#### Janssen Vaccines & Prevention B.V.\*

#### Clinical Protocol

A randomized, parallel-group, placebo-controlled, double-blind Phase 1/2a study in healthy HIV uninfected adults to assess the safety/tolerability and immunogenicity of 2 different prime/boost regimens; priming with trivalent Ad26.Mos.HIV and boosting with trivalent Ad26.Mos.HIV and Clade C gp140 plus adjuvant OR priming with tetravalent Ad26.Mos4.HIV and Clade C gp140 plus adjuvant

#### VAC89220HPX2004

## IPCAVD-011

## Protocol VAC89220HPX2004 Amendment 5; Phase 1/2a

JNJ-55471468, JNJ-55471494, JNJ-55471520, JNJ-55471585, JNJ-64219324

These compounds are being investigated in Phase 1/2a clinical studies.

\*Janssen Vaccines & Prevention B.V. (formerly known as Crucell Holland B.V.) is a Janssen pharmaceutical company of Johnson & Johnson and is hereafter referred to as the sponsor of the study. The sponsor is identified on the Contact Information page that accompanies the protocol.

**Status:** Approved

**Date:** 28 October 2021

**EDMS number:** EDMS-ERI-109992464, 12.0

**GCP Compliance:** This study will be conducted in compliance with Good Clinical Practice, and applicable regulatory requirements.

#### **Confidentiality Statement**

The information provided herein contains Company trade secrets, commercial or financial information that the Company customarily holds close and treats as confidential. The information is being provided under the assurance that the recipient will maintain the confidentiality of the information under applicable statutes, regulations, rules, protective orders or otherwise.

Status: Approved, Date: 28 October 2021

# **TABLE OF CONTENTS**

| TABLE OF CONTENTS | 2 |
|---|---|
| LIST OF ATTACHMENTS | 4 |
| LIST OF IN-TEXT TABLES AND FIGURES | 4 |
| PROTOCOL AMENDMENTS | 5 |
| SYNOPSIS | 11 |
| TIME AND EVENTS SCHEDULE | 17 |
| ABBREVIATIONS | |
| 1.1. Background | |
| 1.1.1. Nonclinical Studies | |
| 1.1.1.1. Repetitive gp120/gp140 Vaccinations | |
| 1.1.1.2. Ad26/gp140 and Ad26/Ad35 Vaccinations | |
| 1.1.1.3. Ad26/Ad5 and Repetitive gp140 Vaccinations | |
| 1.1.1.4. Tetravalent Ad26 Vaccinations | |
| 1.1.2. Clinical Studies | |
| 1.1.2.1. Prototypes and Similar Vaccines | |
| 1.1.2.1.1. Ad5 and Ad26 Vaccines | |
| 1.1.2.1.2. gp120 Vaccines | |
| 1.1.2.2. Current Studies | |
| 1.2. Overall Rationale for the Study | 28 |
| 2. OBJECTIVES, ENDPOINTS, AND HYPOTHESIS | |
| 2.1. Objectives and Endpoints | |
| 2.1.1. Objectives | |
| 2.1.2. Endpoints | |
| 2.2. Hypothesis | 30 |
| 3. STUDY DESIGN AND RATIONALE | 30 |
| 3.1. Overview of Study Design | |
| 3.2. Study Design Rationale | |
| 4. SUBJECT POPULATION | 32 |
| 4.1. Inclusion Criteria for the Main Study | |
| 4.2. Exclusion Criteria for the Main Study | |
| 4.3. Prohibitions and Restrictions | |
| 4.4. Inclusion and Exclusion Criteria for the Optional Long-term Extension Phase | |
| 5. TREATMENT ALLOCATION AND BLINDING | 38 |
| 6. DOSAGE AND ADMINISTRATION | 39 |
| 7. TREATMENT COMPLIANCE | |
| 9. STUDY EVALUATIONS | |
| 9.1. Study Procedures | |
| 9.1.1. Overview | 41 |
| 9.1.2. Visit Windows | 42 |
| 9.1.3. Screening Phase (Weeks -4 to 0) | 44 |

| 9.1.4. | Vaccination | 45 |
|---|---|---|
| 9.1.5. | Post-vaccination Follow-Up Phase | 47 |
| 9.1.6. | Follow-Up Phase | |
| 9.1.7. | Early Withdrawal/Exit Visit | |
| 9.1.8. | Optional Long-term Extension Phase | |
| 9.2. | Immunogenicity Evaluations | 49 |
| 9.3. | Safety Evaluations | |
| 9.4. | Human Immunodeficiency Virus Testing and Vaccine Induced Seropositivity | 54 |
| 9.4.1. | Human Immunodeficiency Testing | 54 |
| 9.4.2. | Management of Subjects who Become HIV-infected During the Study | |
| 9.4.3. | VISP | |
| 9.4.4. | Social Impact | |
| 9.5. | Sample Collection and Handling | 55 |
| 10. S | UBJECT COMPLETION/DISCONTINUATION OF STUDY TREATMENT/WITHDRAWAL | |
| | ROM THE STUDY | 56 |
| 10.1. | Completion | |
| 10.2. | Discontinuation of Study Treatment | |
| 10.3. | Contraindications to Vaccination | |
| 10.4. | Withdrawal From the Study | |
| 10.5. | Withdrawal From the Use of Samples in Future Research | |
| 10.0. | William and Trom the Coo of Campios in Fataro Rossaron | |
| 11. S | TATISTICAL METHODS | <mark>58</mark> |
| 11.1. | Subject Information | 58 |
| 11.2. | Analysis Populations | 58 |
| 11.3. | Sample Size Determination | <mark>58</mark> |
| 11.4. | Immunogenicity Analyses | <mark>59</mark> |
| 11.5. | Safety Analyses | <mark>59</mark> |
| 11.6. | Analysis Time Points | 60 |
| 11.7. | PSRT | <mark>61</mark> |
| 11.8. | DRC | |
| 11.9. | Study Holding Rules | 62 |
| 40 4 | E DEDODTINO | |
| | E REPORTING | |
| 12.1. | Definitions | |
| 12.1.1. | | |
| 12.1.2. | Attribution Definitions | |
| 12.1.3. | Severity Criteria | |
| 12.2. | Situations Requiring Special Notification | |
| 12.2.1. | AESI | |
| 12.3. | Procedures | |
| 12.3.1. | All AEs | |
| 12.3.2. | SAEs | |
| 12.3.3. | HIV Infection | |
| 12.3.4. | Pregnancy | |
| 12.4. | Contacting Sponsor Regarding Safety | 70 |
| 13. P | RODUCT QUALITY COMPLAINT HANDLING | 70 |
| 13.1. | Procedures | |
| 13.1. | Contacting Sponsor Regarding Product Quality | |
| 10.2. | Contacting Openior Regarding Freduct Quality | 10 |
| 14. V | ACCINE INFORMATION | <mark>71</mark> |
| 14.1. | Physical Description of Study Vaccines | |
| 14.2. | Packaging and Labeling | |
| 14.3. | Preparation, Handling, and Storage | |
| 14.4. | Vaccine Accountability | |
| | · | |
| 15. S | TUDY-SPECIFIC MATERIALS | <b>73</b> |

| 16. ETI | HICAL ASPECTS | <mark>74</mark> |
|---|---|---|
| 16.1. S | Study-specific Design Considerations | 74 |
| 16.2. F | Regulatory Ethics Compliance | <mark>76</mark> |
| 16.2.1. | Investigator Responsibilities | |
| 16.2.2. | Independent Ethics Committee or Institutional Review Board | <mark>76</mark> |
| 16.2.3. | Informed Consent | <mark>78</mark> |
| 16.2.4. | Privacy of Personal Data | |
| 16.2.5. | Long-term Retention of Samples for Additional Future Research | 79 |
| 17. AD | MINISTRATIVE REQUIREMENTS | 80 |
| 17.1. F | Protocol Amendments | 80 |
| | Regulatory Documentation | |
| 17.2.1. | Regulatory Approval/Notification | |
| 17.2.2. | Required Prestudy Documentation | |
| 17.3. S | Subject Identification, Enrollment, and Screening Logs | 81 |
| | Source Documentation | |
| | Case Report Form Completion | |
| | Data Quality Assurance/Quality Control | |
| | Record Retention | |
| | Monitoring | |
| 17.9. S | Study Completion/Termination | |
| 17.9.1. | Study Completion/End of Study | |
| 17.9.2. | Study Termination | |
| | On-Site Audits | |
| 17.11. L | Jse of Information and Publication | 85 |
| | VID-19 APPENDIX: GUIDANCE ON STUDY CONDUCT DURING THE COVID-19 | |
| PAI | NDEMIC | <mark>87</mark> |
| | NDEMIC | |
| REFERE | NCES | 89 |
| REFERE<br>INVESTI | GATOR AGREEMENT | 89<br>117 |
| REFERE<br>INVESTI | NCES | 89<br>117 |
| REFERE<br>INVESTI | GATOR AGREEMENT | 89<br>117 |
| REFERE<br>INVESTIC | GATOR AGREEMENT | 89<br>117 |
| REFERE INVESTIC LAST PA | GATOR AGREEMENT AGE F ATTACHMENTS ent 1: Division of Aids Table for Grading the Severity of Adult and Pediatric AEs – | 89<br>117<br>117 |
| REFERE INVESTION LAST PA | GATOR AGREEMENT AGE F ATTACHMENTS ent 1: Division of Aids Table for Grading the Severity of Adult and Pediatric AEs – Including Modifications | <b>89</b><br><b>117</b><br><b>117</b> |
| REFERE INVESTION LAST PA LIST ON Attachmen | GATOR AGREEMENT AGE F ATTACHMENTS ent 1: Division of Aids Table for Grading the Severity of Adult and Pediatric AEs – Including Modifications | <b>89 117 117 91</b> 113 |
| REFERE INVESTION LAST PA LIST ON Attachment Attachment Attachment | GATOR AGREEMENT AGE The property of Adult and Pediatric AEs — Including Modifications Includi | <b>89 117 117 91</b> 113 |
| REFERE INVESTION LAST PA LIST ON Attachmen | GATOR AGREEMENT AGE F ATTACHMENTS ent 1: Division of Aids Table for Grading the Severity of Adult and Pediatric AEs – Including Modifications | <b>89 117 117 91</b> 113 |
| REFERE INVESTION LAST PA LIST ON Attachment Attachment Attachment Attachment Attachment | F ATTACHMENTS ent 1: Division of Aids Table for Grading the Severity of Adult and Pediatric AEs – Including Modifications | <b>89 117 117 91</b> 113 |
| REFERE INVESTION LAST PA LIST ON Attachment Attachment Attachment Attachment Attachment | GATOR AGREEMENT AGE The property of Adult and Pediatric AEs — Including Modifications Includi | <b>89 117 117 91</b> 113 |
| REFERE INVESTION LAST PA LIST ON Attachment Attachment Attachment Attachment Attachment | GATOR AGREEMENT AGE F ATTACHMENTS ent 1: Division of Aids Table for Grading the Severity of Adult and Pediatric AEs – Including Modifications ent 2: HIV-risk Assessment ent 3: Test of Understanding ent 4: Social Impact Questionnaire F IN-TEXT TABLES AND FIGURES | <b>89 117 117 91</b> 113 |
| REFERE INVESTION LAST PA LIST ON Attachment Attachment Attachment Attachment LIST ON | GATOR AGREEMENT AGE F ATTACHMENTS ent 1: Division of Aids Table for Grading the Severity of Adult and Pediatric AEs – Including Modifications ent 2: HIV-risk Assessment ent 3: Test of Understanding ent 4: Social Impact Questionnaire F IN-TEXT TABLES AND FIGURES | <b>89 117 117 91</b> 115 116 |

### PROTOCOL AMENDMENTS

| <b>Protocol Version</b> | Issue Date |
|-------------------------|-------------------|
| Original Protocol | 21 Jan 2016 |
| Amendment 1 | 16 Sep 2016 |
| Amendment 2 | 20 September 2017 |
| Amendment 3 | 27 March 2020 |
| Amendment 4 | 28 July 2020 |
| Amendment 5 | This document |

Amendments below are listed beginning with the most recent amendment.

### <u>Amendment 5</u> (This document)

**The overall reason for the amendment:** In this amendment, the LTE phase is being shortened by one year, since this vaccine regimen did not provide statistically significant protection against HIV infection in study HPX2008/HVTN 705.

**Rationale:** The LTE phase is being shortened by one year. Visit 26 and Visit 27 will be removed and Visit 25 will become the last visit in the study. Participants who already had their Visit 25 or Visit 26 will be contacted to perform an extra unscheduled exit visit, to be performed within 6 weeks after local approval of protocol amendment 5.

#### **SYNOPSIS**

Time and Events Schedule

- 1.2 Overall Rationale for the Study
- 3.1 Overview of Study Design
- 9.1.1 Overview
- 9.1.2 Visit Windows
- 9.1.8 Optional Long-term Extension Phase
- 10.1 Completion
- 11.6 Analysis Time Points
- 16.1 Study-specific Design Considerations
- 16.2.3 Informed Consent

**Rationale:** The background section of the protocol has been updated with a summary of the HPX2008/HVTN 705 results.

1.1.2.2 Current Studies

**REFERENCES** 

## **Amendment 4** (28 July 2020)

The overall reason for the amendment: In this amendment, it is clarified that if a visit of the LTE phase can't be scheduled within the allowed window, it will be assessed on a case-by-case basis whether this visit can still be performed. In addition, an appendix has been included to outline temporary measures while access to the sites is restricted during public health crises such as e.g., COVID-19 outbreak and to provide investigators with flexibility to conduct study assessments while ensuring the safety and well-being of the subjects and site staff during the pandemic. These measures will not be described in the body of the protocol but rather outlined in an Appendix (Section 18).

**Rationale:** It is clarified that if a visit of the LTE phase can't be scheduled within the allowed window, it will be assessed on a case-by-case basis upon discussion between investigator and sponsor whether this visit can still be performed. In addition, a clarification has been added to interpret 1 month as 30 days, and 1 week as 7 days; hence, the visit window for visit 23 ought to be interpreted as -28 days/+60 days.

Time and Events Schedule

9.1.2 Visit Windows

**Rationale:** A COVID-19 Appendix has been added to provide guidance to investigators for managing study-related procedures during the COVID-19 pandemic. For health and safety reasons, subjects may not be able to come to the study site for scheduled procedures.

#### **SYNOPSIS**

Time and Events Schedule

- 3.1 Overview of Study Design
- 9.1.2 Visit Windows

18 COVID-19 APPENDIX: GUIDANCE ON STUDY CONDUCT DURING THE COVID-19 PANDEMIC

#### Amendment 3 (27 March 2020)

The overall reason for the amendment: In this amendment, Janssen is offering an additional optional 2-year extension to those participants who have completed the current optional 3-year LTE phase. This will allow a total LTE phase of 5 years after the end of the main study to assess durability of immunologic responses.

**Rationale:** Based on the currently available durability data of immune responses<sup>22,23</sup>, the sponsor aims to evaluate the persistence of these responses over 5.5 years after the last (4th) vaccination. Therefore, an optional 2-year extension of the 3-year LTE phase was introduced.

#### **SYNOPSIS**

Time and Events Schedule

- 1.2 Overall Rationale for the Study
- 3.1 Overview of Study Design
- 4.4 Inclusion and Exclusion Criteria for the Optional Long-term Extension Phase
- 9.1.1 Overview
- 9.1.2 Visit Windows
- 9.1.8 Optional Long-term Extension Phase
- 10.1 Completion
- 11.6 Analysis Time Points
- 16.1 Study-specific Design Considerations
- 16.2.3 Informed Consent

**REFERENCES** 

**Rationale:** It is clarified that subjects may be excluded from donating blood following vaccination in the study due to vaccine induced seropositivity (VISP) for as long as VISP persists, as the screening HIV tests most often used on donated blood (ELISA) will often be positive.

#### 4.3 Prohibitions and Restrictions

**Rationale:** Text has been added to allow modifications in study visits and assessments in the event of emergencies (possibly affecting a site, a region, a country or world-wide).

Time and Events Schedule

- 9.1.1 Overview
- 9.1.2 Visit Windows

**Rationale:** The Confidentiality Statement was revised and the statement 'CONFIDENTIAL – FOIA Exemptions Apply in U.S.' was added to the running footer, to comply with an update from Janssen's Legal department.

Title page

## Amendment 2 (20 September 2017)

The overall reason for the amendment: In this amendment, an optional Long-term Extension (LTE) phase was introduced to assess the durability of immunologic responses up to approximately 3 years after the end of the main study. In addition, clarifications and adjustments were added with regards to the Week 16 interim immunogenicity analysis, the eligibility criteria of the main study, the need for microscopic reflex testing, the definition of the per protocol immunogenicity population, the possibility to perform guest visits, and the follow-up procedures of the main study.

**Rationale:** To assess the durability of the immune responses, an optional LTE phase of approximately 3 years was introduced for subjects randomized to Group 2A, who have received all 4 vaccinations and are negative for HIV infection at the end of the main study. The vaccination regimen of Group 2A (including Ad26.Mos4.HIV and Clade C gp140) forms the basis for the regimens that will likely be evaluated in future studies.

### **SYNOPSIS**

Time and Events Schedule

- 1.2 Overall Rationale for the Study
- 2.1.1 Objectives
- 2.1.2 Endpoints
- 3.1 Overview of Study Design
- 4.1 Inclusion Criteria for the Main Study
- 4.2 Exclusion Criteria for the Main Study
- 4.3 Prohibitions and Restrictions
- 4.4 Inclusion and Exclusion Criteria for the Optional Long-term Extension Phase
- 5 TREATMENT ALLOCATION AND BLINDING
- 8 PRESTUDY AND CONCOMITANT THERAPY
- 9.1.1 Overview
- 9.1.2 Visit Windows
- 9.1.6 Follow-Up Phase
- 9.1.7 Early Withdrawal/Exit Visit
- 9.1.8 Optional Long-term Extension Phase
- 9.3 Safety Evaluations
- 9.4.1 Human Immunodeficiency Testing
- 9.4.2 Management of Subjects who Become HIV-infected During the Study
- 10.1 Completion
- 10.2 Discontinuation of Study Treatment
- 10.4 Withdrawal From the Study
- 11.3 Sample Size Determination
- 11.6 Analysis Time Points
- 12.3.1 All AEs
- 12.3.2 SAEs
- 12.3.3 HIV Infection
- 16.1 Study-specific Design Considerations
- 16.2.3 Informed Consent

**Rationale:** In order to accelerate the availability of preliminary immunogenicity data, an interim immunogenicity analysis will be performed once approximately 60 subjects have completed the Week 16 visit.

#### 5 TREATMENT ALLOCATION AND BLINDING

11.6 Analysis Time Points

**Rationale:** It was clarified that subjects are not eligible for participation to the study if they received an experimental vaccine (other than a prophylactic or therapeutic HIV vaccine candidate) within the last 12 months prior to the Day 1 visit (Vaccination 1).

### 4.2 Exclusion Criteria for the Main Study

#### 8 PRESTUDY AND CONCOMITANT THERAPY

**Rationale:** It was indicated that microscopic reflex testing will not be carried out in the event of abnormal urinalysis tests that are considered by the investigator to have a menstrual origin.

#### 9.3 Safety Evaluations

**Rationale:** A definition of the per protocol immunogenicity population was added to exclude subjects with major protocol deviations from the immunogenicity population.

#### 11.2 Analysis Populations

#### 11.4 Immunogenicity Analyses

**Rationale:** It was indicated that subjects who are temporarily not able to attend the per protocol visits at their clinical site due to travel (eg, vacation, business travel) may visit any other clinical site participating in this clinical study for non-vaccination visits.

#### 9.1.1 Overview

**Rationale:** It was clarified that a (remote) safety follow-up communication 24-72 hours post vaccination is not required if the vaccination was missed.

#### Time and Events Schedule

#### 9.1.5 Post-vaccination Follow-Up Phase

**Rationale:** It was clarified that subjects who prematurely discontinue study treatment will be encouraged to complete the post-vaccination follow-up visits of the last vaccination received and a 12 and 24 weeks follow-up visit after the last vaccination received.

#### Time and Events Schedule

10.2 Discontinuation of Study Treatment

| Dationala | Minor | alarifications | and corrections |
|-----------|-------|----------------|-----------------|

| SYNOPSIS | An error in the abbreviation of Protocol Safety Review Team (PSRT) was corrected |
|---|---|
| 9.3 Safety Evaluations | Added language that laboratory test ranges will be applied according to subject's sex at birth. |
| 9.4.3 VISP | It was indicated that the central lab will carry out a follow-up testing algorithm in response to a positive result in an HIV-Ab test. |
| 9.4.4 Social Impact | It was indicated that more details regarding completion<br>of the social impact questionnaire can be found in the<br>Study Procedures Manual. |
| 10.4 Withdrawal From the Study | It was clarified that subjects who are vaccinated and who withdraw will not be replaced. |
| 12.3.2 SAEs | Administrative change |
| Attachment 4 | It was clarified that adaptations to the social impact<br>questionnaire are allowed for local purposes, after IRB<br>and sponsor approval. |

#### **Amendment 1** (16 Sep 2016)

The overall reason for the amendment: The contraceptive requirements have been adapted, to align with recent changes in company policy to become aligned with the general standards for contraceptive use in vaccine trials...

**Rationale:** Changes in the contraceptive requirement in the inclusion criteria to align with updated company policies regarding standard contraceptive use in vaccine studies.

- 4.1. Inclusion Criteria
- 4.3. Prohibitions and Restrictions

Rationale: Omission of stratification by region in original protocol rectified.

#### **SYNOPSIS**

- 3.1. Overview of Study Design
- 5. TREATMENT ALLOCATION AND BLINDING

**Rationale:** The HIV RNA test at screening and baseline has been deleted, since evaluation of VISP is not relevant at these timepoints.

#### TIME AND EVENTS SCHEDULE

- 9.4.1. Human Immunodeficiency Testing
- 12.3.3. HIV Infection

**Rationale:** Specifications added for the screening window: Eligible subjects who are late for the baseline visit should have screening tests repeated.

9.1.3 Screening Phase (Weeks -4 to 0)

**Rationale:** From 1 Jun 2016 onwards, the name of Crucell Holland B.V. has been changed to Janssen Vaccines & Prevention B.V.

Title page

**Rationale:** It is clarified that the extra 2 weeks of screening to allow for start of hormonal contraception are applicable for female subjects and for female partners of male subjects.

#### **SYNOPSIS**

TIME AND EVENTS SCHEDULE

- 3.1 Overview of Study Design
- 4. SUBJECT POPULATION
- 9.1.2 Visit Windows
- 9.1.3 Screening Phase (Weeks -4 to 0)

| Rationale: Minor clarifications | |
|---|---|
| TIME AND EVENTS SCHEDULE 9.3. Safety Evaluations | Changed wordings from 'positive' to 'abnormal' urinalysis. |
| SYNOPSIS TIME AND EVENTS SCHEDULE 9.1.5. Post-vaccination Follow-Up Phase 11.7. PSRT | Time indication of 72 hours simplified to 3 days. |
| 5. TREATMENT ALLOCATION AND BLINDING | Specified that blind should not be broken before eDC (electronic data capture) database is closed. |
| Rationale: Minor corrections | |
| 9.3. Safety Evaluations | Removed redundant reference to Section 12.1.1. |
| 1.1.2.2. Current Studies | Typographical error corrected |

# Clinical Protocol VAC89220HPX2004 Amendment 5

| 12.3.2. SAEs | Updated methods of reporting SAE to include email |
|---|---|
| 12.1.2. Attribution Definitions | Definition of 'related AE' has been altered to align with definition in more recent study protocols |
| 17.5. Case Report Form Completion | Removed statement that all data should be recorded in CRF |
| <ul><li>10.5. Withdrawal From the Use of Samples in Future Research</li><li>16.2.3. Informed Consent</li></ul> | Removed wordings in reference to optional research samples as this is not applicable for this study. |
| 16.2.5. Long-term Retention of Samples for Additional Future Research | Corrected the cross-reference to Section 10.5 |

Approved, Date: 28 October 2021

### **SYNOPSIS**

A randomized, parallel-group, placebo-controlled, double-blind Phase 1/2a study in healthy HIV uninfected adults to assess the safety/tolerability and immunogenicity of 2 different prime/boost regimens; priming with trivalent Ad26.Mos.HIV and boosting with trivalent Ad26.Mos.HIV and Clade C gp140 plus adjuvant OR priming with tetravalent Ad26.Mos4.HIV and boosting with tetravalent Ad26.Mos4.HIV and Clade C gp140 plus adjuvant

The proposed clinical study will be a first-in-human evaluation (for Ad26.Mos4.HIV) to evaluate the safety/tolerability and immunogenicity of a regimen including trivalent Ad26.Mos.HIV and a regimen including tetravalent Ad26.Mos4.HIV.

#### **OBJECTIVES, ENDPOINTS, AND HYPOTHESIS**

## **Objectives**

#### **Primary Objectives**

- To assess safety/tolerability of the 2 different vaccine regimens.
- To assess Envelope (Env)-binding antibody (Ab) responses of the 2 different vaccine regimens.

## Secondary Objectives

- To assess neutralizing Ab (nAb) responses, Ab functionality (as assessed by phagocytosis), and Ab isotyping.
- To assess T-cell responses.

## **Exploratory Objectives**

- To explore Ab functionality (other than phagocytosis).
- To explore Ab Fc characterization.
- To explore T-cell and Ab epitope mapping.
- To explore gene expression of peripheral blood mononuclear cells (PBMCs).
- To explore B-cell responses.
- To explore immune responses against the viral vector.
- To assess the social impact of participation in a human immunodeficiency virus (HIV)-vaccine study for subjects via a social impact questionnaire.
- To explore durability of the immune responses to the vaccine regimen in the group selected for the optional Long-term Extension (LTE) phase.

### **Endpoints**

## **Primary Endpoints**

• AEs throughout the study

Local and systemic solicited adverse events (AEs) for 7 days post-vaccination.

AEs for 28 days after each vaccination.

Discontinuations from vaccination/from study due to AEs.

Serious AEs (SAEs) and AEs of special interest (AESIs) during the course of the study, including the optional LTE phase.

• Env-specific binding Abs (titers and breadth).

### Secondary Endpoints

- Env-specific nAbs (titers and breadth) (for Tier 1 and Tier 2 viruses; note: Tier 2 will be assessed only if Tier 1 shows positive results).
- Env-specific functional Abs (phagocytosis score and breadth).
- Env-specific binding Ab isotypes (IgA, IgG1-4) (titers and breadth).
- Interferon (IFN)γ PBMC responders to mosaic peptide pools of Env/group-specific antigen (Gag)/polymerase (Pol) and potential T-cell epitopes (PTE).
- Cluster of differentiation (CD)4<sup>+</sup> and CD8<sup>+</sup> T-cell functionality (% cells producing ia, IFNγ, IL-2, IL-4, TNFα).
- T-cell development with emphasis on follicular helper T-cells and memory differentiation.
- Available samples from time points after last vaccination until the final main study visit at Week 72 will be used for determination of durability of the immune responses.

## **Exploratory Endpoints**

- Ab functionality evaluation (by other than phagocytosis).
- Ab Fc (sub)typing.
- Epitope mapping of Ab to Env and T-cell responses to Gag/Pol/Env and PTE.
- Regulation of genes (clusters) that predict specific immune responses and human leukocyte antigen typing.
- Ab-producing B-cells and characterization of B-cell memory development.
- Adenovirus serotype 26 (Ad26) nAbs (titer).
- Available samples from time points during the optional LTE phase will be used for determination of long-term durability of the immune responses.

## **Hypothesis**

No formal statistical hypothesis will be tested. This study will evaluate whether 2 vaccine regimens, priming with Ad26.Mos.HIV or Ad26.Mos4.HIV and boosting with Clade C gp140 together with Ad26.Mos.HIV or Ad26.Mos4.HIV, are safe, well-tolerated, and immunogenic, providing broad, functional, and durable humoral and cellular responses.

### **OVERVIEW OF STUDY DESIGN**

This is a randomized, double-blind, placebo-controlled, parallel, interventional, Phase 1/2a study in healthy HIV-uninfected adult men and women aged 18 through 50 years. A target of 198 subjects will participate in this study, randomized into one of 4 subgroups: 55 subjects will receive vaccination with Ad26.Mos.HIV and Clade C gp140 in Subgroup 1A, 11 subjects will receive placebo in Subgroup 1B, 110 subjects will receive vaccination with Ad26.Mos4.HIV and Clade C gp140 in subgroup 2A and 22 subjects will receive placebo in Subgroup 2B. Randomization will be stratified by region. Subjects will be enrolled regardless of their baseline Ad26 seropositivity.

The main study will be conducted in 3 phases: a 4-week screening period (with 2 extra weeks to allow for start of hormonal contraception for female subjects or female partners of male subjects); a 48-week vaccination period during which subjects will be vaccinated at baseline (Week 0) and Weeks 12, 24, and 48; and a follow-up period to the final main study visit at Week 72. An optional LTE phase (approximately 3 or 4 years after Week 72, depending on the length of follow-up which subjects consent to) will be performed for subjects randomized to Group 2A, who have received all 4 vaccinations and are negative for HIV infection at Week 72. The vaccination regimen of Group 2A (including Ad26.Mos4.HIV and Clade C gp140) forms the basis for the regimens that will likely be evaluated in future studies. The duration of the subject's participation will be approximately 76 weeks for subjects not participating in the optional LTE phase and approximately 220 or 268 weeks for subjects participating in the optional LTE phase (approximately 3 or 4 years after the end of the main study, respectively).

After vaccination, subjects will remain under observation at the study site for at least 30 minutes for presence of any acute reactions and solicited events. In addition, subjects will record solicited local (at injection site) and systemic events in a diary for 7 days post-vaccination. Further safety evaluations will include monitoring of AEs, physical examinations, vital sign measurements, clinical laboratory tests, and pregnancy testing until Week 72. Blood samples will be taken at specific clinic visits to assess immune responses. Subjects will complete a social impact questionnaire at specific clinic visits. A Protocol Safety Review Team (PSRT) and Data Review Committee (DRC) will be commissioned for this study.

A COVID-19 Appendix provides guidance to investigators for managing study-related procedures during the COVID-19 pandemic.

| Study De | sign VAC892 | 20HPX | 2004 | | | |
|---|---|---|---|---|---|---|
| Group | Subgroup | N | Week 0 | Week 12 | Week 24 | Week 48 |
| Group 1 | | | | | Ad26.Mos.HIV | Ad26.Mos.HIV |
| | A | 55 | Ad26.Mos.HIV | Ad26.Mos.HIV | + | + |
| Group 1 | | 55 Ad26.Mos.l | | | Clade C gp140<br>(250 mcg + adjuvant) <sup>a</sup> | Clade C gp140<br>(250 mcg + adjuvant) <sup>a</sup> |
| • | | | | | Placebo | Placebo |
| | В | 11 | Placebo | Placebo | + | + |
| | | | | | Placebo | Placebo |
| | | | | | Ad26.Mos4.HIV | Ad26.Mos4.HIV |
| | $A^b$ | p N 55 | Ad26.Mos4.HIV | Ad26.Mos4.HIV | + | + |
| Group 2 | | | | | Clade C gp140<br>(250 mcg + adjuvant) <sup>a</sup> | Clade C gp140 (250<br>mcg + adjuvant) <sup>a</sup> |
| - ··r - | | | | | Placebo | Placebo |
| | В | 22 | Placebo | Placebo | + | + |
| | | | | | Placebo | Placebo |

 $<sup>^{</sup>a}250$  mcg refers to total protein content; sterile aluminum phosphate suspension will be used as adjuvant. Aluminum content will be 0.425 mg/0.5 mL dose.

## **PSRT**

The PSRT will review blinded safety data reports on a regular basis (at least 2 times per month) starting from one week after first vaccination until the last subject has completed the Week 52 visit, and thereafter as needed.

<sup>&</sup>lt;sup>b</sup>An optional LTE phase (approximately 3 or 4 years after Week 72 depending on the length of follow up which subjects consent to) will be performed for subjects randomized to Group 2A, who have received all 4 vaccinations and are negative for HIV infection at Week 72.

After a sentinel group of 10 subjects received the first injection, further vaccinations will be paused until a 3-day safety evaluation is performed. This evaluation will be performed by the PSRT and the PI(s) of the subjects involved and will be based on the information received from the investigator(s) by email/telephone.

If an administration of vaccine is considered, by PSRT review, to raise significant safety concerns, all enrollment and vaccinations will be suspended until recommendations are issued. In specific cases a Data Review Committee (DRC) meeting will be triggered.

The PSRT will include, but will not be limited to medical and safety representatives from the sponsor, sites, Division of Acquired Immune Deficiency Syndrome (DAIDS), Beth Israel Deaconess Medical Center (BIDMC), HIV Vaccine Trials Network (HVTN), International AIDS Vaccine Initiative (IAVI), and Military HIV Research Program (MHRP). The PSRT responsibilities, authorities, and procedures will be documented in its charter.

#### DRC

A DRC will be established for this study, which will monitor data to ensure the safety and well-being of the subjects enrolled. The DRC will review data as indicated below. The conclusions of the DRC will be communicated to the investigators, the Institutional Review Board/Independent Ethics Committee, and the national regulatory authorities, as appropriate.

The DRC will specifically review safety data (solicited and unsolicited AEs, SAEs, and available laboratory assessments) at 3 time points:

- Review blinded safety data (4 weeks of follow-up) after 15% of subjects have received their first
  injection. The DRC will review these interim safety results and will allow administration of the first
  dose of Ad26.Mos4.HIV/placebo (first injection) in the VAC89220HPX2003 study only if no
  significant safety concerns are identified.
- Review blinded safety data (4 weeks of follow-up) after 30% of subjects have received their first injection.
- Review blinded safety data (4 weeks of follow-up) after 30% of subjects have received their third injection.

In addition, ad hoc review may be performed further to the occurrence of any AE/SAE leading to a study holding situation or at request of the PSRT.

The DRC will include medical experts in vaccines and the HIV therapeutic area and at least one statistician. The DRC may include members from both inside and outside Janssen, but will not include any study team personnel or people otherwise directly involved in the study conduct, data management, or statistical analysis for the study. The DRC responsibilities, authorities, and procedures will be documented in its charter.

#### SUBJECT POPULATION

Screening for eligible subjects will be performed within 4 weeks (with 2 extra weeks to allow for start of hormonal contraception for female subjects or female partners of male subjects) before the first administration of study vaccine/placebo at Week 0.

Study subjects must be healthy (on the basis of physical examination, medical history, laboratory assessments, and vital signs measurement), HIV-uninfected adult men and women, aged  $\geq$ 18 to  $\leq$ 50 years, and assessed by the clinic staff as being at low risk for HIV infection.

For entering the optional LTE phase, subjects must have been randomized to Group 2A during the main study, have received all 4 vaccinations and be negative for HIV infection at the end of the main study.

#### DOSAGE AND ADMINISTRATION

Each subject will receive study vaccine/placebo at 4 time points (see Table Study Design) according to randomization, on Day 1 and Weeks 12, 24, and 48, administered by intramuscular injection into the deltoid. For visits with only one injection (ie, at Weeks 0 and 12), preferably the deltoid of the non-dominant upper arm is used. When 2 injections are to be given at one visit (ie, at Weeks 24 and 48), it is required to use a different deltoid for each injection. Exceptions on injection site are allowed only if medically indicated.

#### Ad26.Mos4.HIV:

Total dose is  $5x10^{10}$  virus particles (vp) per 0.5 mL injection

#### • Ad26.Mos.HIV:

Total dose is 5x10<sup>10</sup> vp per 0.5 mL injection

Ad26.Mos4.HIV and Ad26.Mos.HIV are classified as genetically modified organisms (GMOs). Based on nonclinical biodistribution and shedding data with related vectors, the investigational vaccine is not expected to pose any risk to the environment. Any local requirements related to GMOs must be fulfilled by the investigator.

## • Clade C gp140:

Clade C gp140 with 250 mcg total protein, mixed with aluminum phosphate adjuvant (0.425 mg aluminum) at the pharmacy, per 0.5 mL injection

#### • Placebo:

0.9% saline, 0.5 mL injection

#### **IMMUNOGENICITY EVALUATIONS**

Humoral immune response assays will include, but are not limited to Env-Ab-binding assays, virus neutralization assay, and assays for Ab functionality.

Cellular immune response assays will include, but are not limited to interferon gamma enzyme-linked immunospot assay, intracellular cytokine staining, and multiparameter flow cytometry.

#### SAFETY EVALUATIONS

All AEs and situations requiring special notification will be reported from the time a signed and dated informed consent form (ICF) is obtained until 28 days after first dose of study vaccine, and thereafter, pre-dose and for 28 days after each subsequent dose of study vaccine/placebo. All SAEs and AEs leading to discontinuation from the study vaccination (regardless of the causal relationship) and AESIs (ie, confirmed HIV infection) are to be reported for the duration of the main study. During the optional LTE phase, only SAEs and AESIs are to be reported. Other AEs are not collected during the optional LTE phase as the optional LTE phase begins 6 months after the last vaccination and it is very unlikely that an AE related to the study vaccine would only present that long after the last vaccination.

After each vaccination, subjects will remain under observation at the study site for at least 30 minutes for presence of any acute reactions and solicited events.

In addition, symptoms of the following solicited AEs will be collected via a diary for 7 days post-vaccination (day of vaccination and the subsequent 7 days). The diary will be used as a source document.

- Solicited local AEs: pain/tenderness, erythema, and swelling/induration (measured using the ruler supplied).
- Solicited systemic AEs: fever (temperature measurement), fatigue, headache, nausea, myalgia, and chills.
- Temperature should be measured at approximately the same time each day using the thermometer supplied.

#### STATISTICAL METHODS

Anticipating a dropout rate of approximately 10%, the sample sizes will allow detection of approximately 1.5-fold differences in Env-binding Ab titers between the groups with Ad26.Mos4.HIV (approximately 100 evaluable subjects) and their corresponding group with Ad26.Mos.HIV only (approximately 50 evaluable subjects); with 80% probability, assuming a 1-sided 5% Type I error and a standard deviation of 0.4 on the log<sub>10</sub> scale.

While mild to moderate vaccine reactions (local site and systemic responses) are expected, AEs that preclude further vaccine administration or more serious ones that would limit product development are not anticipated. With 110 individuals in the tetravalent Ad26.Mos4.HIV vaccine regimen, the observation of 0 such reactions would be associated with a 95% confidence that the true rate is <2.7%. For the combined active groups (n=165), there would be 95% confidence that the true rate is <1.8% when 0 events are observed.

## **Immunogenicity Analyses**

No formal hypothesis on immunogenicity will be tested. Descriptive statistics (actual values and changes from reference with 95% confidence interval) will be calculated for continuous parameters. Frequency tabulations will be calculated for discrete parameters. Graphical representations of changes in immunologic parameters will be made as applicable.

## **Safety Analyses**

No formal statistical testing of safety data is planned. Safety data will be analyzed descriptively.

CONFIDENTIAL – FOIA Exemptions Apply in U.S.

# TIME AND EVENTS SCHEDULE

Approved, Date: 28 October 2021

# Time and Events Schedule for Treatment Phase and Follow-up Phase until Week 72

| Phase | Scr | Vac | P | ost va | ıc. FU | IJ | Vac | Post vac. FU | | | Vac Post vac. FU | | | T | Vac | Post vac. FU | | | Sec.<br>Year | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit# | 1 <sup>1</sup> | 2 | 2a <sup>5</sup> | 3 | 4 | 5 | 6 | 6a⁵ | <b>7</b> <sup>2</sup> | 82 | 9 | 9a5 | 10 <sup>2</sup> | 11 <sup>2</sup> | 12 | 13 | 13a <sup>5</sup> | 14 <sup>2</sup> | 15 <sup>2</sup> | 16 | 17 <sup>3</sup> | Exit <sup>4</sup> |
| Visit Week | to 0 | 0 | | 1 | 2 | 4 | 12 | | 14 | 16 | 24 | | 26 | 28 | 36 | 48 | | 50 | 52 | 60 | 72 | |
| Visit Day | 28<br>to<br>0 | 1 | to<br>4 | 8<br>±<br>1 | 15<br>±<br>5 | 29<br>±<br>5 | 85<br>1/+3<br>wks | 86<br>to<br>88 | 99<br>±<br>5 | 113<br>±<br>5 | 169<br>1/+3<br>wks | 170<br>to<br>172 | 183<br>±<br>5 | 197<br>±<br>5 | 253<br>±<br>5 | 337<br>1/+3<br>wks | 338<br>to<br>340 | 351<br>±<br>5 | 365<br>±<br>5 | 421<br>± 3<br>wks | 505<br>± 3<br>wks | |
| Visit Type | Scr | VAC<br>1 | S | S | S<br>+<br>I | S<br>+<br>I | VAC<br>2 | s | S<br>+ I | S+<br>I | VAC<br>3 | S | S+<br>I | S+<br>I | s | VAC<br>4 | S | S+<br>I | S+<br>I | S+<br>I | S+<br>I | Early<br>exit |
| Informed consent <sup>6</sup> | • | | | | | | | | | | | | | | | | | | | | ●3 | |
| Medical history | • | | | | | | | | | | | | | | | | | | | | | |
| Physical exam <sup>7</sup> (incl height <sup>8</sup> and weight <sup>9</sup> ) | • | 0 | | • | • | • | 0 | | • | • | 0 | | • | • | • | 0 | | • | • | • | • | • |
| Vital signs | • | € | | • | • | • | € | | • | • | 8 | | • | • | • | 8 | | • | • | • | • | • |
| HIV-risk assessment | • | • | | • | • | • | • | | • | • | • | | • | • | • | • | | • | • | • | • | • |
| Counseling on HIV | • | • | | • | • | • | • | | • | • | • | | • | • | • | • | | • | • | • | • | • |
| Test of Understanding | • | | | | | | | | | | | | | | | | | | | | | |
| Concomitant meds | • | 0 | | • | • | • | 0 | | • | • | 0 | | • | • | • | 0 | | • | • | • | • | • |
| Review of inclusion/ | • | 0 | | | | | | | | | | | | | | | | | | | | |
| exclusion criteria <sup>10</sup> | | • | | | | | | | | | | | | | | | | | | | | |
| Randomization | | • | | | | | | | | | | | | | | | | | | | | |
| Vaccination | | • | | | | | • | | | | • | | | | | • | | | | | | |
| Post-vac observation (30 min) <sup>11</sup> | | • | | | | | • | | | | • | | | | | • | | | | | | |
| AE recording <sup>12</sup> | • | 8 | • | • | • | • | € | • | • | • | 8 | • | • | • | | 8 | • | • | • | | | • |
| SAE, AE leading to<br>treatment discontinuation,<br>AESI recording <sup>12</sup> | • | 8 | • | • | • | • | 6 | • | • | • | 8 | • | • | • | • | 8 | • | • | • | • | • | • |
| Diary distribution | | • | | | | | • | | | | • | | | | | • | | | | | | |
| Diary review by site staff | | | | Ш | • | | | | • | | | | • | | | | | • | | | | |
| 24h-72h contact | | | ●13 | | | | | • | | | | • | | | | | • | | | | | |
| Social impact questionnaire | | | | | | | • | | | | | | | | | • | | | | | • | • |

| Phase | Scr | Vac | P | ost ve | ac. Fl | U | Vac | Pos | st vac. | <b>FU</b> | Vac | | Post v | ac. FU | T | Vac | Pos | st vac. | FU | | ond<br>FU <sup>3</sup> | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit # | 11 | 2 | 2a <sup>5</sup> | 3 | 4 | 5 | 6 | 6a5 | <b>7</b> <sup>2</sup> | 8 <sup>2</sup> | 9 | 9a5 | 10 <sup>2</sup> | 11 <sup>2</sup> | 12 | 13 | 13a <sup>5</sup> | 14 <sup>2</sup> | 15 <sup>2</sup> | 16 | 173 | Exit <sup>4</sup> |
| Visit Week | to<br>0 | 0 | | 1 | 2 | 4 | 12 | | 14 | 16 | 24 | | 26 | 28 | 36 | 48 | | 50 | 52 | 60 | 72 | |
| Visit Day | 28<br>to<br>0 | 1 | to 4 | 8<br>±<br>1 | 15<br>±<br>5 | 29<br>±<br>5 | 85<br>1/+3<br>wks | 86<br>to<br>88 | 99<br>±<br>5 | 113<br>±<br>5 | 169<br>1/+3<br>wks | 170<br>to<br>172 | 183<br>±<br>5 | 197<br>±<br>5 | 253<br>±<br>5 | 337<br>1/+3<br>wks | 338<br>to<br>340 | 351<br>±<br>5 | 365<br>±<br>5 | 421<br>± 3<br>wks | 505<br>± 3<br>wks | |
| Visit Type | Scr | VAC<br>1 | s | s | S<br>+<br>I | S<br>+<br>I | VAC<br>2 | s | S<br>+ I | S+<br>I | VAC<br>3 | s | S+<br>I | S+<br>I | s | VAC<br>4 | s | S+<br>I | S+<br>I | S+<br>I | S+<br>I | Early<br>exit |
| Urinalysis <sup>14</sup> | • | 0 | | | | | 0 | | | | 0 | | | | | 0 | | | | | • | • |
| Serum pregnancy test <sup>15</sup> | • | | | | | | | | | | | | | | | | | | | | | |
| Urine pregnancy test <sup>15</sup> | | 0 | | | | | 0 | | | | 0 | | | | | 0 | | | | | | • |
| Pregnancy counseling <sup>16</sup> | • | • | | | | | • | | | | • | | | | | • | | | | | | • |
| CBC with differential and platelets <sup>17</sup> | • | 0 | | | • | | 0 | | • | | 0 | | • | | • | • | | • | | • | • | • |
| Serum chemistry <sup>17</sup> | • | 0 | | | • | | 0 | | • | | 0 | | • | | • | 0 | | • | | • | • | • |
| Hepatitis B/C serologies | 2 | | | | | | | | | | | | | | | | | | | | | |
| Syphilis serology | 2 | | | | | | | | | | | | | | | | | | | | | |
| Urine chlamydia/ | • | | | | | | | | | | | | | | | | | | | | | |
| gonorrhea | | | | | | | | | | | | | | | | | | | | | | |
| Trichomonas <sup>15,18</sup> | • | | | | | | | | | | | | | | | | | | | | | |
| HIV EIA | • | • | | | | | • | | | | • | | | | | • | | | | | • | • |
| HIV RNA | | | | | | | 2 | | | | 2 | | | | | 0 | | | | | 0 | 0 |
| HLA test | | 2 | | | | | | | | | | | | | | | | | | | | |
| Humoral immuno. assays | | 0 | | | • | • | 0 | | • | • | 0 | | • | • | | • | | • | • | • | • | • |
| Cellular immuno. assays | | 0 | | | | • | | | • | • | | | • | • | | | | • | • | • | • | • |

AE = adverse event; AESI = AE of special interest; CBC = complete blood count; EIA = enzyme immunoassay; FU = follow-up; HIV = human immunodeficiency virus; h = hour; HLA = human leukocyte antigen; min = minutes; immuno. = immunogenicity; incl = including; RNA = ribonucleic acid; S = safety; S + I = safety + immunogenicity; SAE = serious adverse event; scr = screening; vac = vaccination; wk = week

<sup>•</sup> pre-dose; • no extra blood required; • pre- and post-dose

<sup>&</sup>lt;sup>1</sup>Screening visit may be split into multiple days/visits. The maximum screening period is 4 weeks, with the exception of female subjects or female partners of male subjects starting hormonal contraception. In this case, the maximum screening period is 6 weeks.

<sup>&</sup>lt;sup>2</sup>Timings of visits at 2 and 4 weeks post-vaccination will be determined relative to the actual day of vaccination.

<sup>&</sup>lt;sup>3</sup>All subjects will be followed up until Week 72 to assess durability of immune response. Subjects who prematurely discontinue study treatment will be encouraged to complete the post-vaccination follow-up visits of the last vaccination received and a 12 and 24 weeks follow-up visit after the last vaccination received, specified as Week 60 and Week 72. Upon sponsor unblinding at the Week 28 analysis, subjects randomized to Group 2A who have received all 4 vaccinations, will be asked to participate in the optional LTE phase and sign the ICF appendix for the optional LTE phase at Week 72. During the first visit of the optional LTE phase, the

remaining eligibility criteria for the optional LTE phase will be verified. Subjects who attend their Week 72 visit prior to the sponsor's unblinding at the Week 28 analysis, will be enrolled in the optional LTE phase if they consent and sign the ICF appendix for the optional LTE phase and meet the eligibility criteria for the optional LTE phase. When the Week 28 sponsor unblinding subsequently occurs, subjects that started the optional LTE phase but turn out not to be in Group 2A of the main study will be withdrawn from the optional LTE phase. If signing the ICF appendix is not possible at Week 72, signing should be performed at an extra visit (Visit 17bis) as soon as possible after Week 72 and at the latest before any assessment is done on the first visit of the optional LTE phase. See Time and Events Schedule for the Optional Long-term Extension Phase.

<sup>4</sup>For those subjects who are unable to continue participation in the study, an exit visit will be conducted as soon as possible.

<sup>5</sup>Within 24-72 hours post-vaccination a member of the site staff will have a (remote) safety follow-up communication with the subject (by e-mail, telephone, or visit; according to the subject's preference). A (remote) safety follow-up communication 24-72 hours post-vaccination is not required if the vaccination was missed. 
<sup>6</sup>Must be signed before first study-related activity.

<sup>7</sup>Complete physical exam will be performed at screening and final main study visits. At all other visits, an abbreviated, symptom-directed exam will be performed as indicated by the investigator. Weight will be measured at every visit.

<sup>8</sup>Only at screening.

<sup>9</sup>Only pre-dose.

<sup>10</sup>Minimum criteria for the availability of documentation supporting the eligibility criteria are described in Section 17.4. Check clinical status again before first dose of study vaccine.

<sup>11</sup>Observation at the study site for at least 30 min for presence of any acute reactions and solicited events.

<sup>12</sup>Local and systemic solicited events will be recorded for 7 days post-vaccination; AEs will be recorded from signing of ICF onwards until 28 days after first vaccination, and thereafter, pre-dose and for 28 days after each subsequent vaccination; SAEs, AEs leading to treatment discontinuation, and AESIs will be recorded throughout the study.

<sup>13</sup>For the sentinel group of 10 subjects, this will need to be an actual visit at 3 days post vaccination.

<sup>14</sup>Microscopic reflex testing in the event of abnormal urinalysis.

<sup>15</sup>For female subjects only.

<sup>16</sup>For both male and female subjects.

<sup>17</sup>If medical status and physical examination on Day 1 suggests significant changes may have occurred since screening, the clinically relevant screening assessments will be repeated and the Day 1 visit rescheduled. If the repeat screening assessment causes the subject to fall outside the screening window, all screening safety procedures should be repeated so that they are not more than 28 days prior to the Day 1 visit. In case a Grade 3 or 4 laboratory abnormality, or any laboratory abnormality accompanied by clinically relevant signs or symptoms occurs (from the baseline visit onwards), all attempts will be made to perform a confirmatory test within 48 hours after the results have become available. After that, laboratory tests will be repeated weekly until values are resolved or stable.

<sup>18</sup>Urine or vaginal swab may be used.

Approved, Date: 28 October 2021

Approved, Date: 28 October 2021

| Phase | | Long-term Extension 4 years <sup>3</sup> | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | Long-term Extension 3 years <sup>3</sup> | | | | | | | |
| Visit # | 17<br>bis <sup>1</sup> | 18 <sup>1</sup> | 19 | 20 | 21 | 22 | 23/Final Visit <sup>4</sup> | 24 | 25/Final Visit <sup>4</sup> |
| Visit Week | | 96¹ | 120 | 144 | 168 | 192 | 216 | 240 | 264 |
| Visit Day <sup>5</sup> | | 673<br>± 4 wks | 841<br>± 4<br>wks | 1009<br>± 4<br>wks | 1177<br>± 4<br>wks | 1345<br>± 4 wks | 1513<br>- 4 wks/+ 2 months | 1681<br>± 4 wks | 1849<br>± 4 wks |
| Informed consent | • | | | | | | •3 | | |
| Review of inclusion/<br>exclusion criteria | | • | | | | | | | |
| HIV-risk assessment | | • | • | • | • | • | • | • | • |
| Counseling on HIV | | • | • | • | • | • | • | • | • |
| Concomitant meds <sup>2</sup> | | • | • | • | • | • | • | • | • |
| SAE and AESI recording | | • | • | • | • | • | • | • | • |
| Social impact questionnaire | | • | • | • | • | • | • | • | • |
| HIV EIA | | • | • | • | • | • | • | • | • |
| HIV RNA | | • | • | • | • | • | • | • | • |
| Humoral immuno. assays | | • | • | • | • | • | • | • | • |
| Cellular immuno. assays | | • | • | • | • | • | • | • | • |

AESI = adverse event of special interest; EIA = enzyme immunoassay; HIV = human immunodeficiency virus; RNA = ribonucleic acid; SAE = serious adverse event; wks = weeks.

The timing and events outlined here are subject to modification in the event of emergencies (possibly affecting a site, a region, a country or world-wide). Instructions on specific modifications will depend on the particular situation and could vary by site. At a minimum, all efforts will be made to interact with a participant via telemedicine at the time of a protocol-defined visit. Whereas the implementation of alternative processes should be consistent with the protocol to the extent possible, it may, therefore, not be possible to conduct all assessments at the defined time (or within the designated window). The health and safety of the participant and site staff will be the driving factor in such decision making along with government and/or institutional guidances/mandates. Any such deviations and the reason for any contingency measures implemented, would clearly be described in the study report and IRB/EC and HA notification would be made if required. The COVID 19 Appendix in Section 18 provides guidance to investigators for managing study related procedures during the COVID 19 pandemic.

<sup>1</sup>This visit only needs to occur if the ICF appendix for the optional LTE phase is not signed at Week 72. Visit 17bis should occur as soon as possible after the Week 72 visit. The ICF appendix for the optional LTE phase needs to be signed at the latest before any assessment is done on the first visit of the optional LTE phase.

<sup>2</sup>Restricted to concomitant therapies given in conjunction with an SAE and any chronic or recurrent use of immunomodulators/suppressors and oral or parenteral corticosteroids. Subjects will also be asked during all visits whether they are participating in another clinical study.

- <sup>3</sup> An optional 2-year extension of this 3-year optional LTE is introduced in protocol amendment 3. Subjects will be informed of the option to participate in this 2-year extension at the next possible visit after approval of this amendment. Subjects willing to participate will need to sign the ICF appendix for the 2-year extension at Visit 23. As of protocol amendment 5, this optional extension is reduced from 2 years to 1 year.
- <sup>4</sup> Subjects not willing to participate in the 2-year extension will have their final study visit at Visit 23. For subjects willing to participate: As of protocol amendment 5, the LTE will be shortened by one year, so Visit 26 and Visit 27 have been removed and Visit 25 will be the final visit. Participants who already had their Visit 25 or Visit 26 will be contacted to perform an extra unscheduled exit visit, to be performed within 6 weeks after local approval of protocol amendment 5. This can be either a telephone call or an actual site visit and will need to include the same assessments as in the current Visit 25, except for the social impact questionnaire and blood sampling for HIV and immunogenicity testing. In case a safety issue (including a recent HIV exposure) emerges during the call, the participant might be asked to come to the site for further evaluation.
- <sup>5</sup> If a visit can't be scheduled within the allowed window, it will be assessed on a case-by-case basis upon discussion between the investigator and the sponsor whether this visit can still be performed. Note that 1 month should be interpreted as 30 days and 1 week as 7 days; hence, the visit window for visit 23 ought to be interpreted as -28 days/+60 days.

## **ABBREVIATIONS**

Ab antibody

Ad26 adenovirus serotype 26

ADCP antibody-dependent cellular phagocytosis

AE adverse event

AESI adverse event of special interest
ALT alanine aminotransferase
AST aspartate aminotransferase
β-hCG β-human chorionic gonadotropin
BIDMC Beth Israel Deaconess Medical Center

CBC complete blood count CD cluster of differentiation CRF case report form

DAIDS Division of Acquired Immune Deficiency Syndrome

DMC Data Monitoring Committee
DRC Data Review Committee
eDC electronic Data Capturing

ELISA enzyme-linked immunosorbent assay ELISPOT enzyme-linked immunospot assay

Env envelope

FDA Food and Drug Administration

FIH first-in-human

FSH follicle stimulating hormone
Gag group-specific antigen
GMO genetically modified organism

gp glycoprotein HCV hepatitis C virus

HIV(-1) human immunodeficiency virus (type 1)

HLA human leukocyte antigen HHS Health and Human Services

HVTN Human immunodeficiency virus Vaccine Trials Network

IAVI International Acquired Immune Deficiency Syndrome Vaccine Initiative

ICF informed consent form
ICS intracellular cytokine staining
IEC Independent Ethics Committee

IFN interferon IM intramuscular

IRB Institutional Review Board IWRS interactive web response system

LTE Long-term Extension

MHRP Military Human immunodeficiency virus Research Program

Mos mosaic

MVA Modified Vaccinia Ankara nAb neutralizing antibody

OHRP Office for Human Research Protections PBMC peripheral blood mononuclear cell

Pol polymerase

PSRT Protocol Safety Review Team
PTE potential T-cell epitope
RNA ribonucleic acid

SAE serious adverse event
SIV simian immunodeficier

SIV simian immunodeficiency virus SHIV simian human immunodeficiency virus

TOU Test Of Understanding ULN upper limit of normal

US United States

VISP Vaccine Induced Seropositivity

vp viral particle

### 1. INTRODUCTION

A safe and effective human immunodeficiency virus (HIV) vaccine is the presently elusive cornerstone of HIV prevention.<sup>21</sup> Optimally, both a robust cluster of differentiation (CD) CD4<sup>+</sup> and CD8<sup>+</sup> T-cell responses and a potent humoral response with multiple effectors should be induced by a vaccine. An objective of the HIV-vaccine development program being pursued by the sponsor and its partners is to optimize a vaccine candidate for improved potency, where potency is defined as the quantitative response, frequency, and amplitude of a variety of potent antibody (Ab) and Ab-mediated cellular effector mechanisms, coupled with appropriate cellular responses. A second objective is to increase the breadth of response, defined as immune recognition of diverse strains/clades of HIV to include multiple clades.

A successful global prophylactic HIV vaccine will likely need to protect against the diverse strains and clades of HIV that may be encountered. Improving the magnitude and breadth of epitope coverage is thought to be key to development of a successful Ab and T-cell based preventive HIV vaccine. Strategies to accomplish this include the use of vaccines containing immunogens from a number of prevalent clades and/or using mosaic sequences, ie, proteins assembled from natural sequences of the different clades by in silico recombination, optimized for potential T-cell epitopes.<sup>5</sup>

Vaccines used in this study are Ad26.Mos4.HIV, Ad26.Mos.HIV, and Clade C gp140 (for details see Section 14).

For the most comprehensive nonclinical and clinical information regarding Ad26.Mos4.HIV, Ad26.Mos.HIV, and Clade C gp140, see the latest version of the Investigator's Brochures and Addenda for Ad26.Mos4.HIV, Ad26.Mos.HIV, and Clade C gp140. 12,13

The term "sponsor" used throughout this document refers to the entities listed in the Contact Information page(s), which will be provided as a separate document.

Other organizations are also involved in this study, referred to in this protocol as "partners". For this protocol, the partners are the Division of Acquired Immune Deficiency Syndrome (DAIDS), Beth Israel Deaconess Medical Center (BIDMC), HIV Vaccine Trials Network (HVTN), International AIDS Vaccine Initiative (IAVI), and Military HIV Research Program (MHRP).

## 1.1. Background

### 1.1.1. Nonclinical Studies

## 1.1.1.1. Repetitive gp120/gp140 Vaccinations

In order to mimic the native trimeric structure of the HIV Env gp "spike" (glycoprotein 120 [gp120]/gp41) and induce native Envelope (Env)-reactive antibodies, trimeric gp140 proteins based on human Clade A and Clade C sequences were developed and found to induce significantly higher titers of potent neutralizing antibody (nAb) responses for a cross-clade set of tier 1 (Clades A, B, and C) and tier 2 (Clade C) viruses than the corresponding gp120 monomers in guinea pigs. <sup>18</sup> Although tier 1/2 pseudovirus neutralization is likely not predictive of neutralization capacity

against circulating HIV-1 viruses, the results suggest a broader and more avid Ab recognition of native HIV-1 Env.

## 1.1.1.2. Ad26/gp140 and Ad26/Ad35 Vaccinations

The protective efficacy of boosting with gp140 protein following priming with adenovirus serotype 26 (Ad26) vectors was evaluated in stringent simian immunodeficiency virus (SIV)- and simian-human immunodeficiency (SHIV)-challenge models in non-human primates (Part 1). Boosting with adjuvanted SIV<sub>MAC32H</sub> gp140 protein afforded 50% protection against the complete series of 6 heterologous, intrarectal challenges with SIV<sub>MAC251</sub> in animals that were primed with the Ad26 vector expressing SIV<sub>SME543</sub> Env/group-specific antigen (Gag)/polymerase (Pol) antigens, which was significantly higher than in animals that were similarly primed, but boosted with the corresponding Ad35 vector expressing SIV<sub>SME543</sub> Env/Gag/Pol antigens (17% protection). Binding Ab titers and Ab-dependent cellular phagocytosis (ADCP) responses correlated with protection against acquisition of infection. Cellular immune responses measured by interferon (IFN)γ enzyme-linked immunospot assay (ELISPOT) assays in response to SIV<sub>MAC239</sub> and SIV<sub>SME543</sub> Env/Gag/Pol peptide pools were also detected in all animals after vaccination. By intracellular cytokine staining (ICS) assays, gp140 boosting primarily expanded Env-specific IFNγ CD4<sup>+</sup> T-lymphocyte responses in the Ad26/gp140 group.

## 1.1.1.3. Ad26/Ad5 and Repetitive gp140 Vaccinations

A similar level of protection (40%) was seen after a series of 6 heterologous, intrarectal challenges with SHIV-SF162P3 in a first group of animals primed with Ad26 and Ad5<sub>HVR48</sub> vectors expressing mosaic, consensus, or natural Clade C HIV-1 Env/Gag/Pol antigens and boosted six times 2 years later with HIV-1 Clade C Env gp140 trimer (Part 2). A second group of animals received only the 6 gp140 immunizations. Although the gp140 vaccine afforded only minimal protection, 40% of Ad/gp140-vaccinated animals were completely protected against this challenge series. As for Section 1.1.1.2, binding Ab titers and ADCP responses correlated with protection against acquisition of infection.

#### 1.1.1.4. Tetravalent Ad26 Vaccinations

In ongoing clinical trials the trivalent Ad26.Mos.HIV viral vector is being used. But subsequent non-clinical data in rabbits have shown that the addition of a vector, expressing Mos2S Env protein, to Ad26.Mos1.Env increases the magnitude of binding Ab titers and neutralizing capacity for Tier 1A Clade C HIV virus in the absence of negative effects on Clade B neutralization capacity. Thus, addition of Ad26.Mos2S.Env to Ad26.Mos.HIV has the potential to substantially increase the breadth of humoral immune responses.

## 1.1.2. Clinical Studies

### 1.1.2.1. Prototypes and Similar Vaccines

There is considerable clinical experience with vaccines similar to Ad26.Mos.HIV and Clade C gp140 that demonstrated their class safety and tolerability.

## 1.1.2.1.1. Ad5 and Ad26 Vaccines

In 2 previous HIV-efficacy studies utilizing Ad5, a trend towards increased HIV-1 infection was observed in vaccine recipients as compared with placebo recipients.<sup>3,7</sup> The HVTN 502/Step (Merck Ad5) study showed no efficacy and a trend towards increased HIV-1 infections in vaccine recipients as compared with placebos. A significant but unexplained increase of HIV-1 infections was seen in vaccine recipients as compared with placebos in the subgroup of men who were baseline Ad5 seropositive and uncircumcised.<sup>3</sup> The HVTN 503/Phambili (Merck Ad5, MRKAd5) study was terminated and unblinded early, but follow-up of these individuals revealed increased HIV-1 infections in vaccine recipients as compared with placebo, particularly in men, which occurred after approximately 24 months of follow-up during the unblinded period. There was also differential dropout of high-risk placebos during this time period. Additionally, a third study, the HVTN 505 (NIH VRC deoxyribonucleic acid [DNA]/Ad5) study<sup>8</sup>, revealed no efficacy at the interim analysis. More HIV-1 infections were observed in vaccine recipients as compared with placebos in this study, including after the DNA prime and prior to the Ad5 boost, but these differences were not statistically meaningful. To clearly understand whether vaccine-associated increase of HIV-1 acquisition has occurred in one or more studies, a meta-analysis was recently conducted using up-to-date participant-level data from the 3 efficacy trials and three Phase 1-2 studies. The meta-analysis provides evidence for increased risk associated with the MRKAd5 vaccine overall and in various subgroups except circumcised and Ad5-negative men. While the meta-analysis does not provide a reliable basis for predicting whether rAd5-vectored vaccines for other pathogens or other rAd-vectored vaccines for HIV-1 would increase susceptibility to infection in HIV-1 at-risk populations, for large efficacy trials of such vaccines it provides a rationale for adding monitoring plans enabling detection of such increased susceptibility.

The mechanism for this possible increase in HIV-1 acquisition risk remains unclear, but a leading hypothesis involves activation of vector-specific CD4<sup>+</sup> T-lymphocytes at mucosal surfaces following Ad5 vaccination, potentially resulting in increased targets for HIV-1 infection. <sup>2,10</sup> This hypothesis has never been directly evaluated in humans with Ad5 vectors. Nevertheless, to assess the extent of mucosal CD4<sup>+</sup> T-cell activation with Ad26 vectors, a randomized, double-blinded, placebo-controlled clinical study (IPCAVD-003) was performed to determine whether vaccination of healthy human subjects with an Ad26 vector expressing HIV-1 Env would result in increased numbers or activation status of total or vector-specific CD4<sup>+</sup> T-lymphocytes in the colorectal mucosa. The findings of this study are reassuring in that this vector did not detectably increase the numbers or activation status of total or vector-specific CD4<sup>+</sup> T-cells in colorectal mucosa in humans.

The rationale to continue clinical development of Ad26 vector-based vaccines for HIV-1 is based on data showing that: (1) Ad26 is biologically substantially different than Ad5; (2) Ad26-based vaccines afford superior protective efficacy compared with Ad5-based vaccines against SIV<sub>MAC251</sub> challenges in rhesus monkeys; and (3) Ad26 did not increase the number or activation status of total or vector-specific CD4<sup>+</sup> T-lymphocytes at mucosal surfaces in humans following vaccination in a randomized, double-blind, placebo-controlled clinical study (IPCAVD-003).

In 3 Phase 1 studies (IPCAVD-001, IPCAVD-003, and IPCAVD-004)<sup>12</sup>, Ad26.ENVA.01, at intramuscular (IM) doses over the range  $10^9$  to  $10^{11}$  virus particles (vp), was found to induce Env-specific humoral and cell-mediated responses when given on up to 3 occasions to more than 200 healthy subjects. Ad26.ENVA.01 was generally well tolerated in these studies. An IM dose of  $5x10^{10}$  vp was found to provide the optimal balance of immunogenicity and reactogenicity. Therefore, this is the dose of Ad26.Mos.HIV chosen for further evaluation in this study.

In IPCAVD-003, 24 HIV-1 negative subjects were randomized 3:1 to receive a single vaccination with Ad26.ENVA.01 or placebo. Eight of the subjects were Ad26 seropositive at screening. The T-cell responses by IFNγ ELISPOT assays were slightly lower in the baseline Ad26-seropositive subjects; ICS and enzyme-linked immunosorbent assay (ELISA) responses proved comparable between subjects who were Ad26 seropositive and Ad26 seronegative at baseline, both in peripheral blood and in colorectal mucosa. In addition, systemic and mucosal responses persisted for at least 1 year in the majority of subjects after a single IM vaccine dose. These data suggest that the impact of baseline Ad26 nAbs, at the titers observed in that study, on the immunogenicity of this Ad26 vaccine is modest. Additionally, there were no consistent increases in Ad26-specific CD4<sup>+</sup> T-lymphocyte responses at mucosal surfaces following vaccination in either Ad26-seronegative or Ad26-seropositive subjects.

## 1.1.2.1.2. gp120 Vaccines

A monovalent gp120 protein (AIDSVAX B) was tested in 671 healthy subjects at 3 doses, 100, 300, and 600 mcg. <sup>11</sup> The 300-mcg dose was found to be the most effective, inducing a higher Ab response without significant side effects. In the Thai trial RV144<sup>20</sup>, the only vaccine study to date to demonstrate efficacy in prevention of acquisition of HIV, a bivalent gp120 protein (AIDSVAX B/E; 300-mcg dose) was used as a booster following priming with a recombinant canarypox vector (ALVAC-HIV) and afforded more than 30% protection from infection in the absence of either CD8<sup>+</sup> T-cells or nAb to primary HIV isolates. Therefore, a similar dose (250 mcg) of Clade C gp140 was chosen for evaluation in this study.

### 1.1.2.2. Current Studies

Currently, 2 first-in-human (FIH) studies in healthy HIV-uninfected subjects are evaluating safety/tolerability and immunogenicity of the following vaccines:

- Clade C gp140 (HIV-V-A003).
- Ad26.Mos.HIV, Modified Vaccinia Ankara (MVA)-Mosaic, and Clade C gp140 (HIV-V-A004; FIH for Ad26.Mos.HIV).

HIV-V-A003 is a single-center, randomized, placebo-controlled, double-blind, Phase 1 study to evaluate safety/tolerability, and immunogenicity of 2 dose levels (50 and 250 mcg) of Clade C gp140, with or without aluminum phosphate adjuvant, in healthy HIV-uninfected adult subjects. The blinded evaluation that was performed by the Data Monitoring Committee (DMC) at Week 6 (2 weeks after all of the 50 enrolled subjects had received their second and last vaccination) showed that Clade C gp140, administered as 50 or 250 mcg, with or without aluminum phosphate adjuvant, was well tolerated and no safety concerns were identified. All reported adverse events (AEs) were

of mild and moderate severity, there were no serious AEs (SAEs), withdrawals, or discontinuations. The DMC concurred with proceeding with the clinical development as planned and with administration of Clade C gp140 in HIV-V-A004.

HIV-V-A004 is a multi-center, randomized, parallel-group, placebo-controlled, double-blind Phase 1/2a study to evaluate safety/tolerability, and immunogenicity of various prime/boost regimens containing Ad26.Mos.HIV, MVA-Mosaic, and/or Clade C gp140 (with aluminum phosphate adjuvant) components in approximately 400 healthy HIV-uninfected adult subjects. As pre-specified in the protocol, enrollment was paused when approximately 10% of subjects had received their first injection (Ad26.Mos.HIV) and the Protocol Safety Review Team (PSRT) has reviewed blinded safety data of 2 weeks after this first injection of 39 subjects and on 18 June 2015 all members agreed that the study could resume enrollment. Most AEs were of mild and moderate severity. Three Grade 3 AEs were reported that were considered related to vaccination: headache, chills, and myalgia. There were no SAEs, withdrawals, or discontinuations. The independent Data Monitoring Committee (DMC) also reviewed the 2 week safety data after 30% of subjects had their first vaccination. They recommended continuing the study without modification. A 50 yearold male subject reported a severe allergic reaction having started 12 hours after first vaccination administration. Symptoms and signs mentioned by the subject included facial swelling, blurred vision, difficulty swallowing, and generalized rash of the face, extremities, and chest tightness. There was an emergency room (ER) visit (per ambulance) with administration of benadryl, but no hospitalization. Clinical observations by ER physician noted an alert and oriented person, with clinical signs of allergic reaction symptoms but with no lip/tongue/oropharyngeal/uvular swelling, normal findings of cardiovascular and respiratory system). Reaction was resolved within one day of onset. Concurrent diseases were drug abuse and bipolar disorder (not disclosed by subject to the investigator), with hallucinatory decompensation and chest pain one week after the severe allergic reaction. Following that, the subject was withdrawn from study due to non-compliance (history of drug abuse and non-reported psychiatric issues).

Study VAC89220HPX2008/HVTN 705 (hereafter abbreviated to HPX2008/HVTN 705) is an ongoing, multicenter, randomized, parallel-group, placebo-controlled, double-blind Phase 2b proof-of-concept efficacy study in approximately 2,600 HIV-uninfected sexually active women aged 18 to 35 years. The study is being conducted in approximately 25 sites, with the majority of these throughout South Africa. Study participants were selected from populations at high risk of acquiring HIV infection in southern Africa settings with overall moderate to high HIV incidence. The predominant circulating HIV-1 is a Clade C virus. The study is investigating the preventive vaccine efficacy, safety, and tolerability of a heterologous regimen with 4 vaccinations consisting of tetravalent Ad26.Mos4.HIV and aluminum phosphate-adjuvanted Clade C gp140, with vaccinations at Months 0, 3, 6, and 12. The primary analysis recently demonstrated that the vaccine regimen did not provide statistically significant protection against HIV infection. The vaccine efficacy over Months 7 to 24 in the per-protocol cohort did not differ significantly from zero, with a point estimate (95% confidence interval) of 25% (-10% to 49%). The regimen did not cause harm and was generally well-tolerated. 15

## 1.2. Overall Rationale for the Study

The proposed clinical study will be an FIH evaluation (for Ad26.Mos4.HIV) in healthy HIV-uninfected subjects to evaluate the safety/tolerability and immunogenicity of a regimen including trivalent Ad26.Mos4.HIV and a regimen including tetravalent Ad26.Mos4.HIV. Better Clade C responses are to be expected with the tetravalent Ad26.Mos4.HIV compared to the trivalent Ad26.Mos.HIV.

To assess the durability of the immune responses, an optional Long-term Extension (LTE) phase of approximately 3 years was introduced for subjects randomized to Group 2A, who have received all 4 vaccinations and are negative for HIV infection at the end of the main study. The vaccination regimen of Group 2A (including Ad26.Mos4.HIV and Clade C gp140) forms the basis for the regimens that will likely be evaluated in future studies.

Based on the currently available durability data of immune responses<sup>22,23</sup> the sponsor aims to evaluate the persistence of these responses over 5.5 years after the last (4th) vaccination. Therefore, an optional 2-year extension of the 3-year LTE phase was introduced with protocol amendment 3.

Recent results of study HPX2008/HVTN 705 demonstrated that the vaccine regimen used in HPX2008 (which is the same regimen being used in HPX2004) did not provide statistically significant protection against HIV infection (see Section 1.1.2.2). Therefore, with protocol amendment 5, the 2-year LTE extension was shortened to 1 year (corresponding to a follow-up of approximately 4,5 years after the last [4<sup>th</sup>] vaccination).

## 2. OBJECTIVES, ENDPOINTS, AND HYPOTHESIS

## 2.1. Objectives and Endpoints

## 2.1.1. Objectives

### **Primary Objectives**

The primary objectives are to assess:

- Safety/tolerability of the 2 different vaccine regimens of priming with trivalent Ad26.Mos.HIV and boosting with trivalent Ad26.Mos.HIV and Clade C gp140 plus adjuvant or priming with tetravalent Ad26.Mos4.HIV and boosting with Ad26.Mos4.HIV and Clade C gp140 plus adjuvant.
- Env-binding Ab responses of the 2 different vaccine regimens.

## **Secondary Objectives**

The secondary objectives are to assess:

- Neutralizing Ab responses, Ab functionality (as assessed by phagocytosis), and Ab isotyping.
- T-cell responses.

## **Exploratory Objectives**

The exploratory objectives are:

- Ab functionality (other than phagocytosis).
- Ab Fc characterization.
- T-cell and Ab epitope mapping.
- Gene expression of peripheral blood mononuclear cells (PBMCs).
- B-cell responses.
- Immune responses against the viral vector.
- The social impact of participation in an HIV-vaccine study for subjects via a social impact questionnaire.
- To explore durability of the immune responses to the vaccine regimen in the groups selected for the optional LTE phase.

## 2.1.2. Endpoints

## **Primary Endpoints**

• AEs throughout the study

Local and systemic solicited AEs for 7 days post-vaccination.

AEs for 28 days after each vaccination.

Discontinuations from vaccination/from study due to AEs.

SAEs and AEs of special interest (AESIs) during the course of the study, including the optional LTE phase.

• Env-specific binding Abs (titers and breadth).

## **Secondary Endpoints**

- Env-specific nAbs (titers and breadth) (for Tier 1 and Tier 2 viruses; note: Tier 2 will be assessed only if Tier 1 shows positive results).
- Env-specific functional Abs (phagocytosis score and breadth).
- Env-specific binding Ab isotypes (IgA, IgG1-4) (titers and breadth).
- IFNy PBMC responders to mosaic peptide pools of Env/Gag/Pol and PTE.
- CD4<sup>+</sup> and CD8<sup>+</sup> T-cell functionality (% cells producing ia, IFNγ, IL-2, IL-4, TNFα).
- T-cell development with emphasis on follicular helper T-cells and memory differentiation.
- Available samples from time points after last vaccination until the final main study visit at Week 72 will be used for determination of durability of the immune responses.

## **Exploratory Endpoints**

• Ab functionality evaluation (by other than phagocytosis).

- Ab Fc (sub)typing.
- Epitope mapping of Ab to Env and T-cell responses to Gag/Pol/Env and PTE.
- Regulation of genes (clusters) that predict specific immune responses and human leukocyte antigen (HLA) typing.
- Ab-producing B-cells and characterization of B-cell memory development.
- Ad26 nAbs (titer).
- Available samples from time points during the optional LTE phase will be used for determination of long-term durability of the immune responses.

## 2.2. Hypothesis

No formal statistical hypothesis will be tested. This study will evaluate whether 2 vaccine regimens, priming with Ad26.Mos.HIV or Ad26.Mos4.HIV and boosting with Clade C gp140 together with Ad26.Mos.HIV or Ad26.Mos4.HIV, are safe, well-tolerated, and immunogenic, providing broad, functional, and durable humoral and cellular responses.

## 3. STUDY DESIGN AND RATIONALE

## 3.1. Overview of Study Design

This is a randomized, double-blind, placebo-controlled, parallel, interventional, Phase 1/2a study in healthy HIV-uninfected adult men and women aged 18 through 50 years. A target of 198 subjects will participate in this study, randomized into one of 4 subgroups: 55 subjects will receive vaccination with Ad26.Mos.HIV and Clade C gp140 in Subgroup 1A, 11 subjects will receive placebo in Subgroup 1B, 110 subjects will receive vaccination with Ad26.Mos4.HIV and Clade C gp140 in subgroup 2A and 22 subjects will receive placebo in Subgroup 2B. Randomization will be stratified by region. Subjects will be enrolled regardless of their baseline Ad26 seropositivity. Subjects will receive study vaccine or placebo according to the time points in Table 1.

The main study will be conducted in 3 phases: a 4-week screening period (with 2 extra weeks to allow for start of hormonal contraception for female subjects or female partners of male subjects); a 48-week vaccination period during which subjects will be vaccinated at baseline (Week 0) and Weeks 12, 24, and 48; and a follow-up period to the final main study visit at Week 72. An optional LTE phase (approximately 3 or 4 years after Week 72 depending on the length of follow-up which subjects consent to) will be performed for subjects randomized to Group 2A, who have received all 4 vaccinations and are negative for HIV infection at Week 72. The vaccination regimen of Group 2A (including Ad26.Mos4.HIV and Clade C gp140) forms the basis for the regimens that will likely be evaluated in future studies. The duration of the subject's participation will be approximately 76 weeks for subjects not participating in the optional LTE phase and approximately 220 or 268 weeks for subjects participating in the optional LTE phase (approximately 3 or 4 years after the end of the main study, respectively).

After vaccination, subjects will remain under observation at the study site for at least 30 minutes for presence of any acute reactions and solicited events. In addition, subjects will record solicited

local (at injection site) and systemic events as described in Section 9.1.1. See Section 12.1.3 for grading of severity of solicited AEs. Further safety evaluations will include monitoring of AEs, physical examinations, vital sign measurements, clinical laboratory tests, and pregnancy testing until Week 72. Blood samples will be taken at specific clinic visits to assess immune responses. Subjects will complete a social impact questionnaire at specific clinic visits. For details see Attachment 4. A PSRT and Data Review Committee (DRC) will be commissioned for this study. See Sections 11.7 and 11.8 for details.

For details on Analysis Time Points, see Section 11.6.

The COVID-19 Appendix in Section 18 provides guidance to investigators for managing study-related procedures during the COVID-19 pandemic.

| Table 1: | Study Design VAC89220HPX2004 | | | | | |
|---|---|---|---|---|---|---|
| Group | Subgroup | N | Week 0 | Week 12 | Week 24 | Week 48 |
| Group 1 | A | | Ad26.Mos.HIV | | Ad26.Mos.HIV | Ad26.Mos.HIV |
| | | 55 | | Ad26.Mos.HIV | Clade C gp140<br>(250 mcg +<br>adjuvant) <sup>a</sup> | Clade C gp140<br>(250 mcg +<br>adjuvant) <sup>a</sup> |
| | В | 11 | Placebo | Placebo | Placebo<br>+ | Placebo<br>+ |
| | | | | | Placebo | Placebo |
| Group 2 | A <sup>b</sup> | 110 | Ad26.Mos4.HIV | | Ad26.Mos4.HIV | Ad26.Mos4.HIV |
| | | | | | + | + |
| | | | | Ad26.Mos4.HIV | Clade C gp140<br>(250 mcg +<br>adjuvant) <sup>a</sup> | Clade C gp140<br>(250 mcg +<br>adjuvant) <sup>a</sup> |
| | В | 22 | Placebo | | Placebo | Placebo |
| | | | | Placebo | + | + |
| | | | | | Placebo | Placebo |

<sup>&</sup>lt;sup>a</sup>250 mcg refers to total protein content; sterile aluminum phosphate suspension will be used as adjuvant. Aluminum content will be 0.425 mg/0.5 mL dose.

## 3.2. Study Design Rationale

#### Vaccines and Dose Selection Rationale

The rationale behind selection of study vaccines and doses is described in Section 1.1.

### Blinding, Control, Study Phase/Periods, Treatment Groups

A placebo control will be used to establish the frequency and magnitude of changes in clinical endpoints that may occur in the absence of active treatment. Randomization will be used to

<sup>&</sup>lt;sup>b</sup>An optional LTE phase (approximately 3 or 4 years after Week 72 depending on the length of follow-up which subjects consent to) will be performed for subjects randomized to Group 2A, who have received all 4 vaccinations and are negative for HIV infection at Week 72.

minimize bias in the assignment of subjects to treatment groups, to increase the likelihood that known and unknown subject attributes (eg, demographic and baseline characteristics) are evenly balanced across treatment groups, and to enhance the validity of statistical comparisons across treatment groups. Blinded treatment will be used to reduce potential bias during data collection and evaluation of clinical endpoints.

## 4. SUBJECT POPULATION

Screening for eligible subjects will be performed within 4 weeks (with 2 extra weeks to allow for start of hormonal contraception for female subjects or female partners of male subjects) before the first administration of study vaccine/placebo at Week 0.

The inclusion and exclusion criteria for enrolling subjects in this study are described in the following 2 subsections. If there is a question about the inclusion or exclusion criteria below, the investigator must consult with the appropriate sponsor representative and resolve any issues before enrolling a subject in the study. Waivers are not allowed.

For a discussion of the statistical considerations of subject selection see Section 11.3.

## 4.1. Inclusion Criteria for the Main Study

Each potential subject must satisfy all of the following criteria to be enrolled in the study.

- 1. Each subject must sign an informed consent form (ICF) indicating that he or she understands the purpose of and procedures required for the study and is voluntarily willing to participate in the study.
- 2. Subjects are  $\geq 18$  to  $\leq 50$  years old on the day of signing the ICF.
- 3. Subject must be healthy on the basis of physical examination, medical history, and vital signs measurement performed at screening.
- 4. Subjects must meet following laboratory criteria prior to randomization\*:
  - a) Hemoglobin: Women  $\geq 10.5$  g/dL; Men  $\geq 11.0$  g/dL
  - b) White cell count: 2,500 to 11,000 cells/mm<sup>3</sup>, inclusive
  - c) Absolute neutrophil count: >1,000 cells/mm<sup>3</sup>
  - d) Platelets: 125,000 to 450,000 per mm<sup>3</sup>, inclusive
  - e) Urinalysis: protein <1+, blood <1+ (men) and <2+ (women), and glucose negative
  - f) Alanine aminotransferase/aspartate aminotransferase: <1.25x upper limit of normal (ULN)
  - g) Creatinine: <1.1x ULN

<sup>\*</sup>If laboratory screening tests are out of range, repeat of screening tests is permitted once.

- 5. Subjects are negative for HIV infection at screening<sup>a</sup>.
- 6. All female subjects of childbearing potential must have a negative serum ( $\beta$ -human chorionic gonadotropin [ $\beta$ -hCG]) at the screening visit, and a negative urine pregnancy test pre-dose on Day 1<sup>b</sup>.
- 7. Contraceptive requirements for heterosexually active female subjects (from 28 days prior first vaccination up until 3 months after last vaccination)<sup>c</sup>:
  - a) If not of childbearing potential: postmenopausal (>45 years of age with amenorrhea for at least 2 years, or any age with amenorrhea for at least 6 months and a serum follicle stimulating hormone [FSH] level >40 IU/L) or surgically sterile: no additional contraception required.
  - b) If of child-bearing potential, but has a vasectomized partner (after vasectomy: sperm count below the limit of detection if procedure occurred <1 year ago<sup>d</sup>): no additional contraception required.
  - c) If of child-bearing potential, but has a non-vasectomized partner, or partner had a positive sperm count after a vasectomy procedure of <1 year ago<sup>d</sup>, should be practicing an acceptable effective method of contraception. Acceptable methods for this study include:
    - Hormonal contraception,
    - Intrauterine device (IUD),
    - Intrauterine hormone-releasing system (IUS),
    - Male or female condom with or without spermicide,
    - Cap, diaphragm or sponge with vaginal spermicide, or
    - Sexual abstinence \*

\*Sexual abstinence is considered an effective method **only** if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study vaccine. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the study and the preferred and usual lifestyle of the subject.

Women who are not heterosexually active at screening, but become sexually active during the study must agree to utilize an effective method of birth control as mentioned above.

8. Contraceptive requirements for heterosexually active male subjects (from day of first vaccination until 3 months after last vaccination):

<sup>&</sup>lt;sup>a</sup> If possible, the site should select an assay that is US FDA-approved

<sup>&</sup>lt;sup>b</sup> Note: negative urine pregnancy also required prior to the second, third, and fourth vaccinations

c Verbal assurance should be given that adequate birth control measures have been followed for 28 days prior to first vaccination

<sup>&</sup>lt;sup>d</sup> Based on verbal confirmation

- a) If male subject had a vasectomy (after vasectomy: sperm count below the limit of detection if procedure occurred <1 year ago<sup>d</sup>): no additional contraception required.
- b) If male subject did not have a vasectomy or had a positive sperm count after a vasectomy procedure of <1 year ago<sup>d</sup>: contraceptive methods will depend on child-bearing potential of female partner: same criteria to be followed as for female subjects in inclusion criterion 7.
- 9. A woman must agree not to donate eggs (ova, oocytes) for the purpose of assisted reproduction after the first dose until 3 months after receiving the last dose of study vaccine/placebo. A man must agree not to donate sperm after the first dose until 3 months after receiving the last dose of study vaccine/placebo.
- 10. Subjects are willing/able to adhere to the prohibitions and restrictions specified in the protocol and study procedures.
- 11. Subjects are amenable to HIV-risk reduction counseling and committed to maintaining behavior consistent with low risk of HIV exposure through the last required protocol clinic visit.
- 12. Subjects are assessed by the clinic staff as being at low risk for HIV infection (see Attachment 2).
- 13. Passed the Test Of Understanding (TOU). The TOU must be completed by all subjects, as the first assessment after signing of the ICF.

# 4.2. Exclusion Criteria for the Main Study

Any potential subject who meets any of the following criteria will be excluded from participating in the study:

- 1. Subject has chronic hepatitis B (measured by hepatitis B surface antigen test) or active hepatitis C (measured by hepatitis C virus [HCV] Ab test; if positive, HCV ribonucleic acid [RNA] PCR test will be used to confirm active versus past HCV infection), active syphilis infection, chlamydia, gonorrhea, or trichomonas<sup>e</sup>. Active syphilis documented by serology unless positive serology is due to past treated infection.
- 2. In the 12 months prior to randomization, subject has a history of newly acquired herpes simplex virus type 2, syphilis, gonorrhea, non-gonococcal urethritis, chlamydia, pelvic inflammatory disease, trichomonas, mucopurulent cervicitis, epididymitis, proctitis, lymphogranulomavenereum, chancroid, or hepatitis B.
- 3. Subject has any condition, including any clinically significant acute or chronic medical condition, for which, in the opinion of the investigator, participation would not be in the best interest of the subject (eg, compromise the well-being) or that could prevent, limit, or

\_

<sup>&</sup>lt;sup>e</sup> Trichomonas testing will only be performed for female subjects

- confound the protocol-specified assessments. In case of questions, the investigator is encouraged to contact the study responsible physician.
- 4. Subject has had major surgery (eg, requiring general anesthesia) within the 4 weeks before screening, or will not have fully recovered from surgery, or has surgery planned through the course of the study.
  - Note: Subjects with planned surgical procedures to be conducted under local anesthesia may participate.
- 5. Subject has had a thyroidectomy or active thyroid disease requiring medication during the last 12 months (not excluded: a stable thyroid supplementation).
- 6. Subject has had major psychiatric illness and/or substance abuse problems during the past 12 months (including hospitalization or periods of work disability) that in the opinion of the investigator would preclude participation.
- 7. Subject is a woman who is pregnant, or breast-feeding, or planning to become pregnant while enrolled in this study, or within 3 months after the last dose of vaccine/placebo.
- 8. Subject is a man who plans to father a child while enrolled in this study, or within 3 months after the last dose of vaccine/placebo.
- 9. Subject has been in receipt of any licensed vaccine within 14 days prior to the first dose of study vaccine/placebo, plans to receive within 14 days after the first study vaccination, or plans to receive within 14 days before or after the second, third or fourth vaccination.
- 10. Subject has used experimental therapeutic drugs within 30 days of randomization. For experimental vaccines see exclusion criterion 11.
- 11. Subject is a recipient of a prophylactic or therapeutic HIV vaccine candidate at any time, or a recipient of other experimental vaccine(s) within the last 12 months prior to the Day 1 visit (Vaccination 1). For subjects who received an experimental vaccine (except HIV vaccine) more than 12 months prior to the Day 1 visit (Vaccination 1), documentation of the identity of the experimental vaccine must be provided to the sponsor, who will determine eligibility on a case-by-case basis.
  - Exceptions: Subjects can be included where the vaccine received was subsequently licensed (see exclusion criterion 9). Subjects with proof of having received only a placebo vaccine can also be included.
- 12. Subject is currently in, or plans participation in, another interventional study during the study period. Participation in an observational study is allowed with prior approval of the sponsor.
- 13. Subject has been in receipt of blood or immunoglobulin products in the past 3 months.
- 14. Subject has known allergies, hypersensitivity, or intolerance to vaccines or its excipients 12,13.

- 15. Subject has a history of chronic urticaria (recurrent hives) or a history of chronic or recurrent eczema and/or atopic dermatitis that requires oral/parenteral immunomodulators/immunosuppressors.
- 16. Subject has chronic or recurrent use of immunomodulators/suppressors, eg, cancer chemotherapeutic agents, and oral or parenteral corticosteroids. Inhaled, ocular, and topical steroids are allowed.
- 17. Subject who cannot communicate reliably with the investigator.
- 18. Subject is an employee of the investigator or study site, with direct involvement in the proposed study or other studies under the direction of that investigator or study site, as well as family members of the employees or the investigator.

**NOTE:** Investigators should ensure that all study enrollment criteria have been met during the screening period. If a subject's clinical status changes (including any available laboratory results or receipt of additional medical records) after screening but before the first dose of study vaccine is given such that he or she no longer meets all eligibility criteria, then the subject should be excluded from participation in the study. Section 17.4 describes the required documentation to support meeting the enrollment criteria.

### 4.3. Prohibitions and Restrictions

Potential subjects must be willing and able to adhere to the following prohibitions and restrictions during the course of the study to be eligible for participation:

- 1. Agree to follow the contraceptive requirements as noted in Section 4.1 during the main study.
- 2. Following vaccination subjects may be excluded from donating blood products due to induced vaccine seropositivity (see Section 9.4.3) for as long as VISP persists.
- 3. Male subjects must agree not to donate sperm from the first administration of study vaccine/placebo until 3 months after the last dose of study vaccine/placebo.
- 4. Female subjects must agree not to donate eggs (ova, oocytes) for the purpose of assisted reproduction until 3 months after the last dose of study vaccine/placebo.
- 5. Use of any experimental medication (including experimental vaccines other than the study vaccine) during the main study is disallowed. Vaccination with any licensed vaccine within 14 days prior to or after any of the study vaccinations is disallowed. However, if a vaccine is indicated in a post-exposure setting (eg, rabies or tetanus), it must take priority over the study vaccine. Subjects who enter the optional LTE phase are allowed to use any experimental medication during the optional LTE phase, except for prophylactic or therapeutic HIV vaccine candidates which are disallowed and experimental immunomodulators/suppressors which need prior sponsor approval.
- 6. Chronic or recurrent use of immunomodulators/suppressors, eg, cancer chemotherapeutic agents, and oral or parenteral corticosteroids is prohibited during the main study. During the optional LTE phase, use of these medications is discouraged, except when required by
the medical condition of the subject, and each use should be reported during clinical visits. Inhaled, ocular, and topical steroids are allowed (see Section 8).

7. Concurrent participation in another clinical study without prior sponsor approval is disallowed during the main study. Subjects who enter the optional LTE phase are allowed to participate in another clinical study, except for studies with prophylactic or therapeutic HIV vaccine candidates which are disallowed and studies with experimental immunomodulators/suppressors which need prior sponsor approval.

# 4.4. Inclusion and Exclusion Criteria for the Optional Long-term Extension Phase

Each potential subject must satisfy all of the following inclusion criteria to be enrolled in the optional LTE phase of the study upon completion of the final main study visit at Week 72. For the optional 2-year extension of the LTE phase, there are no inclusion criteria, except for the signing of the ICF appendix in criterion 1.

- 1. Each subject must sign an ICF appendix for the optional 3-year LTE phase indicating that he or she understands the purpose of and procedures required for the optional LTE phase and is voluntarily willing to participate in the optional LTE phase of the study. Subjects willing to participate in the optional 2-year extension of the LTE phase will need to sign the ICF appendix for the 2-year extension at Visit 23.
- 2. Subject must be randomized to Group 2A of the main study.
  - Note: Upon sponsor unblinding at the Week 28 analysis, subjects randomized to Group 2A who have received all 4 vaccinations, will be asked to participate in the optional LTE phase and sign the ICF appendix for the optional LTE phase at Week 72. Subjects who attend their Week 72 visit prior to the sponsor's unblinding at the Week 28 analysis, will be enrolled in the optional LTE phase if they consent and sign the ICF appendix for the optional LTE phase and meet the eligibility criteria for the optional LTE phase. When the Week 28 sponsor unblinding subsequently occurs, subjects that started the optional LTE phase but turn out not to be in Group 2A of the main study will be withdrawn from the optional LTE phase.
- 3. Subject must have received all 4 vaccinations of the main study.
- 4. Subject must be negative for HIV infection at the final main study visit at Week 72.
- 5. Subject must be willing/able to adhere to the prohibitions and restrictions for the optional LTE phase, as specified in the protocol and study procedures.

Any potential subject who meets any of the following exclusion criteria at the end of the main study will be excluded from participating in the optional LTE phase of the study. For the optional 2-year extension of the LTE phase, there are no exclusion criteria.

- 1. Subject has any condition for which, in the opinion of the investigator, participation would not be in the best interest of the subject (eg, compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments.
- 2. Subject is planning to participate in an interventional study during the optional LTE phase, concerning a prophylactic or therapeutic HIV vaccine candidate.
- 3. Subject is planning to participate in an interventional study during the optional LTE phase, concerning an experimental immunomodulator/suppressor that is not allowed per the sponsor. Documentation of the identity of the experimental immunomodulator/suppressor must be provided to the sponsor, who will determine eligibility on a case-by-case basis.

## 5. TREATMENT ALLOCATION AND BLINDING

#### **Treatment Allocation**

## **Procedures for Randomization**

Central randomization will be implemented in this study. Subjects will be randomly assigned to one of 2 treatment groups and to one of 2 subgroups within each group based on a computer-generated randomization schedule prepared before the study by or under the supervision of the sponsor. The randomization will be evaluated by using randomly permuted blocks and stratified by region.

The interactive web response system (IWRS) will assign a unique treatment code, which will dictate the treatment assignment and matching study vaccine for the subject. The requestor must use his or her own user identification and personal identification number when contacting the IWRS, and will then give the relevant subject details to uniquely identify the subject.

#### **Blinding**

The subjects, study-site personnel (except for those with primary responsibility for study vaccine preparation and dispensing), and investigator will be blinded to study vaccine allocation until Week 72, with the exception of the partial unblinding for the start of the optional LTE phase (see below). The sponsor will be blinded to study vaccine allocation until the Week 28 analysis (see Section 11.6).

An interim immunogenicity analysis will be performed once approximately 60 subjects have completed the Week 16 visit and will be unblinded at the group level, but not at the subject level. Study-site personnel (except for those with primary responsibility for study vaccine preparation and dispensing), the sponsor (except for programming, statistics, clinical, and clinical immunology personnel involved in the analysis, and the sponsor committee involved in making future decisions for the program) and subjects will remain blinded to study vaccine allocation.

The pharmacist with primary responsibility for vaccine preparation (see Section 14.3) will not be blinded to the study vaccine. In order to preserve blinding, he/she will place an overlay on the syringes.

The investigator will not be provided with randomization codes. The codes will be maintained within the IWRS, which has the functionality to allow the investigator to break the blind for an individual subject.

Data that may potentially unblind the treatment assignment will be handled with special care to ensure that the integrity of the blind is maintained and the potential for bias is minimized. This can include making special provisions, such as segregating the data in question from view by the investigators, clinical team, or others as appropriate until the time of database lock and unblinding.

Under normal circumstances, the blind should not be broken by the investigator until the Week 72 electronic Data Capture (eDC) database is locked for the subjects, study-site personnel (except for those with primary responsibility for study vaccine preparation and dispensing), and investigator. However, for the purpose of the optional LTE phase, the investigator, the study-site personnel, and the subject will be informed if the subject qualifies for the optional LTE phase (ie, if the subject is randomized to Group 2A) when the subject reaches the Week 72 visit, or as soon as possible following Week 72 upon sponsor unblinding at the Week 28 analysis. This will result in the partial unblinding of the investigator, the study-site personnel, and the subjects as only those subjects randomized to Group 2A qualify for the optional LTE phase. Subjects randomized to Groups 1A, 1B and 2B will not be informed of their treatment assignment until after the Week 72 eDC database lock.

Otherwise, the blind should be broken only if specific emergency treatment/course of action would be dictated by knowing the treatment status of the subject. In such cases, the investigator may in an emergency determine the identity of the treatment by contacting the IWRS. It is recommended that the investigator contacts the sponsor or its designee if possible to discuss the particular situation, before breaking the blind. Telephone contact with the sponsor or its designee will be available 24 hours per day, 7 days per week. In the event the blind is broken, the sponsor must be informed as soon as possible. The date and reason for the unblinding must be documented by the IWRS, in the appropriate section of the Case Report Form (CRF), and in the source document. The documentation received from the IWRS indicating the code break must be retained with the subject's source documents in a secure manner.

Subjects who have had their treatment assignment unblinded should continue to return for safety and immunogenicity evaluations, but will be withdrawn from study vaccine administration (see Section 10.2).

In general, randomization codes will be disclosed fully only if the study is completed and the clinical eDC database is closed. However, if an interim analysis is specified, the randomization codes and, if required, the translation of randomization codes into treatment and control groups will be disclosed to those authorized and only for those subjects included in the interim analysis. See Section 11.6.

## 6. DOSAGE AND ADMINISTRATION

Each subject will receive study vaccine/placebo at 4 time points according to randomization, on Day 1 and Weeks 12, 24, and 48, administered by IM injection into the deltoid. For visits with

only one injection (ie, at Weeks 0 and 12), preferably the deltoid of the non-dominant upper arm is used. When 2 injections are to be given at one visit (ie, at Weeks 24 and 48), it is required to use a different deltoid for each injection. Exceptions on injection site are allowed only if medically indicated.

For information on vaccination windows, see Section 9.1.2. If a subject cannot be vaccinated within the allowed window, then that vaccination should not be administered. However, if the window is missed due to a study pause (see Section 11.9), vaccination will be assessed on a case-by-case basis, upon discussion between sponsor and investigator. If a subject misses more than one study vaccination, he/she will be withdrawn from further study vaccination (see Section 10.4). Study vaccines are as follows:

### Ad26.Mos4.HIV:

Total dose is  $5x10^{10}$  vp per 0.5 mL injection

Ad26.Mos.HIV:

Total dose is  $5x10^{10}$  vp per 0.5 mL injection

• Clade C gp140:

Clade C gp140 with 250 mcg total protein, mixed with aluminum phosphate adjuvant (0.425 mg aluminum) at the pharmacy, per 0.5 mL injection

Placebo:

0.9% saline, 0.5 mL injection

#### 7. TREATMENT COMPLIANCE

Subjects will receive doses of study vaccine/placebo at 4 time points administered by IM injection by qualified study-site personnel at the study sites.

The date and time of each study vaccine administration will be recorded in the CRF.

#### 8. PRESTUDY AND CONCOMITANT THERAPY

Prestudy therapies administered up to 30 days before the screening visit will be recorded in the CRF at screening. In case a subject received an experimental vaccine more than 12 months prior to the Day 1 visit (Vaccination 1) and is determined to be eligible, administration of this experimental vaccine will be recorded in the CRF.

Concomitant therapies must be recorded in the CRF throughout the study from the signing of the ICF to the final main study visit at Week 72. Beyond Week 72 (during the optional LTE phase), only concomitant therapies given in conjunction with an SAE will be collected, as well as any chronic or recurrent use of immunomodulators/suppressors and oral or parenteral corticosteroids (see below).

Use of any experimental medication (including experimental vaccines other than the study vaccine) during the main study is disallowed. Vaccination with any licensed vaccine within the

14 days prior to or after any dose of study vaccine/placebo is prohibited. However, if a vaccine is indicated in a post-exposure setting (eg, rabies or tetanus), it must take priority over the study vaccine. Subjects who enter the optional LTE phase are allowed to use any experimental medication during the optional LTE phase, except for prophylactic or therapeutic HIV vaccine candidates which are disallowed and experimental immunomodulators/suppressors which would need prior sponsor approval.

Study subjects can receive medications, such as acetaminophen, non-steroidal anti-inflammatory drugs, or antihistamines as needed, although their use must be documented and use of these medications as routine prophylaxis prior to study vaccination is discouraged.

Chronic or recurrent use of:

- Immunomodulators/suppressors, eg, cancer chemotherapeutic agents
- Oral or parenteral corticosteroids, eg, glucocorticoids

is an exclusion criterion (Section 4.2), and these medications are prohibited during the main study. During the optional LTE phase, use of these medications is discouraged, except when required by the medical condition of the subject, and each use should be reported during clinical visits. Ocular and topical steroids are allowed, as well as inhaled steroids for the treatment of pulmonary conditions.

The sponsor must be notified in advance (or as soon as possible thereafter) of any instances in which prohibited therapies are administered.

### 9. STUDY EVALUATIONS

## 9.1. Study Procedures

## 9.1.1. Overview

The Time and Events Schedule summarizes the frequency and timing of safety and immunogenicity measurements applicable to the main study and the optional LTE phase.<sup>f</sup>

Evaluation of the safety/tolerability and immunogenicity of the vaccine regimens will include laboratory assessments, physical assessment by clinical staff, and subject reports on signs and

\_

f The timing and events outlined in the Time and Events Schedule are subject to modification in the event of emergencies (possibly affecting a site, a region, a country or world-wide). Instructions on specific modifications will depend on the particular situation and could vary by site. At a minimum, all efforts will be made to interact with a participant via telemedicine at the time of a protocol-defined visit. Whereas the implementation of alternative processes should be consistent with the protocol to the extent possible, it may, therefore, not be possible to conduct all assessments at the defined time (or within the designated window). The health and safety of the participant and site staff will be the driving factor in such decision making along with government and/or institutional guidances/mandates. Any such deviations and the reason for any contingency measures implemented, would clearly be described in the study report and IRB/EC and HA notification would be made if required.

symptoms following vaccinations. Additional study visits may be required if in the investigator's opinion, further clinical or laboratory evaluation is needed.

Subjects will be provided with a thermometer, ruler, and subject diary to measure and record body temperature and solicited local (at injection site) and systemic events.

The diary includes instructions how to capture the data and grading scales to assess severity of the symptoms. The study staff is responsible for providing appropriate training to the subject to avoid missing or incorrect data. The diary card will be reviewed by the study personnel at visits indicated on the Time and Events Schedule.

From screening to the final main study visit at Week 72, the total blood volume to be collected from each subject will be approximately 1,200 mL. The total blood volume to be collected during the optional LTE phase (Group 2A only) will be approximately 470 mL over a 3-year period or 628 mL over a 4-year period for subjects who consent to the optional 1-year extension of the optional LTE phase. The total blood volume to be collected is considered to be within the United States (US) Department of Health and Human Services (HHS) Office for Human Research Protections (OHRP), and US FDA guidelines of 550 mL in any 8-week period. Daily volumes for humoral immunogenicity testing will be approximately 20 mL/visit and for cellular immunogenicity testing approximately 50-102 mL/visit during the main study and 50 mL/visit during the optional LTE phase.

Repeat or unscheduled samples may be taken for safety reasons or for technical issues with the samples.

Subjects who are temporarily not able to attend the per protocol visits at their clinical site due to travel (eg, vacation, business travel) may visit any other clinical site participating in this clinical study for non-vaccination visits. Please refer to the Study Procedures Manual for the guest visit procedure details.

## 9.1.2. Visit Windows

The maximum screening period is 4 weeks, with the exception of female subjects or female partners of male subjects starting hormonal contraception. In this case, the maximum screening period is 6 weeks.

For the study visits, following windows will be allowed as indicated:

- Visit 3: Day  $8 \pm 1$  day
- Visit 4: Day  $15 \pm 5$  days
- Visit 5: Day  $29 \pm 5$  days
- Visit 6: Day 85 -1 week, +3 weeks (second vaccination)
- Visit 7\*: Visit 6 + 14 days (Day 99)  $\pm 5$  days

- Visit 8\*: Visit 6 + 28 days (Day 113)  $\pm 5$  days
- Visit 9: Day 169 -1 week, +3 weeks (third vaccination)
- Visit  $10^*$ : Visit 9 + 14 days (Day 183)  $\pm 5$  days
- Visit 11\*: Visit 9 + 28 days (Day 197)  $\pm$  5 days
- Visit 12: Day  $253 \pm 5$  days
- Visit 13: Day 337 -1 week, +3 weeks (fourth vaccination)
- Visit 14\*: Visit 13 + 14 days (Day 351)  $\pm$  5 days
- Visit 15\*: Visit 13 + 28 days (Day 365)  $\pm$  5 days
- Visit 16: Day  $421 \pm 3$  weeks
- Visit 17: Day  $505 \pm 3$  weeks
- Visit 18 to 22 inclusive and Visit 24-25 inclusive: Days 673, 841, 1009, 1177, 1345, 1681, 1849, ± 4 weeks
- Visit 23: 1513 -4 weeks/+2 months

\*If a subject is not vaccinated on the given day of vaccination, the timings of the visits 2 and 4 weeks post-vaccination (see Time and Events Schedule) will be determined relative to the actual day of vaccination.

If a subject cannot be vaccinated within the allowed window, then that vaccination should not be administered. However, if the window is missed due to a study pause (see Section 11.9), vaccination will be assessed on a case-by-case basis upon discussion between investigator and sponsor. If a subject misses more than 1 study vaccination, he/she will be withdrawn from further study vaccination.

For the LTE phase (from Week 72 onwards): If a visit can't be scheduled within the allowed window, it will be assessed on a case-by-case basis upon discussion between investigator and sponsor whether this visit can still be performed.

In the event of emergencies (possibly affecting a site, a region, a country or world-wide), it may not be possible to conduct all assessments at the defined time (or within the designated window). See Section 9.1.1 and Appendix 18, COVID-19 APPENDIX: GUIDANCE ON STUDY CONDUCT DURING THE COVID-19 PANDEMIC for details.

# 9.1.3. Screening Phase (Weeks -4 to 0)

Only healthy subjects negative for HIV infection (if possible, the site should select an assay that is FDA-approved) and complying with the inclusion and exclusion criteria specified in Section 4 will be included into the study. The investigator will provide detailed information on the study to the subjects and will obtain written informed consent prior to each subject's participation in the study. All the procedures described in the Time and Events Schedule will only take place after written informed consent has been obtained.

Screening may be conducted in part after a sponsor- and Independent Ethics Committee (IEC)/Institutional Review Board (IRB)-pre-approved non-study specific screening consent process, but only if the relevant pre-screening tests are identical to the per protocol screening tests and are within 4 weeks (with 2 extra weeks to allow for start of hormonal contraception for female subjects and female partners of male subjects) prior to first vaccination. However, no study specific procedures, other than screening assessments, will be performed until the subject has signed the study-specific ICF. The non-study specific ICF will be considered source data.

During screening, subjects must pass the TOU, a questionnaire provided to the subject to document his/her understanding of the study (see Section 16.1 and Attachment 3). The TOU must be completed by all subjects, as the first assessment after signing of the ICF.

The following evaluations will be performed to determine eligibility requirements as specified in the inclusion and exclusion criteria:

- Medical history
- Physical examination, including weight and height
- Vital signs measurement
- Review of pre-study medications
- HIV-risk assessment (see Attachment 2) and counseling on avoidance of HIV infection
- Review of inclusion/exclusion criteria
- Blood sampling for complete blood count (CBC) with differential and platelets, blood chemistry, hepatitis B/C serology, and HIV testing (including pre- and post-HIV-test counseling)
- Sexually-transmitted infection testing (syphilis, chlamydia, gonorrhea, trichomonas [for female subjects; urine or vaginal swab may be used])
- Pregnancy counseling for both male and female subjects
- Female subjects of childbearing potential: serum β-hCG pregnancy testing
- Urinalysis

General eligibility for this clinical study will be dependent on results of laboratory tests and the medical assessment. Study subjects who qualify for inclusion based on the medical history, physical examination, and laboratory results will be contacted and scheduled for vaccination (Visit

2) within 28 days from signing ICF (with 2 extra weeks to allow for start of hormonal contraception for female subjects or female partners of male subjects).

Subjects with laboratory values or vital signs (eg, elevated blood pressure) not meeting eligibility criteria on the screening visit may have one repeat testing if the abnormality is not clinically significant and may be a testing aberrancy. The screening visit may be split into multiple days/visits. If the repeat screening assessment causes the subject to fall outside the screening window, all screening safety procedures should be repeated so that they are not more than 28 days prior to the Day 1 visit. These subjects will not be considered screen failures, if their repeat labs meet the inclusion criteria.

After medical history, physical examination, and laboratory data have been reviewed for completeness and adherence to inclusion/exclusion criteria, the subject can be deemed to be eligible for the study.

All pre-dose AEs will be recorded on the CRF, together with information about any concomitant medications.

In case a subject meets all eligibility criteria but is unable to adhere to the allowed screening period, all screening procedures (except ICF and TOU) should be repeated so that they fall within the allowed screening period.

If a subject is a screen failure but at some point in the future is expected to meet the subject eligibility criteria, the subject may be rescreened on one occasion only. Subjects who are rescreened will be assigned a new subject number, undergo the informed consent process, and then restart a new screening phase.

#### 9.1.4. Vaccination

#### Visit 2/Randomization/Vaccination 1

After re-check of inclusion/exclusion criteria (including concomitant medication), abbreviated physical examination (including weight measurement), measurement of vital signs, and a urine pregnancy test (for women of childbearing potential), eligible subjects will be randomized as described in Section 5.

If medical status and/or physical examination suggest(s) significant changes have occurred since screening, the clinically relevant screening assessments will be repeated and the Day 1 visit rescheduled. If the repeat screening assessment causes the subject to fall outside the screening window, all screening safety procedures should be repeated so that they are not more than 28 days prior to the Day 1 visit. These subjects will not be considered screen failures, if their repeat labs meet the inclusion criteria.

Pre-dose samples for hematology, biochemistry, HIV testing, urinalysis, and immunogenicity will be collected. Human leukocyte antigen will also be tested using the baseline blood sample. Pre-dose AEs will also be collected, together with information about any concomitant medications.

Study vaccine will be prepared by the site pharmacist, who will place an overlay on the syringes (to preserve blinding) and will send it to the clinic. After each vaccination, subjects will remain under observation at the study site for at least 30 minutes for presence of any acute reactions and solicited local (at injection site) and systemic events (see Section 9.3), and vital signs measurement will be repeated.

Subjects will be provided with a thermometer, ruler, and subject diary to measure and record body temperature and solicited local (at injection site) and systemic events for 7 days post-vaccination (day of vaccination and the subsequent 7 days).

In addition to an HIV-risk assessment, counseling related to avoidance of HIV infection, pre- and post-HIV-test counseling, and pregnancy counseling will be provided to all subjects (men and women).

#### Visit 6/Vaccination 2

An abbreviated physical examination (including weight measurement) and measurement of vital signs, will be performed for all subjects pre-vaccination. A urine pregnancy test must be performed before vaccination for women of childbearing potential, and results must be available and negative prior to vaccination. Pre-dose samples for hematology, biochemistry, HIV testing, and urinalysis will be collected. A pre-dose blood sample for the immunogenicity assays will be drawn. Pre-dose AEs will also be collected, together with information about any concomitant medications. After each vaccination, subjects will remain under observation at the study site for at least 30 minutes for presence of any acute reactions and solicited local (at injection site) and systemic events (see Section 9.3), and vital signs measurement will be repeated.

Subjects will be provided with a thermometer, ruler, and subject diary to measure and record body temperature and solicited local (at injection site) and systemic events for 7 days post-vaccination (day of vaccination and the subsequent 7 days).

In addition to an HIV-risk assessment, counseling related to avoidance of HIV infection, pre- and post-HIV-test counseling, and pregnancy counseling will be provided to all subjects (men and women).

Subjects will complete a social impact questionnaire (Attachment 4).

## Visit 9/Vaccination 3

The procedures for Visit 9 will be the same as at Visit 6 as detailed above, with the exception of the social impact questionnaire which will not be completed.

### Visit 13/Vaccination 4

The procedures for Visit 13 will be the same as at Visit 6 as detailed above.

## 9.1.5. Post-vaccination Follow-Up Phase

## Visits 2a, 3, 4, and 5

At Visit 2a (24-72 hours post-vaccination), a member of the site staff will have a (remote) safety follow-up communication with the subject (by e-mail, telephone, or visit, according to the subject's preference). The subject will be brought in for a clinic visit based on this assessment, if deemed necessary by the investigator/sub-investigator or upon request of the subject. Exception: for the sentinel group of 10 subjects, this will need to be an actual visit at 3 days post first vaccination. A (remote) safety follow-up communication 24-72 hours post-vaccination is not required if the vaccination was missed.

Visit 3 is a clinic visit for safety follow-up only, and will include an abbreviated physical examination (including weight measurement), vital signs measurement, and recording of concomitant medications and any AEs. In addition to an HIV-risk assessment, counseling related to avoidance of HIV infection will be provided to all subjects.

Visit 4 is a clinic visit that will include an abbreviated physical examination (including weight measurement), vital signs measurement, recording of concomitant medications and any AEs, and review of the diary for 7 days post-vaccination (day of vaccination and the subsequent 7 days). Samples will be collected for safety laboratory testing (CBC and serum chemistry) and humoral immunogenicity assays. In addition to an HIV-risk assessment, counseling related to avoidance of HIV infection will be provided to all subjects.

Visit 5 is a clinic visit that will include an abbreviated physical examination (including weight measurement), vital signs measurement, recording of concomitant medications and any AEs, and collection of samples for humoral and cellular immunogenicity assays. In addition to an HIV-risk assessment, counseling related to avoidance of HIV infection will be provided to all subjects.

### Visits 6a, 7, and 8

The procedures for Visits 6a, 7, and 8 will be the same as for Visits 2a, 4, and 5, respectively. Exception: no special requirements for the sentinel group for Visit 6a. At visits 7 and 8, both humoral and cellular immunogenicity samples will be collected.

### Visits 9a, 10, and 11

The procedures for Visits 9a, 10, and 11 will be the same as for Visits 2a, 4, and 5, respectively. Exception: no special requirements for the sentinel group for Visit 9a. At Visits 10 and 11, both humoral and cellular immunogenicity samples will be collected.

### Visit 12

Visit 12 is a clinic visit for safety follow-up only, and will include an abbreviated physical examination (including weight measurement), vital signs measurement, recording of concomitant medication, recording of SAEs, AEs leading to treatment discontinuation, and AESIs, and collection of samples for safety laboratory testing (CBC and serum chemistry). In addition to an

HIV-risk assessment, counseling related to avoidance of HIV infection will be provided to all subjects.

## Visits 13a, 14, and 15

The procedures for Visits 13a, 14, and 15 will be the same as at Visits 2a, 4, and 5, respectively. Exception: no special requirements for the sentinel group for Visit 13a. At Visits 14 and 15, both humoral and cellular immunogenicity samples will be collected.

# 9.1.6. Follow-Up Phase

Follow-up visits will be performed at the clinic at Week 60 and 72. Each visit includes a vital signs measurement, recording of concomitant medications, recording of SAEs, AEs leading to treatment discontinuation, and AESIs, and collection of samples for immunogenicity and safety laboratory testing (CBC and serum chemistry). In addition to an HIV-risk assessment, counseling related to avoidance of HIV infection will be provided to all subjects.

A complete physical exam will be performed at the final main study visit (Week 72). At Week 60, an abbreviated, symptom-directed exam will be performed as indicated by the investigator. Weight will be measured at both visits.

At the final main study visit (Week 72), samples for HIV testing and urinalysis will be collected. Pre- and post-HIV-test counseling will be provided to all subjects. Subjects will also complete a social impact questionnaire (Attachment 4).

# 9.1.7. Early Withdrawal/Exit Visit

In the event of early withdrawal from the main study (ie, before Week 72), the following procedures will be performed: an abbreviated physical examination (including weight measurement), vital signs measurement, recording of concomitant medications and any AEs, and collection of samples for safety laboratory testing (CBC and serum chemistry), the immunogenicity assays, urinalysis, and HIV testing. In addition to an HIV-risk assessment, counseling related to avoidance of HIV infection, pre- and post-HIV-test counseling, and pregnancy counseling will be provided to all subjects (men and women). A urine pregnancy test will be carried out for women of childbearing potential. Additionally, subjects will complete a social impact questionnaire (Attachment 4).

## 9.1.8. Optional Long-term Extension Phase

An optional LTE phase (approximately 3 years after Week 72) will be performed for subjects randomized to Group 2A, who have received all 4 vaccinations and are negative for HIV infection at Week 72.

The sponsor will be unblinded to study treatment at the Week 28 analysis and will notify the investigator and study-site personnel of subjects randomized to Group 2A. At Week 72, subjects randomized to Group 2A who have received all 4 vaccinations, will be asked to participate in the optional LTE phase and sign the ICF appendix for the optional LTE phase. During the first visit of the optional LTE phase, the remaining eligibility criteria for the optional LTE phase will be

verified. Subjects who attend their Week 72 visit prior to the sponsor's unblinding at the Week 28 analysis, will be enrolled in the optional LTE phase if they consent and sign the ICF appendix for the optional LTE phase and meet the eligibility criteria for the optional LTE phase. When the Week 28 sponsor unblinding subsequently occurs, subjects that started the optional LTE phase but turn out not to be in Group 2A of the main study will be withdrawn from the optional LTE phase.

If signing the ICF appendix is not possible at Week 72, signing should be performed at an extra visit (Visit 17bis) as soon as possible after Week 72 and at the latest before any assessment is done on the first visit of the optional LTE phase.

An optional 2-year extension of this 3-year optional LTE is introduced in protocol amendment 3. Subjects will be informed of the option to participate in this 2-year extension at the next possible visit after approval of this amendment. Subjects willing to participate will need to sign the ICF appendix for the 2-year extension at Visit 23. Subjects not willing to participate in the 2-year extension will have their final study visit at Visit 23. For subjects willing to participate: As of protocol amendment 5, the LTE will be shortened by one year, so Visit 26 and Visit 27 have been removed and Visit 25 will be the final visit. Participants who already had their Visit 25 or Visit 26 will be contacted to perform an extra unscheduled exit visit, to be performed within 6 weeks after local approval of protocol amendment 5. This can be either a telephone call or an actual site visit and will need to include the same assessments as in the current Visit 25, except for the social impact questionnaire and blood sampling for HIV and immunogenicity testing. In case a safety issue (including a recent HIV exposure) emerges during the call, the participant might be asked to come to the site for further evaluation.

Subjects will attend follow-up visits at the clinic from Week 96 until the final visit at Week 216 (for subjects who consent to be followed-up for approximately 3 years after week 72) or Week 264 (for subjects who consent to be followed-up for approximately 4 years after week 72). Each visit includes recording of any SAEs, AESIs, and concomitant medications (any medication given in conjunction with an SAE, as well as any recurrent or chronic use of immunomodulators/suppressors and corticosteroids), and collection of samples for cellular and humoral immunogenicity assays.

Samples for HIV testing will be collected. In addition to an HIV-risk assessment, counseling related to avoidance of HIV infection, pre- and post-HIV test counseling will be provided to all subjects.

Also, at each visit, subjects will complete a social impact questionnaire (Attachment 4).

## 9.2. Immunogenicity Evaluations

Humoral immune response assays will include, but are not limited to Env-Ab-binding assays, virus neutralization assay, and assays for Ab functionality.

Cellular immune response assays will include, but are not limited to IFN $\gamma$  ELISPOT assay, ICS, and multiparameter flow cytometry.

## 9.3. Safety Evaluations

Details regarding the PSRT and DRC are provided in Section 11.7 and 11.8, respectively.

Any clinically relevant changes occurring during the study must be recorded on the AE section of the CRF.

Any clinically significant abnormalities persisting at the end of the study/early withdrawal will be followed by the investigator until resolution or until a clinically stable endpoint is reached.

The study will include the following evaluations of safety and tolerability according to the time points provided in the Time and Events Schedule:

#### **AEs**

All AEs will be reported from the time a signed and dated ICF is obtained until 28 days after first dose of study vaccine, and thereafter, pre-dose and for 28 days after each subsequent dose of study vaccine/placebo. Unsolicited AEs with the onset date outside the timeframe defined above (>28 days after previous study vaccination), which are ongoing on the day of the subsequent vaccination, should be recorded on the CRF AE page. All SAEs and AEs leading to discontinuation from the study vaccination and AESIs (ie, confirmed HIV infection) are to be reported for the duration of the main study (see Section 12.3.1 for details). During the optional LTE phase, only SAEs and AESIs are to be reported. Other AEs are not collected during the optional LTE phase as the optional LTE phase begins 6 months after the last vaccination and it is very unlikely that an AE related to the study vaccine would only present that long after the last vaccination.

Adverse events will be followed by the investigator as specified in Section 12.

For solicited AEs, the following applies.

#### **Solicited AEs**

After vaccination, subjects will remain under observation at the study site for at least 30 minutes for presence of any acute reactions and solicited events. In addition, subjects will record solicited events in a diary for 7 days post-vaccination. All subjects will be provided with a diary and instructions on how to complete the diary (Section 9.1.1). Diary information will be transcribed by the study personnel in the appropriate CRF pages.

## Injection Site (Local) AEs

Subjects will be asked to note in the diary occurrences of pain/tenderness, erythema and induration/swelling at the study vaccine injection site daily for 7 days post-vaccination (day of vaccination and the subsequent 7 days). The extent (largest diameter) of any erythema, and induration/swelling should be measured (using the ruler supplied) and recorded daily.

## • Injection Site Pain/Tenderness

Injection site pain (eg, stinging, burning) is an unpleasant sensory and emotional experience associated with actual or potential tissue damage and occurring at the immunization site (with

or without involvement of surrounding tissue). Injection site tenderness is a painful sensation localized at the injection site upon palpation and/or movement of the limb. Due to subjective nature of the reaction, the severity assessment of pain/tenderness is self-reported (if a subject is unable to provide self-report, other reporters include parent/care giver or health care provider).<sup>6</sup>

## • Injection Site Erythema

Injection site erythema is a redness of the skin caused by dilatation and congestion of the capillaries localized at the injection site. It can best be described by looking and measuring.

# • Injection Site Swelling/Induration

Injection site swelling is a visible enlargement of an injected limb. It may be either soft (typically) or firm (less typical). Injection site induration is a palpable thickening, firmness, or hardening of soft tissue, usually has well-demarcated palpable borders, can be visible (raised or sunken compared to surrounding skin), is often 'woody' to touch and has a flat shape. As differentiation between swelling and induration may be difficult without health care professional's assessment, both symptoms have been combined to allow self-assessment by the subjects. Both swelling and induration can best be described by looking and measuring. <sup>16,17</sup>

Note: any other injection site events not meeting the above case definitions should be reported separately as unsolicited AEs.

## Systemic AEs

Subjects will be instructed on how to record daily temperature using a thermometer provided for home use. Subjects should record the temperature in the diary in the evening of the day of vaccination, and then daily for the next 7 days approximately at the same time each day. If more than one measurement is made on any given day, the highest temperature of that day will be used in the CRF.

Fever is defined as endogenous elevation of body temperature  $\ge 38^{\circ}$ C, as recorded in at least one measurement.<sup>19</sup>

Subjects will also be instructed on how to note daily in the diary symptoms for 7 days post-vaccination (day of vaccination and the subsequent 7 days) of the following events: fatigue, headache, nausea, myalgia, and chills.

The severity of these solicited systemic AEs will be graded according to the criteria presented in Section 12.1.3.

### **AESI**

Confirmed HIV infection in a subject during the study is considered an AESI. All AESIs, irrespective if considered serious or not by the investigator, shall be reported to the sponsor immediately and aggregate analyses performed either at the end of study and possibly at interim time points during the study.

## **Clinical Laboratory Tests**

Blood samples for serum chemistry and hematology and a urine sample for urinalysis will be collected. The investigator must review the laboratory results, document this review, and record any clinically relevant changes occurring during the study in the AE section of the CRF. The laboratory reports must be filed with the source documents.

In case a Grade 3 or Grade 4 laboratory abnormality, or any laboratory abnormality accompanied by clinically relevant signs or symptoms occurs (from the baseline visit onwards), all attempts will be made to perform a confirmatory test within 48 hours after the results have become available. After that, laboratory tests will be repeated weekly until values are resolved or stable.

The following tests will be performed by the local laboratory (\*parameters only measured at screening):

- Hematology Panel
  - -hemoglobin -platelet count
  - -hematocrit
  - -red blood cell (RBC) count
  - -white blood cell (WBC) count with differential

A WBC evaluation may include any abnormal cells, which will then be reported by the laboratory. A RBC evaluation may include abnormalities in the RBC count and/or RBC parameters and/or RBC morphology, which will then be reported by the laboratory.

In addition, any other abnormal cells in a blood smear will also be reported.

• Serum Chemistry Panel

-creatinine -creatine phosphokinase\*

-glucose\* -bilirubin\*

-aspartate aminotransferase (AST) -FSH (post-menopausal women only)\*

-alanine aminotransferase (ALT)

Urinalysis

Dipstick -protein
-specific gravity -blood
-pH -ketones

-glucose

Microscopic reflex testing will be carried out in the event of abnormal urinalysis tests, except when the investigator considers the abnormal urinalysis result to be from menstrual origin.

In the microscopic examination, observations other than the presence of WBC, RBC, and casts may also be reported by the laboratory.

Laboratory values will be graded according to a modified version of the Division of Acquired Immunodeficiency Syndrome (DAIDS) grading table, Version 2.0 (Attachment 1), and, if clinically significant, reported as AEs. Laboratory reference ranges will be applied according to the subject's sex at birth.

Additional clinical laboratory assessments to be performed are as follows:

- Serum (at screening) and Urine (pre-dose at vaccinations and the early Exit visit) Pregnancy Testing for women of childbearing potential only
- Serology (hepatitis B surface antigen, HCV Ab; at screening)
- HIV testing (at screening, vaccinations, Week 72, the early Exit visit, and at each visit of the optional LTE phase)
- Syphilis, chlamydia, gonorrhea, trichomonas [for female subjects; urine or vaginal swab may be used] (at screening)

## Vital Signs (oral or tympanic temperature, pulse/heart rate, blood pressure)

Vital sign measurements will be performed at time points specified in the Time and Events Schedule.

Blood pressure and pulse/heart rate measurements will be assessed with a completely automated device. Manual techniques will be used only if an automated device is not available.

Blood pressure and pulse/heart rate measurements should be preceded by at least 5 minutes of rest in a quiet setting without distractions (eg, television, cell phones).

If any clinically significant changes in vital signs are noted, they will be reported as AEs and followed to resolution, or until reaching a clinically stable endpoint.

## **Physical Examination**

Full physical examination will be carried out at screening and at the final main study visit (Week 72). At all other main study visits, an abbreviated, symptom-directed exam will be performed as indicated by the investigator based on any clinically relevant issues, clinically relevant symptoms, and medical history. Symptom-directed physical examination may be repeated if deemed necessary by the investigator. Height will be measured at screening. Weight will be measured at every main study visit.

Physical examinations will be performed by the investigator or designated medically-trained clinician. Any screening or baseline abnormality should be documented in the medical history page of the CRF. Any clinically relevant post-baseline abnormality or any clinically relevant worsening versus baseline conditions should be documented in the AE pages of the CRF.

# 9.4. Human Immunodeficiency Virus Testing and Vaccine Induced Seropositivity

## 9.4.1. Human Immunodeficiency Testing

HIV testing will be performed as indicated in the Time and Events Schedule.

At screening and baseline, subjects will be tested for HIV infection, and must be negative to be entered into the study. If possible, the site should select an assay that is US FDA-approved.

At all other main study visits that include HIV-testing, a study-specific HIV-testing algorithm (detailed in the Laboratory Manual) will be followed. Information provided to the clinical staff of the study site will not include the results of specific tests, but will state only the final interpretation as "infected" or "uninfected". This system allows timely HIV testing without compromising the double-blind nature of the study. The algorithm used for HIV testing throughout the main study aims to differentiate false-positive results (Vaccine Induced Seropositivity [VISP]) from true positives (HIV infection).

During the optional LTE phase, the study-specific HIV-testing algorithm described above will be followed as long as treatment assignment is blinded. Upon study unblinding, unblinded HIV and VISP results will be reported.

If a false-positive HIV test result develops during the study, further VISP testing will be offered via post-study follow-up (see Section 9.4.3).

# 9.4.2. Management of Subjects who Become HIV-infected During the Study

Test results performed to confirm the diagnosis will be forwarded to the study staff. Subjects who become HIV infected during the study, including the optional LTE phase, will be (see Section 12.3.3):

- Excluded from further vaccinations.
- Provided counseling and referred for medical treatment.
- Informed about observational studies monitoring subjects with HIV infection.
- Excluded from initiation of the optional LTE phase.

## 9.4.3. VISP

In general, HIV-uninfected subjects who participate in preventative HIV-vaccine studies may develop HIV-specific antibodies as a result of an immune response to the candidate HIV vaccine, referred to as VISP. These antibodies may be detected in common HIV-serologic tests, causing the test to appear positive even in the absence of actual HIV infection. Vaccine Induced Seropositivity may become evident during the study or after the study has been completed.

Should an HIV-Ab test give a positive result for a particular subject during the study, the central lab will carry out a follow-up testing algorithm either to exclude or confirm HIV infection. Further details of this algorithm are given in the Laboratory Manual.

Subjects should not donate blood during the study. Blood donation options for those subjects who wish to resume blood donation after the study will be explained at the final study follow-up visit.

In the case of VISP, if, either during the study or after the end of the study, a subject requires an HIV test outside the study (eg, to obtain a travel visa or insurance, or for medical reasons), he/she should contact the research center. The center can issue a written statement giving details on VISP and on the testing algorithm to be followed. If requested by a subject, repeat HIV testing will be available at the site at most every 3 months to confirm their HIV status. It is highly preferable that this repeat HIV testing will be performed at the research center. More frequent testing is only allowed after sponsor approval. Testing for a particular subject will be available as long as VISP is present for this subject.

Depending on the local availability of a follow-up protocol, subjects could join into such a study that specifically follows the course of VISP. Such a study may not be available at all sites. However, if such a study is not available, the site will provide HIV testing on request as described in the previous paragraph.

In addition to providing testing, subjects will always receive pre- and post-test counseling.

## 9.4.4. Social Impact

Subjects in preventive HIV-vaccine clinical studies may experience problems with personal relationships, employment, education, health care, housing, health, disability or life insurance, travel, and immigration. In relation to a subject's family, friends, and/or colleagues, the social impact could manifest in one or more ways, resulting in social conflicts and stigmatization:

- 1. The investigational vaccine is thought to be harmful to the subject's health, including a belief that it might cause HIV infection.
- 2. The subject is perceived as HIV infected or at high risk.
- 3. Repercussions from any VISP.

For these reasons, subjects will complete a social impact questionnaire (at the timepoints specified in the Time and Events Schedule) to evaluate any potential consequences of the subject's participation. For more information, please refer to the Study Procedures Manual.

## 9.5. Sample Collection and Handling

The actual dates and times of sample collection must be recorded in the CRF or laboratory requisition form.

See the Time and Events Schedule for the timing and frequency of all sample collections.

Instructions for the collection, handling, storage, and shipment of samples are found in the Laboratory Manual that will be provided. Collection, handling, storage, and shipment of samples must be under the specified, and where applicable, controlled temperature conditions as indicated in the Laboratory Manual.

# 10. SUBJECT COMPLETION/DISCONTINUATION OF STUDY TREATMENT/WITHDRAWAL FROM THE STUDY

## 10.1. Completion

A subject who is not participating in the optional LTE phase will be considered to have completed the study if he or she has completed the assessments at Week 72. A subject who is participating in the optional LTE phase will be considered to have completed the main study if he or she has completed the assessments at Week 72 and will be considered to have completed the optional LTE phase if he or she has completed the assessments at the last visit of the optional LTE phase at Week 216 (for subjects who consent to be followed-up for approximately 3 years after Week 72) or Week 264 (for subjects who consent to be followed-up for approximately 4 years after week 72).

# 10.2. Discontinuation of Study Treatment

Subjects will be withdrawn from study vaccine administration for the reasons listed below. These subjects must not receive any additional dose of study vaccine but should enter the follow-up phase with assessments of safety and immunogenicity. The subject will be encouraged to complete the post-vaccination follow-up visits of the last vaccination received and a 12 and 24 weeks follow-up visit after the last vaccination received, specified as Week 60 and Week 72 in the Time and Events Schedule. Additional unscheduled visits may be performed for safety/tolerability reasons, if needed. In case the subject withdraws before receiving the first vaccination, the subject is not required to attend follow-up visits. In case of questions, the investigator is encouraged to contact the study responsible physician. Subjects who prematurely discontinue study treatment are not eligible for the optional LTE phase.

- Unblinding
- Anaphylactic reaction following vaccination
- Pregnancy
- Any related SAE
- Any related AE, worsening of health status or intercurrent illnesses that, in the opinion of the investigator, requires discontinuation from study vaccine
- Confirmed HIV infection
- Chronic or recurrent use of immunosuppressants (after discussion with the sponsor)
- Missing more than 1 study vaccination
- Any event (eg, overdose, incorrect dosing) that, in the opinion of the investigator (in agreement with the sponsor), would require discontinuation of study vaccine

#### 10.3. Contraindications to Vaccination

The following events constitute a contraindication to vaccination at that point in time. If any of these events occur at the scheduled time for vaccination, the vaccination can be rescheduled (as long as this is in agreement with the allowed windows, see Section 9.1.2):

- Acute illness at the time of vaccination. This does not include minor illnesses, such as diarrhea or mild upper-respiratory tract infection.
- Fever (oral temperature  $\ge 38.0^{\circ}$ C) at the time of vaccination.

# 10.4. Withdrawal From the Study

Each subject has the right to withdraw from the study at any time for any reason without affecting the right to treatment by the investigator. The investigator should make an attempt to contact subjects who did not return for scheduled visits or follow-up. Although the subject is not obliged to give reason(s) for withdrawing prematurely, the investigator should make a reasonable effort to ascertain the reason(s) while fully respecting the subject's rights.

A subject will be withdrawn from the study for any of the following reasons:

- Lost to follow-up
- Withdrawal of consent
- Death
- Repeated failure to comply with protocol requirements
- Decision by the sponsor or the investigator to stop or cancel the study
- Decision by local regulatory authorities and Institutional Review Board/Independent Ethics Committee to stop or cancel the study

If a subject is lost to follow-up, every reasonable effort (at least 2 documented attempts to contact the subject by telephone and at least one documented written attempt) must be made by the study-site personnel to contact the subject and determine the reason for discontinuation/withdrawal. The measures taken to follow-up must be documented.

When a subject withdraws before completing the study, the reason for withdrawal is to be documented in the CRF and in the source document. Study vaccine assigned to the withdrawn subject may not be assigned to another subject. Subjects who are vaccinated and who withdraw will not be replaced. If a subject withdraws early from the study, assessments for early withdrawal should be obtained (see Section 9.1.7).

Subjects who wish to withdraw consent from participation in the study will be offered a single Exit visit for safety follow-up (prior to formal withdrawal of consent). They have the right to refuse. The exit visit is only applicable to the main study until Week 72.

### 10.5. Withdrawal From the Use of Samples in Future Research

The subject may withdraw consent for use of samples for research (see Section 16.2.5). In such a case, samples will be destroyed after they are no longer needed for the clinical study. Details of the sample retention for research are presented in the main ICF.

### 11. STATISTICAL METHODS

Statistical analysis will be done by the sponsor or under the authority of the sponsor. A general description of the statistical methods to be used to analyze the safety and immunogenicity data is outlined below. Specific details will be provided in the Statistical Analysis Plan.

## 11.1. Subject Information

For all subjects, demographic characteristics (eg, age, height, weight, body mass index [BMI], race, and gender), and other baseline characteristics (eg, medical history, concomitant diseases) will be tabulated and summarized with descriptive statistics.

## 11.2. Analysis Populations

The <u>safety population</u> will consist of all subjects who received at least one dose of study vaccine, and for whom any post-dose data is available.

The <u>immunogenicity population</u> will consist of all subjects who received at least one dose of study vaccine, and who have data from at least one evaluable post-dose blood sample.

The <u>per protocol immunogenicity population</u> will consist of all randomized and vaccinated subjects for whom immunogenicity data are available, excluding subject samples with major protocol deviations expecting to impact the immunogenicity outcomes (for example missed vaccinations, natural infections, etc).

# 11.3. Sample Size Determination

The sample sizes in the main study are regarded to be appropriate to assess the safety and tolerability of the different vaccine regimens. Placebo recipients are included for blinding and safety purposes and will provide control specimens for immunogenicity assays.

While mild to moderate vaccine reactions (local site and systemic responses) are expected, AEs that preclude further vaccine administration or more serious ones that would limit product development are not anticipated. With 110 individuals in the tetravalent Ad26.Mos4.HIV vaccine regimen, the observation of 0 such reactions would be associated with a 95% confidence that the true rate is <2.7%. For the combined active groups (n 165), there would be 95% confidence that the true rate is <1.8% when 0 events are observed. The following table shows the probabilities of observing at least one AE given true AE rates.

Probability of Observing at Least one AE in n Subjects

| True AE Rate | n = 55 | n = 110 | n=165 |
|--------------|--------|---------|--------|
| 0.1% | 5% | 10% | 15% |
| 0.5% | 24% | 42% | 56% |
| 1% | 42% | 67% | 81% |
| 2.5% | 75% | 94% | 98.5% |
| 5% | 94% | 99.6% | >99.9% |
| 10% | 99.7% | >99.9% | >99.9% |

The primary population for the safety analyses will consist of all subjects who received at least 1 dose (Ad26.Mos.HIV, Ad26.Mos4.HIV, or placebo).

Anticipating a dropout rate of approximately 10%, the sample sizes will allow detection of approximately 1.5-fold differences in Env-binding Ab titers between the groups with Ad26.Mos4.HIV (approximately 100 evaluable subjects) and their corresponding group with Ad26.Mos.HIV only (approximately 50 evaluable subjects); with 80% probability, assuming a 1-sided 5% Type I error and a standard deviation of 0.4 on the log<sub>10</sub> scale.

The immunogenicity population will consist of all subjects who received at least 1 dose and have at least 1 measured post-dose blood sample collected.

# 11.4. Immunogenicity Analyses

Descriptive statistics (actual values and changes from reference with 95% confidence interval) will be calculated for continuous parameters. Frequency tabulations will be calculated for discrete parameters. Graphical representations of changes in immunologic parameters will be made as applicable.

No formal hypothesis on immunogenicity will be tested. The analysis of immunogenicity will be done on the (per protocol) immunogenicity population as defined in Section 11.2.

Differences between groups at a specific time point will be tested for exploratory purposes by a 2-sample t-test if the data appear to be normally distributed. If not, the non-parametric Wilcoxon rank sum test will be used. If portions of the measurements are censored below the assay quantification limit, the Gehan-Wilcoxon test will be employed. All statistical tests will be 2-sided and will be considered statistically significant if p<0.05.

Frequency tabulations will be calculated for discrete (qualitative) immunologic parameters. Significant differences between groups will be determined by a 2-sided Fisher's exact test.

## 11.5. Safety Analyses

No formal statistical testing of safety data is planned. Safety data will be analyzed descriptively.

Baseline for all safety parameters will be defined as the last evaluation done before the first dose of study vaccine.

#### **AEs**

The verbatim terms used in the CRF by investigators to identify AEs will be coded using the Medical Dictionary for Regulatory Activities (MedDRA). All reported AEs and events-related diary information (solicited local at injection site and systemic, and unsolicited) with onset within 28 days after each vaccination (ie, treatment-emergent AEs, and AEs that have worsened since baseline) will be included in the analysis. For each AE, the number and percentage of subjects who experience at least one occurrence of the given event will be summarized by group and/or by vaccine.

Summaries, listings, datasets, or subject narratives may be provided, as appropriate, for those subjects who die, who discontinue treatment due to an AE, or who experience a severe AE, an SAE, or an AESI.

Summaries and listings may be provided separately for AEs with onset outside the above defined timeframe and that were reported pre-dose at the moment of subsequent vaccinations.

Solicited local (at injection site) and systemic AEs will be summarized descriptively. The overall frequencies per vaccine group as well as frequencies according to severity and duration will be calculated for solicited AEs. In addition, the number and percentages of subjects with at least one solicited local (at injection site) or systemic AE will be presented. Frequencies of solicited and unsolicited AEs, separately for all and vaccination-related only, will be presented by System Organ Class and preferred term.

## **Clinical Laboratory Tests**

Laboratory data will be summarized by type of laboratory test. Laboratory abnormalities will be determined according to a modified version of the DAIDS grading table, Version 2.0 (Attachment 1), and in accordance with the normal ranges of the clinical laboratory. Laboratory abnormalities will be tabulated per treatment group and/or per vaccine.

## **Vital Signs**

The percentage of subjects with values beyond pre-specified limits (see Attachment 1) will be summarized.

## **Physical Examination**

Physical examination findings will not be tabulated separately. Clinically relevant findings will be reported as AE and will be tabulated and listed as AEs. BMI will be calculated using the recording of height at screening.

## **Social Impact Questionnaire**

Data from the Social Impact Questionnaire will be summarized using descriptive statistics.

## 11.6. Analysis Time Points

An interim immunogenicity analysis will be performed once approximately 60 subjects have completed the Week 16 visit and will be unblinded at the group level, but not at the subject level (for details see Section 5).

The primary analysis will be performed in an unblinded fashion (for details see Section 5), once all subjects have completed the Week 28 visit (ie, 4 weeks after the third injection) or discontinued earlier. An additional analysis will be performed once all subjects have completed the Week 52 visit (ie, 4 weeks after the fourth injection) or discontinued earlier. The final analysis of the main study will be performed once all subjects have completed their final main study visit at Week 72 or discontinued earlier. The final analysis of the LTE phase (optional and only for subjects randomized to Group 2A) will be performed once all included subjects have completed the last

visit of the optional LTE phase (Week 216 for subjects who consent to be followed-up for approximately 3 years after Week 72 or Week 264 for subjects who consent to be followed-up for approximately 4 years after Week 72), or discontinued earlier.

### 11.7. PSRT

A PSRT will review blinded safety data reports on a regular basis (at least 2 times per month) starting from one week after first vaccination until the last subject has completed the Week 52 visit, and thereafter as needed.

After a sentinel group of 10 subjects received the first injection, further vaccinations will be paused until a 3 day safety evaluation is performed. This evaluation will be performed by the PSRT and the PI(s) of the subjects involved and will be based on the information received from the investigator(s) by email/telephone.

If an administration of vaccine is considered, by PSRT review, to raise significant safety concerns, all enrollment and vaccinations will be suspended until recommendations are issued (see Section 11.9, Table 2). In specific cases a Data Review Committee (DRC) meeting will be triggered.

The PSRT will include, but will not be limited to medical and safety representatives from the sponsor, sites, DAIDS, BIDMC, HVTN, IAVI, and MHRP. The PSRT responsibilities, authorities, and procedures will be documented in its charter.

### 11.8. DRC

A DRC will be established for this study, which will monitor data to ensure the safety and well-being of the subjects enrolled. The DRC will review data as indicated below. The conclusions of the DRC will be communicated to the investigators, the Institutional Review Board/Independent Ethics Committee, and the national regulatory authorities, as appropriate.

The DRC will specifically review safety data (solicited and unsolicited AEs, SAEs, and available laboratory assessments) at 3 time points:

- Review blinded safety data (4 weeks of follow-up) after 15% of subjects have received their
  first injection. The DRC will review these interim safety results and will allow administration
  of the first dose of Ad26.Mos4.HIV/placebo (first injection) in the VAC89220HPX2003 study
  only if no significant safety concerns are identified.
- Review blinded safety data (4 weeks of follow-up) after 30% of subjects have received their first injection.
- Review blinded safety data (4 weeks of follow-up) after 30% of subjects have received their third injection.

In addition, ad hoc review may be performed further to the occurrence of any AE/SAE leading to a study holding situation as outlined in Section 11.9, or at request of the PSRT.

The DRC will include medical experts in vaccines and at least one statistician. The DRC can include members from both inside and outside Janssen, but will not include any study team personnel or people otherwise directly involved in the study conduct, data management, or statistical analysis for the study. The DRC responsibilities, authorities, and procedures will be documented in its charter.

## 11.9. Study Holding Rules

If an administration of vaccine is considered, by the PSRT, to raise significant safety concerns, all screening and vaccinations will be suspended until recommendations are issued. The AEs that may lead to a safety pause or prompt PSRT AE review are summarized below in Table 2. These study holding rules apply to related AEs that occur up to 4 weeks after vaccination and to SAEs occurring up to 4 weeks after the last vaccination.

| Table 2: AE Notification and Safety Pause/AE Review Rules1 | | | |
|---|---|---|---|
| (S)AE and<br>Relationship <sup>2</sup> | Severity | Site Principal Investigator Action | PSRT/DRC Action <sup>3</sup> |
| SAE, related | Any<br>grade | Notify Study Responsible Physician or designee<br>AND fax SAE form to Global Medical Safety<br>Office, immediately and no later than 24 h after<br>becoming aware of the event | Immediate pause for PSRT review of safety data |
| SAE, not related | Grade 5 | Notify Study Responsible Physician or designee<br>AND fax SAE form to Global Medical Safety<br>Office, immediately and no later than 24 h after<br>becoming aware of the event | PSRT review and consideration of pause |
| AE <sup>4</sup> , related | Grade 3<br>or<br>Grade 4 | Notify Study Responsible Physician immediately and no later than 24 h after becoming aware of the event | PSRT review and consideration of pause |
| Three subjects with a similar related AE <sup>5</sup> | Grade 3<br>or<br>Grade 4 | Not applicable | Immediate pause for DRC review of safety data |

The contact details of the medical team are in the Contact Information page(s). The Study Responsible Physician (or designee) is responsible for the immediate notification of PSRT/DRC members and coordination of a PSRT/DRC meeting.

- Applicable for AEs/SAEs occurring up to 4 weeks after the last vaccination. For a Grade 3/4 laboratory related AE, the test must be repeated at least once, within 48 hours of the site becoming aware of the abnormal value. PSRT evaluation for consideration of a pause will proceed without waiting for repeat testing. Start of DRC review will require a confirmation of the laboratory test within 48 hours.
- Related: suspicion of relationship between the study vaccine and the AE. Not related: no suspicion of relationship between the study vaccine and the AE. (Relationship as assessed by investigator)
- All sites will be notified immediately in case of a safety pause.
- For Grade 3 solicited related AEs, immediate PSRT review is mandatory only if the event persists for longer than 3 consecutive days, and the event doesn't get worse during this time. PSRT evaluation for consideration of a pause will proceed for all other cases not specified in footnote 4.
- <sup>5</sup> Applicable for the following related AEs:
  - All Grade 4 AEs (regardless of duration)
  - Grade 3 unsolicited AEs (regardless of duration)
  - Grade 3 solicited AEs (only if persisting for longer than 3 consecutive days)

After each DRC review of a similar AE, the DRC will indicate the conditions under which they require further notification and/or review of the subsequent similar AEs.

Vaccinations for an individual subject may be suspended for safety concerns other than those described in the table, at the discretion of the investigator if he/she feels the subject's safety may be threatened. The investigator may ask for a PSRT meeting to be held for any single event or combination of multiple events which, in his/her professional opinion, jeopardize the safety of the subjects or the reliability of the data.

Vaccinations for the study may be suspended for safety concerns other than those described in the table, or before pause rules are met, if, in the judgment of the DRC, subject safety may be threatened.

For events in the table above, the investigator notifies the sponsor's study responsible physician (or designee) immediately, and in all cases within 24 hours at the latest after the site observes, or is notified of, the AE, and the study responsible physician (or contacted sponsor's representative) then notifies the PSRT immediately. If the case(s) is (are) deemed to fulfill the potential holding rules, the PSRT will convene within one business day to review these AEs. The PSRT will review and determine disposition, including whether the DRC needs to review the event(s).

If a study pause is triggered by the PSRT, all screening and vaccinations will be held until review by the PSRT or DRC is complete. Resumption of screening and study treatment may be determined by the PSRT or DRC (in consultation with the FDA, if required) following a cumulative review of the available safety data as outlined in the charter. The clinical sites will be allowed to resume activities upon receipt of a written notification from the sponsor. As needed, the appropriate regulatory authorities will be informed in writing of the decision by the PSRT and/or DRC to resume or discontinue study activities. The site is responsible for notifying their IEC/IRB according to local standards and regulations. The sponsor is responsible for notifying the FDA.

### 12. AE REPORTING

Timely, accurate, and complete reporting and analysis of safety information from clinical studies are crucial for the protection of subjects, investigators, and the sponsor, and are mandated by regulatory agencies worldwide. The sponsor has established Standard Operating Procedures in conformity with regulatory requirements worldwide to ensure appropriate reporting of safety information; all clinical studies conducted by the sponsor or its affiliates will be conducted in accordance with those procedures.

### Method of Detecting AEs and SAEs

Care will be taken not to introduce bias when detecting AEs or SAEs. Open-ended and non-leading verbal questioning of the subject is the preferred method to inquire about AE occurrence. For some studies, subjects are not always able to provide valid verbal responses to open-ended questions. In these circumstances, another method of detecting these events is specified.

#### Solicited AEs

Solicited AEs are predefined local (at the injection site) and systemic events for which the subject is specifically questioned and which are noted by subjects in their diary (see Section 9.1.1).

#### **Unsolicited AEs**

Unsolicited AEs are all AEs for which the subject is NOT specifically questioned in the subject diary.

### 12.1. Definitions

#### 12.1.1. AE Definitions and Classifications

#### ΑE

An AE is any untoward medical occurrence in a clinical study subject administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal finding), symptom, or disease temporally associated with the use of a medicinal (investigational or non-investigational) product, whether or not related to that medicinal (investigational or non-investigational) product. (Definition per International Conference on Harmonisation [ICH])

This includes any occurrence that is new in onset or aggravated in severity or frequency from the baseline condition, or abnormal results of diagnostic procedures, including laboratory test abnormalities.

Note: The sponsor collects AEs starting with the signing of the ICF (see Section 12.3.1 for time of last AE recording).

#### SAE

An SAE based on ICH and European Guidelines on Pharmacovigilance for Medicinal Products for Human Use is any untoward medical occurrence that at any dose:

- Results in death
- Is life-threatening
  (The subject was at risk of death at the time of the event. It does not refer to an event that hypothetically might have caused death if it were more severe.)
- Requires inpatient hospitalization or prolongation of existing hospitalization
- Results in persistent or significant disability/incapacity
- Is a congenital anomaly/birth defect
- Is a suspected transmission of any infectious agent via a medicinal product
- Is Medically Important\*

\*Medical and scientific judgment should be exercised in deciding whether expedited reporting is also appropriate in other situations, such as important medical events that may not be immediately life threatening or result in death or hospitalization but may jeopardize the subject or may require intervention to prevent one of the other outcomes listed in the definition above. These should usually be considered serious.

If a serious and unexpected AE occurs for which there is evidence suggesting a causal relationship between the study vaccine and the event (eg, death from anaphylaxis), the event must be reported as a serious and unexpected suspected adverse reaction by the sponsor to the Health Authorities and by the investigator to the IEC/IRB according to regulatory and local requirements.

# Unlisted (Unexpected) AE/Reference Safety Information

An AE is considered unlisted if the nature or severity is not consistent with the applicable product reference safety information. For Ad26.Mos4.HIV, Ad26.Mos.HIV, and Clade C gp140, the expectedness of an AE will be determined by whether or not it is listed in the Investigator's Brochure.

#### **AE** Associated With the Use of the Vaccine

An AE is considered associated with the use of the vaccine if the attribution is related by the definition listed in Section 12.1.2.

### **AESI**

Confirmed HIV infection in a subject is considered an AESI. All AESIs, irrespective if considered serious or not by the investigator, shall be reported to the sponsor immediately and aggregate analyses performed either at the end of study and possible at interim time points during the study.

#### 12.1.2. Attribution Definitions

Every effort should be made by the investigator to explain any AE and assess its potential causal relationship, ie, to administration of the study vaccine or to alternative causes (eg, natural history of the underlying diseases, concomitant therapy). This applies to all AEs, whether serious or non-serious.

Causality of AEs should be assessed by the investigator based on the following:

**Related**: there is a reasonable possibility that the study vaccine contributed to the AE.

**Unrelated**: there is no suspicion that there is a relationship between the study vaccine and the AE; there are other more likely causes and administration of the study vaccine is not suspected to have contributed to the AE.

By definition, all solicited AEs at the injection site (local) will be considered related to the study vaccine administration.

## 12.1.3. Severity Criteria

All AEs, laboratory data, and fever will be coded for severity using a modified version of the DAIDS grading table, Version 2.0 (Attachment 1).

The severity of solicited AEs will be graded in the diary by the subject based on the severity assessment provided in the diary and then verified by the investigator using the DAIDS grading table.

For AEs not identified in the grading table (eg, diagnosis of HIV infection), the following guidelines will be applied:

| Mild | Grade 1 | Symptoms causing no or minimal interference with usual social and functional activities |
|---|---|---|
| Moderate | Grade 2 | Symptoms causing greater than minimal interference with usual social and functional activities |
| Severe | Grade 3 | Symptoms causing inability to perform usual social and functional activities |
| Potentially life-threatening | Grade 4 | Symptoms causing inability to perform basic self-care functions OR medical or operative intervention indicated to prevent permanent impairment, persistent disability |
| Fatal | Grade 5 | For any AE where the outcome is death, the severity of the AE is classified as Grade 5 |

## 12.2. Situations Requiring Special Notification

Safety events of interest on a sponsor study vaccine that require expedited notification to the sponsor or safety evaluation include, but are not limited to:

- Overdose of a sponsor study vaccine
- Suspected abuse/misuse of a sponsor study vaccine
- Accidental or occupational exposure to a sponsor study vaccine
- Medication error involving a sponsor product (with or without subject exposure to the sponsor study vaccine, eg, name confusion)
- Exposure to a sponsor study vaccine from breastfeeding

Subject-specific situations requiring special notification should be recorded in the CRF. Any situation requiring special notification that meets the criteria of an SAE should be recorded on the SAE form. Additional reporting from the sites to IEC/IRB and HA should be performed according to local regulations.

#### 12.2.1. AESI

Confirmed HIV infection in a subject is considered an AESI. All AESIs, irrespective if considered serious or not by the investigator, shall be reported to the sponsor immediately and aggregate analyses performed either at the end of study and possible at interim time points during the study.

Data collection on AESI will be performed through a questionnaire. The questionnaire has to be sent to the sponsor within 24 hours of awareness of the confirmed HIV infection in a subject.

## 12.3. Procedures

### 12.3.1. All AEs

All AEs and situations requiring special notification (see Section 12.2) will be reported from the time a signed and dated ICF is obtained until 28 days (including relevant visit window, if applicable) after first dose of study vaccine, and thereafter, pre-dose and for 28 days (including relevant visit window, if applicable) after each subsequent dose of study vaccine. Unsolicited AEs with the onset date outside the timeframe defined above (>28 days after previous study vaccination), which are ongoing on the day of the subsequent vaccination, should be recorded on the CRF AE page.

All SAEs and AEs leading to discontinuation from the study vaccination (regardless of the causal relationship) and AESIs (ie, confirmed HIV infection) are to be reported for the duration of the main study. During the optional LTE phase, only SAEs and AESIs are to be reported. The sponsor will evaluate any safety information that is spontaneously reported by an investigator beyond the time frame specified in the protocol.

All events that meet the definition of an SAE will be reported as SAEs, regardless of whether they are protocol-specific assessments.

The investigator will monitor and analyze study data including all AE and laboratory data as they become available and will make determinations regarding the severity of the adverse experiences and their relation to study vaccine. Adverse events will be deemed either related to study vaccine or not related to study vaccine, according to Section 12.1.2. To ensure that all AEs are captured in a timely manner, CRFs will be entered in real-time, and subjected to review to identify AEs which may invoke study pausing rules.

The investigator or designee must review both collected solicited events and other AE CRFs to insure prompt and complete identification of all events that require expedited reporting as SAEs, invoke study pausing rules or are other serious and unexpected events.

All AEs, regardless of seriousness, severity, or presumed relationship to vaccine, must be recorded using medical terminology in the source document and the CRF. Whenever possible, diagnoses should be given when signs and symptoms are due to a common etiology (eg, cough, runny nose, sneezing, sore throat, and head congestion should be reported as "upper respiratory infection"). Investigators must record in the CRF their opinion concerning the relationship of the AE to study therapy. All measures required for AE management must be recorded in the source document and reported according to sponsor instructions.

The sponsor assumes responsibility for appropriate reporting of AEs to the regulatory authorities. The sponsor will also report to the investigator (and the head of the investigational institute where required) all suspected unexpected serious adverse reactions (SUSARs). The investigator (or sponsor where required) must report SUSARs to the appropriate IEC/IRB that approved the protocol unless otherwise required and documented by the IEC/IRB. A SUSAR will be reported to

regulatory authorities unblinded. Participating investigators and IEC/IRB will receive a blinded SUSAR summary, unless otherwise specified.

For all studies with an outpatient phase, including open-label studies, the subject must be provided with a "wallet (study) card" and instructed to carry this card with them for the duration of the study indicating the following:

- Study number
- Statement, in the local language(s), that the subject is participating in a clinical study
- Investigator's name and 24-hour contact telephone number
- Local sponsor's name and 24-hour contact telephone number (for medical staff only)
- Site number
- Subject number
- Any other information that is required to do an emergency breaking of the blind

### 12.3.2. SAEs

All SAEs occurring during the study, including the optional LTE phase, must be reported to the appropriate sponsor contact person by study-site personnel within 24 hours of their knowledge of the event.

Information regarding SAEs will be transmitted to the sponsor using the SAE Form, which must be completed and signed by a physician from the study site, and transmitted to the sponsor within 24 hours of their knowledge of the event. The initial and follow-up reports of an SAE should be made by facsimile (fax) and/or email.

All SAEs that have not resolved by the end of the study, or that have not resolved upon discontinuation of the subject's participation in the study, must be followed until any of the following occurs:

- The event resolves
- The event stabilizes
- The event returns to baseline, if a baseline value/status is available
- The event can be attributed to agents other than the vaccine or to factors unrelated to study conduct
- It becomes unlikely that any additional information can be obtained (subject or health care practitioner refusal to provide additional information, lost to follow-up after demonstration of due diligence with follow-up efforts)

Suspected transmission of an infectious agent by a medicinal product will be reported as an SAE. Any event requiring hospitalization (or prolongation of hospitalization) that occurs during the course of a subject's participation in a study must be reported as an SAE, except hospitalizations for the following:

- Hospitalizations not intended to treat an acute illness or AE (eg, social reasons such as pending placement in long-term care facility)
- Surgery or procedure planned before entry into the study (must be documented in the CRF). Note: Hospitalizations that were planned before the signing of the ICF, and where the underlying condition for which the hospitalization was planned has not worsened, will not be considered SAEs. Any AE that results in a prolongation of the originally planned hospitalization is to be reported as a new SAE.

The cause of death of a subject in a study during the entire study period, whether or not the event is expected or associated with the vaccine, is considered an SAE.

#### 12.3.3. HIV Infection

Human immunodeficiency virus testing will be carried out at times indicated in the Time and Events Schedule. Subjects will be tested for HIV infection at screening and baseline, and must be negative to be entered into the study. If possible, the site should select an assay that is US FDA-approved. At all other main study visits that include HIV-testing, a study-specific HIV testing algorithm (as described in the Laboratory Manual) will be followed. During the optional LTE phase, the study-specific HIV-testing algorithm described above will be followed as long as treatment assignment is blinded. Upon study unblinding, unblinded HIV and VISP results will be reported.

Any subject with confirmed HIV infection must be discontinued from any further study vaccine administration, but should remain in the study and be followed up for safety and immunogenicity until the end of the study.

Confirmed HIV infection in a subject during the study is considered an AESI. All AESIs, irrespective if considered serious or not by the investigator, shall be reported to the sponsor immediately (see Section 12.2). An aggregate analysis will be performed either at the end of study and possible at interim time points during the study.

Test results performed to confirm the diagnosis will be forwarded to the study staff. Subjects who become HIV infected during the study, including the optional LTE phase, will be (see Section 9.4.2):

- Excluded from further vaccinations.
- Provided counseling and referred for medical treatment.
- Informed about observational studies monitoring subjects with HIV infection.
- Excluded from initiation of the optional LTE phase

## 12.3.4. Pregnancy

All initial reports of pregnancy in female subjects or partners of male subjects must be reported to the sponsor by the study-site personnel within 24 hours of their knowledge of the event using the appropriate pregnancy notification form. Abnormal pregnancy outcomes (eg, spontaneous abortion, fetal death, stillbirth, congenital anomalies, ectopic pregnancy) are considered SAEs and

must be reported using the SAE Form. Any subject who becomes pregnant during the study must promptly discontinue further vaccinations, but should continue participation in the study for follow-up (see Section 10.2).

Because the effect of the study vaccine on sperm is unknown, pregnancies in partners of male subjects included in the study will be reported as noted above.

Follow-up information regarding the outcome of the pregnancy and any postnatal sequelae in the infant will be required to be sent to the sponsor.

# 12.4. Contacting Sponsor Regarding Safety

The names (and corresponding telephone numbers) of the individuals who should be contacted regarding safety issues or questions regarding the study are listed in the Contact Information page(s), which will be provided as a separate document.

#### 13. PRODUCT QUALITY COMPLAINT HANDLING

A product quality complaint (PQC) is defined as any suspicion of a product defect related to manufacturing, labeling, or packaging, ie, any dissatisfaction relative to the identity, quality, durability, or reliability of a product, including its labeling or package integrity. A PQC may have an impact on the safety and efficacy of the product. Timely, accurate, and complete reporting and analysis of PQC information from studies are crucial for the protection of subjects, investigators, and the sponsor, and are mandated by regulatory agencies worldwide. The sponsor has established procedures in conformity with regulatory requirements worldwide to ensure appropriate reporting of PQC information; all studies conducted by the sponsor or its affiliates will be conducted in accordance with those procedures.

#### 13.1. Procedures

All initial PQCs must be reported to the sponsor by the study-site personnel within 24 hours after being made aware of the event.

If the defect is combined with an SAE, the study-site personnel must report the PQC to the sponsor according to the SAE reporting timelines (see Section 12.3.2). A sample of the suspected product should be maintained for further investigation if requested by the sponsor.

## 13.2. Contacting Sponsor Regarding Product Quality

The names (and corresponding telephone numbers) of the individuals who should be contacted regarding product quality issues are listed in the Contact Information page(s), which will be provided as a separate document.

70

## 14. VACCINE INFORMATION

# 14.1. Physical Description of Study Vaccines

The Ad26.Mos4.HIV, Ad26.Mos.HIV, and Clade C gp140 supplied for this study are formulated as:

#### Ad26.Mos4.HIV

Ad26.Mos4.HIV is a tetravalent vaccine containing the following 4 active pharmaceutical ingredients pre-mixed in a 1:1:1:1 vp ratio:

- Ad26.Mos1.Gag-Pol recombinant, replication-incompetent Ad26 encoding for Mosaic 1 (Mos1) HIV-1 Gag and Pol proteins, manufactured in PER.C6® cells (JNJ-55471494-AAA).
- Ad26.Mos2.Gag-Pol recombinant, replication-incompetent Ad26 encoding Mosaic 2 (Mos2) HIV-1 Gag and Pol proteins, manufactured in PER.C6® cells (JNJ-55471520-AAA).
- Ad26.Mos1.Env recombinant, replication-incompetent Ad26 encoding Mos1 HIV-1 Env protein, manufactured in PER.C6<sup>®</sup> cells (JNJ-55471468-AAA).
- Ad26.Mos2S.Env recombinant, replication-incompetent Ad26 encoding modified (substitute, S) Mos2 HIV-1 Env protein, manufactured in PER.C6® cells (JNJ-64219324-AAA).

The Ad26.Mos4.HIV vaccine is formulated as a tetravalent vaccine, as a clear to slightly opalescent solution for IM injection. The vaccine will be supplied as a frozen liquid to be thawed prior to use, and will be practically free from particles. The vaccine will be provided in individual dosage vials at a concentration of  $1x10^{11}$  vp/mL. Refer to the Investigator's Brochure for a list of excipients.  $^{12}$ 

#### Ad26.Mos.HIV

Ad26.Mos.HIV is a trivalent vaccine containing the following 3 active pharmaceutical ingredients pre-mixed in a 1:1:2 vp ratio:

- Ad26.Mos1.Gag-Pol recombinant, replication-incompetent Ad26 encoding Mos1 HIV-1 Gag and Pol proteins, manufactured in PER.C6® cells (JNJ-55471494-AAA).
- Ad26.Mos2.Gag-Pol recombinant, replication-incompetent Ad26 encoding Mos2 HIV-1 Gag and Pol proteins, manufactured in PER.C6® cells (JNJ-55471520-AAA).
- Ad26.Mos1.Env recombinant, replication-incompetent Ad26 encoding Mos1 HIV-1 Env protein, manufactured in PER.C6® cells (JNJ-55471468-AAA).

The Ad26.Mos.HIV vaccine is formulated as a trivalent vaccine as a clear to slightly opalescent solution for IM injection. The vaccine will be supplied as a frozen liquid to be thawed prior to use, and will be essentially free from particles. The vaccine will be provided in individual dosage vials at a concentration of  $1x10^{11}$  vp/mL. Refer to the Investigator's Brochure for a list of excipients. <sup>12</sup>

Ad26.Mos4.HIV and Ad26.Mos.HIV are classified as genetically modified organisms (GMOs). Based on nonclinical biodistribution and shedding data with related vectors, the investigational vaccine is not expected to pose any risk to the environment. Any local requirements related to GMOs must be fulfilled by the investigator.

## Clade C gp140

Clade C gp140 is a monovalent vaccine containing the following pharmaceutical ingredient:

• Clade C gp140 Drug Substance is a trimeric, recombinant HIV-1 Env gp140 of Clade C, produced on a PER.C6® cell line. Aluminum phosphate suspension is used as adjuvant (JNJ-55471585-AAA: Clade C gp140 + aluminum phosphate adjuvant).

Clade C gp140 is formulated as a colorless to slightly yellowish/brownish solution for IM injection. Clade C gp140 will be supplied as a frozen liquid to be thawed prior to use, and will be practically free from particles. Clade C gp140 will be supplied at a nominal strength of either 1 mg/mL or 0.2 mg/mL. Refer to the Investigator's Brochure for a list of excipients. The aluminum phosphate adjuvant will be supplied as a formulated refrigerated liquid suspension with a nominal aluminum content of 1.7 mg/mL. It will be mixed with Clade C gp140 at the site pharmacy prior to administration.

#### Placebo

Placebo consisting of sterile 0.9% Saline for Injection will be supplied (as commercially available).

Study vaccines will be manufactured and provided under the responsibility of the sponsor.

## 14.2. Packaging and Labeling

All study vaccines were manufactured and packaged in accordance with Current Good Manufacturing Practice (GMP). All study vaccines will be packaged and labeled under the responsibility of the sponsor.

No study vaccine can be repacked or relabeled without prior approval from the sponsor.

Further details for study vaccine packaging and labeling can be found in the Site Investigational Product Procedures Manual.

## 14.3. Preparation, Handling, and Storage

Refer to the Site Investigational Product Procedures Manual for guidance on study vaccine preparation, handling, and storage.

Study vaccine must be stored in a secured location at controlled temperature with no access for unauthorized personnel. The study freezer must be equipped with a continuous temperature monitor and alarm. Study freezers should be equipped with back-up power systems. In the event that study vaccine is exposed to temperatures outside the specified temperature ranges, all relevant data will be sent to the sponsor to determine if the affected study vaccine can be used or will be
replaced. The affected study vaccine must be quarantined and not used until further instruction from the sponsor is received.

All injections should be administered in the deltoid. For visits with only one injection, preferably the deltoid of the non-dominant upper arm is used. When 2 study vaccine injections are to be given at one visit, it is required to use a different deltoid for each injection. Exceptions on injection site are allowed only if medically indicated. No local or topical anesthetic will be used prior to the injection. To account for the product with the shortest stability time, the maximum time allowed between preparation and administration of the study vaccine will be 3 hours.

A site pharmacist will prepare all doses for administration and will provide it to the clinic. In order to preserve blinding, the pharmacist will place an overlay on the syringes.

# 14.4. Vaccine Accountability

The investigator is responsible for ensuring that all study vaccine received at the site is inventoried and accounted for throughout the study. The study vaccine administered to the subject must be documented on the vaccine accountability form. All study vaccine will be stored and disposed of according to the sponsor's instructions.

Study vaccine must be handled in strict accordance with the protocol and the container label, and must be stored at the study site in a limited-access area or in a locked cabinet under appropriate environmental conditions. Unused study vaccine must be available for verification by the sponsor's study site monitor during on-site monitoring visits. The return to the sponsor of unused study vaccine will be documented on the vaccine return form. When the study site is an authorized destruction unit and study vaccine supplies are destroyed on-site, this must also be documented on the vaccine return form.

Potentially hazardous materials such as used ampules, needles, syringes and vials containing hazardous liquids, should be disposed of immediately in a safe manner and therefore will not be retained for accountability purposes.

Study vaccine should be dispensed under the supervision of the investigator or a qualified member of the study-site personnel, or by a hospital/clinic pharmacist. Study vaccine will be supplied only to subjects participating in the study. Study vaccine may not be relabeled or reassigned for use by other subjects. The investigator agrees neither to dispense the study vaccine from, nor store it at, any site other than the study sites agreed upon with the sponsor.

## 15. STUDY-SPECIFIC MATERIALS

The investigator will be provided with the following supplies:

- Investigator's Brochure for Ad26.Mos.HIV and Clade C gp140
- Laboratory Manual, Study Procedures Manual
- IWRS Manual

- Electronic Data Capturing (eDC) Manual/electronic CRF completion guidelines and randomization instructions
- Sample ICF
- Subject diary
- Test of Understanding
- Social Impact Questionnaire
- Ruler (to measure diameter of any erythema and induration/swelling), thermometer
- Subject wallet cards
- Recruitment tools, as applicable

#### 16. ETHICAL ASPECTS

# 16.1. Study-specific Design Considerations

Potential subjects will be fully informed of the risks and requirements of the study and, during the study, subjects will be given any new information that may affect their decision to continue participation. They will be told that their consent to participate in the study is voluntary and may be withdrawn at any time with no reason given and without penalty or loss of benefits to which they would otherwise be entitled. Only subjects who are fully able to understand the risks, benefits, and potential AEs of the study, and provide their consent voluntarily will be enrolled.

From screening to the final main study visit at Week 72, the total blood volume to be collected from each subject will be approximately 1,200 mL. The total blood volume to be collected during the optional LTE phase (Group 2A only) will be approximately 470 mL over a 3-year period or 628 mL over a 4-year period. The total blood volume to be collected is considered to be within the US Department of HHS OHRP, and US FDA guidelines of 550 mL in any 8-week period. Daily volumes for humoral immunogenicity testing will be approximately 20 mL/visit and for cellular immunogenicity testing approximately 50-102 mL/visit during the main study and 50 mL/visit during the optional LTE phase.

#### **Test of Understanding**

The TOU is a short assessment of the subject's understanding of key aspects of the study. The test will help the study staff to determine how well subjects understand the study and their requirements for participation.

The TOU must be completed by all subjects, as the first assessment after signing of the ICF. The TOU is reviewed one-on-one with the subjects and a member of the study team. Subjects are allowed to retake the test as many times as necessary to achieve the passing score (≥90%) required for participation in the study. If a subject fails to achieve the passing score, further information and counseling will be provided by the study team member.

Any subject not capable of understanding the key aspects of the study, and their requirements for participation, should not be enrolled.

#### **Risks Related to Aluminum**

Aluminum is one of the most common metals found in nature and is present in air, food, and water. Aluminum salts, such as aluminum phosphate have been used safely in vaccines for more than 70 years. Aluminum-containing vaccines have been associated with severe local reactions, such as redness, lumps under the skin, contact allergy or irritation, and swelling at the site of injection. There have also been reports, especially in patients with impaired renal function, of systemic accumulation of aluminum, which has been associated with nervous disorders and bone disease. Nonetheless, aluminum intake from vaccines is far less than that received from the diet or medications such as antacids.<sup>4,14</sup>

#### **Risks Related to Vaccines**

Subjects may exhibit general signs and symptoms associated with administration of a vaccine, or vaccination with placebo, including fever, chills, rash, aches and pains, nausea, headache, dizziness and fatigue. These side effects will be monitored, but are generally short-term and do not require treatment.

Subjects may have an allergic reaction to the vaccination. An allergic reaction may cause a rash, hives or even difficulty breathing. Severe reactions are rare. Medications must be available in the clinic to treat serious allergic reactions.

The effect of this vaccine on a fetus or nursing baby is unknown, as well as the effect on semen, so female subjects of child bearing potential, and male subjects having sexual intercourse with females, will be required to agree to use birth control for sexual intercourse beginning prior to the first vaccination and through 3 months after the last vaccination. Women who are pregnant or nursing will be excluded from the main study.

Risks related to VISP are discussed in Section 9.4.3.

#### **Risks from Blood Draws**

Blood drawing may cause pain, bruising, and, rarely, infection at the site where the blood is taken.

#### **Risks from HLA Testing**

Tests results can be used to provide information about how susceptible subjects are to certain diseases. Used inappropriately, this information could be discriminatory (for example, by insurance companies). Human Leukocyte Antigen typing can also be used to determine paternity. However, the blood samples donated will not be used for this purpose; they will be used only to provide study investigators information about the immune system. The results will be coded to protect subject identity.

#### **Unknown Risks**

There may be other serious risks that are not known.

Subjects may believe that this vaccine provides protection against acquiring HIV infection, and therefore practice riskier behavior. They will receive extensive counseling throughout the study to address this potential problem. It is not known if the study vaccines increase or decrease the chance of becoming HIV infected when exposed, or if upon becoming HIV infected, the person's disease course progresses faster or slower to AIDS.

In previous HIV-efficacy studies utilizing Ad5, a trend towards increased HIV-1 infection was observed in vaccine recipients as compared with placebo recipients. Adenovirus serotype 26 is biologically substantially different than Ad5 and Ad26-based vaccines afford superior protective efficacy compared with Ad5-based vaccines against SIV<sub>MAC251</sub> challenges in rhesus monkeys. Further, Ad26 did not increase the number or activation status of total or vector-specific CD4<sup>+</sup> T-lymphocytes at mucosal surfaces in humans following vaccination in a randomized, double-blind, placebo-controlled clinical study.

#### **Potential Benefits**

There is no direct medical benefit to the subject for participation in this clinical study. Although study subjects may benefit from clinical testing and physical examination, they may receive no direct benefit from participation. Others may benefit from knowledge gained in this study that may aid in the development of an HIV vaccine.

# 16.2. Regulatory Ethics Compliance

# 16.2.1. Investigator Responsibilities

The investigator is responsible for ensuring that the study is performed in accordance with the protocol, current ICH guidelines on Good Clinical Practice (GCP), and applicable regulatory and country-specific requirements.

Good Clinical Practice is an international ethical and scientific quality standard for designing, conducting, recording, and reporting studies that involve the participation of human subjects. Compliance with this standard provides public assurance that the rights, safety, and well-being of study subjects are protected, consistent with the principles that originated in the Declaration of Helsinki, and that the study data are credible.

# 16.2.2. Independent Ethics Committee or Institutional Review Board

Before the start of the study, the investigator (or sponsor where required) will provide the IEC/IRB with current and complete copies of the following documents (as required by local regulations):

- Final protocol and, if applicable, amendments
- Sponsor-approved ICF (and any other written materials to be provided to the subjects)
- Investigator's Brochure (or equivalent information) and amendments/addenda
- Sponsor-approved subject recruiting materials
- Information on compensation for study-related injuries or payment to subjects for participation in the study, if applicable

- Investigator's curriculum vitae or equivalent information (unless not required, as documented by the IEC/IRB)
- Information regarding funding, name of the sponsor, institutional affiliations, other potential conflicts of interest, and incentives for subjects
- Any other documents that the IEC/IRB requests to fulfill its obligation

This study will be undertaken only after the IEC/IRB has given full approval of the final protocol, amendments (if any, excluding the ones that are purely administrative, with no consequences for subjects, data or study conduct, unless required locally), the ICF, applicable recruiting materials, and subject compensation programs, and the sponsor has received a copy of this approval. This approval letter must be dated and must clearly identify the IEC/IRB and the documents being approved.

During the study the investigator (or sponsor where required) will send the following documents and updates to the IEC/IRB for their review and approval, where appropriate:

- Protocol amendments (excluding the ones that are purely administrative, with no consequences for subjects, data or study conduct)
- Revision(s) to ICF and any other written materials to be provided to subjects
- If applicable, new or revised subject recruiting materials approved by the sponsor
- Revisions to compensation for study-related injuries or payment to subjects for participation in the study, if applicable
- New edition(s) of the Investigator's Brochure and amendments/addenda
- Summaries of the status of the study at intervals stipulated in guidelines of the IEC/IRB (at least annually)
- Reports of AEs that are serious, unlisted/unexpected, and associated with the vaccine
- New information that may adversely affect the safety of the subjects or the conduct of the study
- Deviations from or changes to the protocol to eliminate immediate hazards to the subjects
- Report of deaths of subjects under the investigator's care
- Notification if a new investigator is responsible for the study at the site
- Development Safety Update Report and Line Listings, where applicable
- Any other requirements of the IEC/IRB

For all protocol amendments (excluding the ones that are purely administrative, with no consequences for subjects, data or study conduct), the amendment and applicable ICF revisions must be submitted promptly to the IEC/IRB for review and approval before implementation of the change(s).

At least once a year, the IEC/IRB will be asked to review and reapprove this study, where required. At the end of the study, the investigator (or sponsor where required) will notify the IEC/IRB about the study completion.

### 16.2.3. Informed Consent

Each subject must give written consent according to local requirements after the nature of the study has been fully explained. The ICF must be signed before performance of any study-related activity. The ICF that is used must be approved by both the sponsor and by the reviewing IEC/IRB and be in a language that the subject can read and understand. The informed consent should be in accordance with principles that originated in the Declaration of Helsinki, current ICH and GCP guidelines, applicable regulatory requirements, and sponsor policy.

Before enrollment in the study, the investigator or an authorized member of the study-site personnel must explain to potential subjects the aims, methods, reasonably anticipated benefits, and potential hazards of the study, and any discomfort participation in the study may entail. Subjects will be informed that their participation is voluntary and that they may withdraw consent to participate at any time. They will be informed that choosing not to participate will not affect the care the subject will receive. Finally, they will be told that the investigator will maintain a subject identification register for the purposes of long-term follow-up if needed and that their records may be accessed by health authorities and authorized sponsor personnel without violating the confidentiality of the subject, to the extent permitted by the applicable law(s) or regulations. By signing the ICF the subject is authorizing such access, which includes permission to obtain information about his or her survival status if applicable. It also denotes that the subject agrees to allow his or her study physician to recontact the subject for the purpose of obtaining consent for additional safety evaluations and subsequent disease-related treatment, if needed.

The subject will be given sufficient time to read the ICF and the opportunity to ask questions. After this explanation and before entry into the study, consent should be appropriately recorded by means of the subject's personally dated signature. After having obtained the consent, a copy of the ICF must be given to the subject.

If the subject is unable to read or write, an impartial witness should be present for the entire informed consent process (which includes reading and explaining all written information) and should personally date and sign the ICF after the oral consent of the subject is obtained.

For participation in the optional 3-year LTE phase of the study, an ICF appendix will be available. Upon sponsor unblinding at the Week 28 analysis, subjects randomized to Group 2A who have received all 4 vaccinations, will be asked to participate in the optional LTE phase and sign the ICF appendix for the optional LTE phase at Week 72. Subjects who attend their Week 72 visit prior to the sponsor's unblinding at the Week 28 analysis, will be enrolled in the optional LTE phase if they consent and sign the ICF appendix for the optional LTE phase and meet the eligibility criteria for the optional LTE phase. When the Week 28 sponsor unblinding subsequently occurs, subjects that started the optional LTE phase but turn out not to be in Group 2A of the main study will be withdrawn from the optional LTE phase. If signing the ICF appendix is not possible at Week 72,

signing should be performed at an extra visit (Visit 17bis) as soon as possible after Week 72 and at the latest before any assessment is done on the first visit of the optional LTE phase.

An optional 2-year extension of this 3-year optional LTE is introduced in protocol amendment 3. Subjects will be informed of the option to participate in this 2-year extension at the next possible visit after approval of this amendment. Subjects willing to participate will need to sign the ICF appendix for the 2-year extension at Visit 23. Subjects not willing to participate in the 2-year extension will have their final study visit at Visit 23. In protocol amendment 5, this 2-year extension was shortened to 1 year. Subject willing to participate will have their final visit at Visit 25. Participants who already had their Visit 25 or Visit 26 will be contacted to perform an extra unscheduled exit visit, to be performed within 6 weeks after local approval of protocol amendment 5.

# 16.2.4. Privacy of Personal Data

The collection and processing of personal data from subjects enrolled in this study will be limited to those data that are necessary to fulfill the objectives of the study.

These data must be collected and processed with adequate precautions to ensure confidentiality and compliance with applicable data privacy protection laws and regulations. Appropriate technical and organizational measures to protect the personal data against unauthorized disclosures or access, accidental or unlawful destruction, or accidental loss or alteration must be put in place. Sponsor personnel whose responsibilities require access to personal data agree to keep the identity of subjects confidential.

The informed consent obtained from the subject includes explicit consent for the processing of personal data and for the investigator/institution to allow direct access to his or her original medical records (source data/documents) for study-related monitoring, audit, IEC/IRB review, and regulatory inspection. This consent also addresses the transfer of the data to other entities and to other countries.

The subject has the right to request through the investigator access to his or her personal data and the right to request rectification of any data that are not correct or complete. Reasonable steps will be taken to respond to such a request, taking into consideration the nature of the request, the conditions of the study, and the applicable laws and regulations.

Exploratory DNA, immunogenicity, and social impact questionnaire research is not conducted under standards appropriate for the return of data to subjects. In addition, the sponsor cannot make decisions as to the significance of any findings resulting from exploratory research. Therefore, exploratory research data will not be returned to subjects or investigators, unless required by law or local regulations. Privacy and confidentiality of data generated in the future on stored samples will be protected by the same standards applicable to all other clinical data.

### 16.2.5. Long-term Retention of Samples for Additional Future Research

Each study subject will be asked to consent voluntarily for their blood samples to be stored for other research studies that may be done after this study is completed. Future testing may involve

deoxyribonucleic acid (DNA)/RNA tests. For subjects unwilling to have their blood samples stored for future use, they can consent to participate in this study only, without having their blood samples stored for future testing (see Section 10.5). In this case, their blood samples will be destroyed after all the tests specified for this study have been concluded.

All samples, for which consent has been obtained and for which additional material is available after study-specified testing is complete, will be stored for future testing. All applicable approvals will be sought before any such samples are used for analysis not specified in the protocol or a protocol amendment approved by the IRB.

Stored samples will be coded throughout the sample storage and analysis process and will not be labeled with personal identifiers. Subjects may withdraw their consent for their samples to be stored for research (see Section 10.5).

#### 17. ADMINISTRATIVE REQUIREMENTS

#### 17.1. Protocol Amendments

Neither the investigator nor the sponsor will modify this protocol without a formal amendment by the sponsor. All protocol amendments must be issued by the sponsor, and signed and dated by the investigator. Protocol amendments must not be implemented without prior IEC/IRB approval, or when the relevant competent authority has raised any grounds for non-acceptance, except when necessary to eliminate immediate hazards to the subjects, in which case the amendment must be promptly submitted to the IEC/IRB and relevant competent authority. Documentation of amendment approval by the investigator and IEC/IRB must be provided to the sponsor. When the change(s) involves only logistic or administrative aspects of the study, the IRB/IEC (where required) only needs to be notified.

During the course of the study, in situations where a departure from the protocol is unavoidable, the investigator or other physician in attendance will contact the appropriate sponsor representative (listed in the Contact Information page(s), which will be provided as a separate document). Except in emergency situations, this contact should be made <u>before</u> implementing any departure from the protocol. In all cases, contact with the sponsor must be made as soon as possible to discuss the situation and agree on an appropriate course of action. The data recorded in the CRF and source documents will reflect any departure from the protocol, and the source documents will describe this departure and the circumstances requiring it.

# 17.2. Regulatory Documentation

# 17.2.1. Regulatory Approval/Notification

This protocol and any amendment(s) must be submitted to the appropriate regulatory authorities in each respective country, if applicable. A study may not be initiated until all local regulatory requirements are met.

# 17.2.2. Required Prestudy Documentation

The following documents must be provided to the sponsor before shipment of vaccine to the study site:

- Protocol and amendment(s), if any, signed and dated by the principal investigator
- A copy of the dated and signed (or sealed, where appropriate per local regulations), written IEC/IRB approval of the protocol, amendments, ICF, any recruiting materials, and if applicable, subject compensation programs. This approval must clearly identify the specific protocol by title and number and must be signed (or sealed, where appropriate per local regulations) by the chairman or authorized designee.
- Name and address of the IEC/IRB, including a current list of the IEC/IRB members and their function, with a statement that it is organized and operates according to GCP and the applicable laws and regulations. If accompanied by a letter of explanation, or equivalent, from the IEC/IRB, a general statement may be substituted for this list. If an investigator or a member of the study-site personnel is a member of the IEC/IRB, documentation must be obtained to state that this person did not participate in the deliberations or in the vote/opinion of the study.
- Regulatory authority approval or notification, if applicable
- Signed and dated statement of investigator (eg, Form FDA 1572), if applicable
- Documentation of investigator qualifications (eg, curriculum vitae)
- Completed investigator financial disclosure form from the principal investigator, where required
- Signed and dated clinical trial agreement, which includes the financial agreement
- Any other documentation required by local regulations

The following documents must be provided to the sponsor before enrollment of the first subject:

- Completed investigator financial disclosure forms from all subinvestigators
- Documentation of subinvestigator qualifications (eg, curriculum vitae)
- Name and address of any local laboratory conducting tests for the study, and a dated copy of current laboratory normal ranges for these tests, if applicable
- Local laboratory documentation demonstrating competence and test reliability (eg, accreditation/license), if applicable

# 17.3. Subject Identification, Enrollment, and Screening Logs

The investigator agrees to complete a subject identification and enrollment log to permit easy identification of each subject during and after the study. This document will be reviewed by the sponsor study-site contact for completeness.

The subject identification and enrollment log will be treated as confidential and will be filed by the investigator in the study file. To ensure subject confidentiality, no copy will be made. All reports and communications relating to the study will identify subjects by subject identification and date of birth. In cases where the subject is not randomized into the study, the date seen and date of birth will be used.

The investigator must also complete a subject screening log, which reports on all subjects who were seen to determine eligibility for inclusion in the study.

#### 17.4. Source Documentation

At a minimum, source documents consistent in the type and level of detail with that commonly recorded at the study site as a basis for standard medical care, must be available for the following: subject identification, eligibility, and study identification; study discussion and date of signed informed consent; dates of visits; results of safety parameters as required by the protocol; record of all AEs and follow-up of AEs; concomitant medication; vaccine receipt/dispensing/return records; vaccine administration information; and date of study completion and reason for early discontinuation of vaccine or withdrawal from the study, if applicable.

The author of an entry in the source documents should be identifiable.

Specific details required as source data for the study and source data collection methods will be reviewed with the investigator before the study and will be described in the monitoring guidelines (or other equivalent document).

An eSource system may be utilized, which contains data traditionally maintained in a hospital or clinic record to document medical care (eg, electronic source documents) as well as the clinical study-specific data fields as determined by the protocol. This data is electronically extracted for use by the sponsor. If eSource is utilized, references made to the CRF in the protocol include the eSource system but information collected through eSource may not be limited to that found in the CRF.

The subject's diary used to collect information regarding solicited events after vaccination will be considered source data.

## 17.5. Case Report Form Completion

Case report forms are prepared and provided by the sponsor for each subject in electronic format. All CRF entries, corrections, and alterations must be made by the investigator or authorized study-site personnel. The investigator must verify that all data entries in the CRF are accurate and correct.

The study data will be transcribed by study-site personnel from the source documents onto an electronic CRF, if applicable. Study-specific data will be transmitted in a secure manner to the sponsor.

Worksheets may be used for the capture of some data to facilitate completion of the CRF. Any such worksheets will become part of the subject's source documents. Data must be entered into CRF in English. The CRF must be completed as soon as possible after a subject visit and the forms should be available for review at the next scheduled monitoring visit.

All subjective measurements (eg, questionnaires) will be completed by the same individual who made the initial baseline determinations whenever possible.

If necessary, queries will be generated in the eDC tool. If corrections to a CRF are needed after the initial entry into the CRF, this can be done in either of the following ways:

- Investigator and study-site personnel can make corrections in the eDC tool at their own initiative or as a response to an auto query (generated by the eDC tool).
- Sponsor or sponsor delegate can generate a query for resolution by the investigator and study-site personnel.

# 17.6. Data Quality Assurance/Quality Control

Steps to be taken to ensure the accuracy and reliability of data include the selection of qualified investigators and appropriate study sites, review of protocol procedures with the investigator and study-site personnel before the study, and periodic monitoring visits by the sponsor. Written instructions will be provided for collection, handling, storage, and shipment of samples.

Guidelines for CRF completion will be provided and reviewed with study-site personnel before the start of the study.

The sponsor will review CRFs for accuracy and completeness during on-site monitoring visits and after transmission to the sponsor; any discrepancies will be resolved with the investigator or designee, as appropriate. After upload of the data into the study database they will be verified for accuracy and consistency with the data sources.

#### 17.7. Record Retention

In compliance with the ICH/GCP guidelines, the investigator/institution will maintain all CRF and all source documents that support the data collected from each subject, as well as all study documents as specified in ICH/GCP Section 8, Essential Documents for the Conduct of a Clinical Trial, and all study documents as specified by the applicable regulatory requirement(s). The investigator/institution will take measures to prevent accidental or premature destruction of these documents.

Essential documents must be retained until at least 2 years after the last approval of a marketing application in an ICH region and until there are no pending or contemplated marketing applications in an ICH region or until at least 2 years have elapsed since the formal discontinuation of clinical development of the investigational product. These documents will be retained for a longer period if required by the applicable regulatory requirements or by an agreement with the sponsor. It is the responsibility of the sponsor to inform the investigator/institution as to when these documents no longer need to be retained.

If the responsible investigator retires, relocates, or for other reasons withdraws from the responsibility of keeping the study records, custody must be transferred to a person who will accept the responsibility. The sponsor must be notified in writing of the name and address of the new

custodian. Under no circumstance shall the investigator relocate or dispose of any study documents before having obtained written approval from the sponsor.

If it becomes necessary for the sponsor or the appropriate regulatory authority to review any documentation relating to this study, the investigator/institution must permit access to such reports.

# 17.8. Monitoring

The sponsor may use a combination of monitoring techniques: central, remote, or on-site monitoring to monitor this study.

The sponsor will ensure on-site monitoring visits as frequently as necessary. The monitor will record dates of the visits in a study site visit log that will be kept at the study site. The first post-initiation visit will be made as soon as possible after enrollment has begun. At these visits, the monitor will compare the data entered into the CRF with the source documents (eg, hospital/clinic/physician's office medical records); a sample may be reviewed. The nature and location of all source documents will be identified to ensure that all sources of original data required to complete the CRF are known to the sponsor and study-site personnel and are accessible for verification by the sponsor study-site contact. If electronic records are maintained at the study site, the method of verification must be discussed with the study-site personnel.

Direct access to source documents (medical records) must be allowed for the purpose of verifying that the recorded data are consistent with the original source data. Findings from this review will be discussed with the study-site personnel. The sponsor expects that, during monitoring visits, the relevant study-site personnel will be available, the source documents will be accessible, and a suitable environment will be provided for review of study-related documents. The monitor will meet with the investigator on a regular basis during the study to provide feedback on the study conduct.

In addition to on-site monitoring visits, remote contacts can occur. It is expected that during these remote contacts, study-site personnel will be available to provide an update on the progress of the study at the site.

Central monitoring will take place for data identified by the sponsor as requiring central review.

### 17.9. Study Completion/Termination

# 17.9.1. Study Completion/End of Study

The study is considered completed with the last visit for the last subject participating in the study. The final data from the study site will be sent to the sponsor (or designee) after completion of the final subject visit at that study site, in the time frame specified in the Clinical Trial Agreement.

### 17.9.2. Study Termination

The sponsor reserves the right to close the study site or terminate the study at any time for any reason at the sole discretion of the sponsor. Study sites will be closed upon study completion. A

study site is considered closed when all required documents and study supplies have been collected and a study-site closure visit has been performed.

The investigator may initiate study-site closure at any time, provided there is reasonable cause and sufficient notice is given in advance of the intended termination.

Reasons for the early closure of a study site by the sponsor or investigator may include but are not limited to:

- Failure of the investigator to comply with the protocol, the requirements of the IEC/IRB or local health authorities, the sponsor's procedures, or GCP guidelines
- Inadequate recruitment of subjects by the investigator
- Discontinuation of further vaccine development

#### 17.10. On-Site Audits

Representatives of the sponsor's clinical quality assurance department may visit the study site at any time during or after completion of the study to conduct an audit of the study in compliance with regulatory guidelines and company policy. These audits will require access to all study records, including source documents, for inspection. Subject privacy must, however, be respected. The investigator and study-site personnel are responsible for being present and available for consultation during routinely scheduled study-site audit visits conducted by the sponsor or its designees.

Similar auditing procedures may also be conducted by agents of any regulatory body, either as part of a national GCP compliance program or to review the results of this study in support of a regulatory submission. The investigator should immediately notify the sponsor if he or she has been contacted by a regulatory agency concerning an upcoming inspection.

### 17.11. Use of Information and Publication

All information, including but not limited to information regarding Ad26.Mos4.HIV, Ad26.Mos.HIV, and Clade C gp140 or the sponsor's operations (eg, patent application, formulas, manufacturing processes, basic scientific data, prior clinical data, formulation information) supplied by the sponsor to the investigator and not previously published, and any data generated as a result of this study, are considered confidential and remain the sole property of the sponsor and/or its partners. The investigator agrees to maintain this information in confidence and use this information only to accomplish this study, and will not use it for other purposes without the sponsor's prior written consent.

The investigator understands that the information developed in the study will be used by the sponsor in connection with the continued development of Ad26.Mos4.HIV, Ad26.Mos.HIV, and Clade C gp140, and thus may be disclosed as required to other clinical investigators or regulatory agencies. To permit the information derived from the clinical studies to be used, the investigator is obligated to provide the sponsor with all data obtained in the study.

The results of the study will be reported in a Clinical Study Report generated by the sponsor and will contain data from all study sites that participated in the study as per protocol. Recruitment performance or specific expertise related to the nature and the key assessment parameters of the study will be used to determine a coordinating investigator. Results of any analyses performed after the Clinical Study Report has been issued will be reported in a separate report and will not require a revision of the Clinical Study Report. Study subject identifiers will not be used in publication of results. Any work created in connection with performance of the study and contained in the data that can benefit from copyright protection (except any publication by the investigator as provided for below) shall be the property of the sponsor as author and owner of copyright in such work.

Consistent with Good Publication Practices and International Committee of Medical Journal Editors guidelines, the sponsor with its partners shall have the right to publish such primary (multicenter) data and information without approval from the investigator. The investigator has the right to publish study site-specific data after the primary data are published. If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. Expedited reviews will be arranged for abstracts, poster presentations, or other materials. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application. In the event that issues arise regarding scientific integrity or regulatory compliance, the sponsor will review these issues with the investigator. The sponsor will not mandate modifications to scientific content and does not have the right to suppress information. For multicenter study designs and substudy approaches, secondary results generally should not be published before the primary endpoints of a study have been published. Similarly, investigators will recognize the integrity of a multicenter study by not submitting for publication data derived from the individual study site until the combined results from the completed study have been submitted for publication, within 12 months of the availability of the final data (tables, listings, graphs), or the sponsor confirms there will be no multicenter study publication. Authorship of publications resulting from this study will be based on the guidelines on authorship, such as those described in the Uniform Requirements for Manuscripts Submitted to Biomedical Journals, which state that the named authors must have made a significant contribution to the design of the study or analysis and interpretation of the data, provided critical review of the paper, and given final approval of the final version.

### Registration of Clinical Studies and Disclosure of Results

The sponsor will register and disclose the existence of and the results of clinical studies as required by law.

# 18. COVID-19 APPENDIX: GUIDANCE ON STUDY CONDUCT DURING THE COVID-19 PANDEMIC

It is recognized that the Coronavirus Disease 2019 (COVID-19) pandemic may have an impact on the conduct of this clinical study due to, for example, self-isolation/quarantine by subjects and study-site personnel; travel restrictions/limited access to public places, including hospitals; study site personnel being reassigned to critical tasks.

In alignment with recent health authority guidance, the sponsor is providing options for study related subject management in the event of disruption to the conduct of the study. This guidance does not supersede any local or government requirements or the clinical judgement of the investigator to protect the health and well-being of subjects and site staff and to maintain oversight of delegated trial activities.

Scheduled visits that cannot be conducted in person at the study site will be performed to the extent possible as a remote visit, a home visit, or delayed until such time that on-site visits can be resumed.<sup>g</sup> At each contact, subjects will be interviewed to collect safety data. Key endpoint assessments should be performed if required and as feasible. Subjects will also be questioned regarding general health status to fulfill any physical examination requirement.

Every effort should be made to adhere to protocol-specified assessments. Modifications to protocol-required assessments may be permitted via COVID-19 Appendix after consultation with the subject, investigator, and the sponsor. Missed assessments/visits will be captured in the clinical trial management system for protocol deviations. Discontinuations of study interventions and withdrawal from the study should be documented with the prefix "COVID-19-related" in the case report form (CRF). Any deviations to study procedures occurring due to the COVID-19 pandemic need to be properly captured in the clinical trial management system (or CRF), with the prefix "COVID-19-related" (including actual visit date) and will be summarized in the clinical study report.

The sponsor will continue to monitor the conduct and progress of the clinical study, and any changes will be communicated to the sites and to the health authorities according to applicable guidance documents and regulations. If a subject has tested positive for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), the investigator should contact the sponsor's responsible medical officer to discuss plans for study intervention and follow-up. Modifications made to the study conduct as a result of the COVID-19 pandemic should be summarized in the clinical study report.

-

<sup>&</sup>lt;sup>g</sup> An on-site visit is defined as a visit during which the subject and the qualified site staff are both present in person at the study site.

A remote visit is defined as a visit during which there is no direct in-person physical presence between the subject and the qualified site staff (telephone or video call).

A home visit is defined as a visit during which the subject and the qualified site staff are both present at the subjects' home.

#### **GUIDANCE SPECIFIC TO THIS PROTOCOL:**

The following emergency provisions are meant to ensure subject safety on study while site capabilities are compromised by COVID-19-related restrictions. When restrictions are lifted, sites should revert to the original protocol conduct as soon as feasible and in accordance with local guidance and regulations and in agreement with the institutions and the investigator's assessment of the safety of site staff and study subjects.

#### **Study Visits and Assessments**

• Subjects may have remote visits for reactogenicity and safety assessments until such time that on-site visits can be resumed. The actual visit date should be captured in the eCRF according to the eCRF completion guidelines.

### Sample Management

• If a site is experiencing a disruption in shipment of specimens from their Site Processing Lab to the centralized HIV diagnostic testing laboratory(ies) due to the COVID-19 pandemic-related challenges, the Site Processing Lab should hold that specimen at the proper temperature for later per-protocol testing.

### **Informed Consent**

Consenting and re-consenting of subjects for the measures taken (including also remote
consenting by phone or video consultation) will be performed as applicable and according to
local guidance for informed consent applicable during the COVID-19 pandemic. The process
is to be documented in the source documents.

#### Source Data Verification/Monitoring

• In case on-site monitoring visits are not possible, the site monitor may contact the investigator to arrange monitoring visits and activities remotely (in accordance with site and local requirements). Additional on-site monitoring visits may be needed in the future to catch up on source data verification.

#### **Site Audits**

 During the COVID-19 pandemic and at the impacted sites, study site GCP audits with direct impact/engagement from the investigator and study site personnel may not be conducted in order to comply with national, local, and/or organizational social distancing restrictions. Additional quality assurance activities such as remote audits or focused review of study-related documents may take place with limited impact/engagement if possible.

#### **REFERENCES**

- 1. Barouch D, Alter G, Broge T, et al. Protective efficacy of adenovirus/protein vaccines against SIV challenges in rhesus monkeys. Science. 2015;349:320-324.
- Benlahrech A, Harris J, Meiser A, et al. Adenovirus vector vaccination induces expansion of memory CD4 T cells with a mucosal homing phenotype that are readily susceptible to HIV-1. Proc Natl Acad Sci USA. 2009; 106: 19940-19945.
- Buchbinder S, Mehrotra D, Duerr A, et al. Efficacy assessment of a cell-mediated immunity HIV-1 vaccine (the Step Study): a double-blind, randomized, placebo-controlled, test-of-concept trial. Lancet. 2008; 372: 1881-1893.
- 4. Eickhoff T, Myers M. Workshop summary. Aluminum in vaccines. Vaccine. 2002; 20 Suppl 3: S1-4.
- 5. Fischer W, Perkins S, Theiler J, et al. Polyvalent vaccines for optimal coverage of potential T-cell epitopes in global HIV-1 variants. Nat Med. 2007; 13: 100-106.
- 6. Gidudu JK, Walco GA, Taddio A, et al. The Brighton Immunization Site Pain Working Group. Immunization site pain: Case definition and guidelines for collection, analysis, and presentation of immunization safety data. http://www.sciencedirect.com/science/article/pii/S0264410X12005063. Accessed 11 June 2015.
- 7. Gray G, Allen M, Moodie Z, et al. Safety and efficacy of the HVTN 503/Phambili study of a clade-B-based HIV-1 vaccine in South Africa: a double-blind, randomized, placebo-controlled test-of-concept phase 2b study. Lancet Infect Dis. 2011; 11: 507-515.
- Hammer S, Sobieszczyk M, Karuna S, et al. Efficacy trial of a DNA/rAd5 HIV-1 preventive vaccine. N Engl J Med. 2013; 369: 2083-2092.
- 9. Huang Y, Follmann D, Nason M, et al. Effect of rAd5-vector HIV -1 preventive vaccines on HIV-1 acquisition: a participant-level meta-analysis of randomized trials. PloS One. 2015. DOI:10.1371.
- 10. Hutnick N, Carnathan D, Dubey S, et al. Baseline Ad5 serostatus does not predict Ad5 HIV vaccine-induced expansion of adenovirus-specific CD4+ T cells. Nat Med. 2009; 15: 876-878.
- 11. Information on Phase 1 clinical studies with monovalent AIDSVAX B conducted by Genentech. Available at http://www.vaxgen.com/hivaids/10k p8 (accessed: October 07, 2014).
- 12. Investigator's Brochure: Ad26.Mos.HIV-Ad26.Mos4.HIV. Edition 3. Crucell Holland BV (09 Dec 2015).
- 13. Investigator's Brochure: Clade C gp140 DP. Edition 2. Crucell Holland BV (06 Nov 2014).
- 14. Jefferson T, Rudin M, Di Pietrantonj C. Adverse events after immunisation with aluminium-containing DTP vaccines: systematic review of the evidence. Lancet Infect Dis. 2004; 4: 84-90.
- 15. Johnson & Johnson: Johnson & Johnson and Global Partners Announce Results from Phase 2b Imbokodo HIV Vaccine Clinical Trial in Young Women in Sub-Saharan Africa. August 31, 2021, News Release. Available at: https://www.jnj.com/johnson-johnson-and-global-partners-announce-results-from-phase-2b-imbokodo-hiv-vaccine-clinical-trial-in-young-women-in-sub-saharan-africa. Accessed: 20 October 2021.
- 16. Kohl KS, Walop W, Gidudu J, et al. The Brighton Collaboration Local Reaction Working Group for Swelling at or near Injection Site. Swelling at or near injection site: Case definition and guidelines for collection, analysis and presentation of immunization safety data. http://www.sciencedirect.com/science/article/pii/S0264410X07004835. Accessed 11 June 2015.
- 17. Kohl KS, Walop W, Gidudu J, et al. The Brighton Collaboration Local Reaction Working Group for Induration at or near Injection Site. Induration at or near injection site: Case definition and guidelines for collection, analysis and presentation of immunization safety data. http://www.sciencedirect.com/science/article/pii/S0264410X07005038. Accessed 11 June 2015.
- 18. Kovacs J, Nkolola J, Peng H, et al. HIV-1 envelope trimer elicits more potent neutralizing antibody responses than monomeric gp120. Proc Natl Acad Sci USA. 2012; 109: 12111-12116.
- 19. Marcy SM, Kohl KS, Dagan R, et al. The Brighton Collaboration Fever Working Group. Fever as an adverse event following immunization: case definition and guidelines of data collection, analysis, and presentation. http://www.sciencedirect.com/science/article/pii/S0264410X03006601. Accessed 11 June 2015.

- 20. Rerks-Ngarm S, Pitisuttithum P, Nitayaphan S, et al. Vaccination with ALVAC and AIDSVAX to prevent HIV-1 infection in Thailand. N Engl J Med. 2009; 361: 2209-2220.
- 21. Vella S. Addressing barriers to the end of AIDS by 2030. The Lancet. 2015;2:e360-e361.
- 22. Investigator's Brochure: Ad26.Mos.HIV Ad26.Mos4.HIV. Edition 7. Janssen Vaccines & Prevention B.V. (February 2020).
- 23. Investigator's Brochure: Clade C gp140 Mosaic gp140. Edition 7. Janssen Vaccines & Prevention B.V. (February 2020).

# Attachment 1: Division of Aids Table for Grading the Severity of Adult and Pediatric AEs – Including Modifications

The Division of AIDS Table for Grading the Severity of Adult and Pediatric AEs (Version 2.0, November 2014), or 'DAIDS grading table', is a descriptive terminology to be utilized for AE reporting in this study. A grading (severity) scale is provided for each AE term. Modifications made by the sponsor are footnoted.

#### **General Instructions**

# Estimating Severity Grade for Parameters Not Identified in the Grading Table

If the need arises to grade a clinical AE that is not identified in the DAIDS grading table, use the category 'Estimating Severity Grade' located at the top of the table on the following page. In addition, all deaths related to an AE are to be classified as Grade 5.

# Grading Adult and Pediatric AEs

The DAIDS grading table includes parameters for grading both adult and pediatric AEs. When a single set of parameters is not appropriate for grading specific types of AEs for both adult and pediatric populations, separate sets of parameters for adult and/or pediatric populations (with specified respective age ranges) are provided. If there is no distinction in the table between adult and pediatric values for a type of AE, then the single set of parameters listed is to be used for grading the severity of both adult and pediatric events of that type.

# **Determining Severity Grade**

If the severity of an AE could fall under either 1 of 2 grades (eg, the severity of an AE could be either Grade 2 or Grade 3), select the higher of the 2 grades for the AE.

Laboratory normal ranges should be taken into consideration to assign gradings to a laboratory value.

#### **Definitions**

Basic Self-care Functions Adult Activities such as bathing, dressing, toileting, transfer or

movement, continence, and feeding.

Young Children Activities that are age and culturally appropriate, such as feeding one's self with culturally

appropriate eating implements.

Usual Social & Functional Activities

Activities which adults and children perform on a routine basis and those which are part of regular activities of daily living, for example:

<u>Adults</u> Adaptive tasks and desirable activities, such as going to work, shopping, cooking, use of transportation, or pursuing a hobby.

Young Children Activities that are age and culturally appropriate, such as social interactions, play activities, or

learning tasks.

Intervention

Medical, surgical, or other procedures recommended or provided by a healthcare professional for the treatment of an AE.

| PARAMETER | GRADE 1<br>MILD | GRADE 2<br>MODERATE | GRADE 3<br>SEVERE | GRADE 4 POTENTIALLY LIFE- THREATENING |
|---|---|---|---|---|
| Clinical adverse<br>event NOT identified<br>elsewhere in the<br>grading table | Mild symptoms causing no or minimal interference with usual social & functional activities with intervention not indicated | Moderate symptoms causing greater than minimal interference with usual social & functional activities with intervention indicated | Severe symptoms causing inability to perform usual social & functional activities with intervention or hospitalization indicated | Potentially life-<br>threatening<br>symptoms causing<br>inability to perform<br>basic self-care<br>functions with<br>intervention<br>indicated to prevent<br>permanent<br>impairment,<br>persistent disability,<br>or death |

| | MAJOR CLINICAL CONDITIONS | | | |
|---|---|---|---|---|
| | МАј | CARDIOVASCULAR | 10113 | |
| PARAMETER | GRADE 1<br>MILD | GRADE 2<br>MODERATE | GRADE 3<br>SEVERE | GRADE 4 POTENTIALLY LIFE- THREATENING |
| Arrhythmia (by ECG or physical examination) Specify type, if applicable | No symptoms AND<br>No intervention<br>indicated | No symptoms AND<br>Non-urgent<br>intervention<br>indicated | Non-life-threatening<br>symptoms AND Non-<br>urgent intervention<br>indicated | Life-threatening<br>arrhythmia OR<br>Urgent intervention<br>indicated |
| Blood Pressure Abnormalities¹ Hypertension (with the lowest reading taken after repeat testing during a | 140 to <160 mmHg<br>systolic OR 90 to<br><100 mmHg diastolic | ≥160 to <180 mmHg<br>systolic OR ≥100 to<br><110 mmHg diastolic | ≥180 mmHg systolic<br>OR ≥110 mmHg<br>diastolic | Life-threatening consequences in a participant not previously diagnosed with hypertension |
| visit)<br>≥18 years of age<br><18 years of age | >120/80 mmHg | ≥95th to <99th percentile + 5 mmHg adjusted for age, height, and gender (systolic and/or diastolic) | ≥99th percentile +<br>5 mmHg adjusted for<br>age, height, and<br>gender (systolic<br>and/or diastolic) | (eg. malignant hypertension) OR Hospitalization indicated Life-threatening consequences in a participant not previously diagnosed with hypertension (eg. malignant |
| Hypotension | No symptoms | Symptoms corrected with oral fluid replacement | Symptoms AND IV fluids indicated | hypertension) OR Hospitalization indicated Shock requiring use of vasopressors or mechanical assistance to maintain blood pressure |
| Tachycardia <sup>h</sup> -<br>beats per minute | 101 - 115 | 116 - 130 | > 130 | ER visit or<br>hospitalization for<br>arrhytmia |
| Bradycardia <sup>a</sup> -<br>beats per minute | 50 - 54 | 45 - 49 | < 45 | ER visit or<br>hospitalization for<br>arrhytmia |
| Cardiac Ischemia or<br>Infarction<br>Report only one | NA | NA | New symptoms with ischemia (stable angina) OR New testing consistent with ischemia | Unstable angina OR<br>Acute myocardial<br>infarction |
| Heart Failure | No symptoms AND<br>Laboratory or cardiac<br>imaging<br>abnormalities | Symptoms with mild<br>to moderate activity<br>or exertion | Symptoms at rest or<br>with minimal activity<br>or exertion (eg,<br>hypoxemia) OR<br>Intervention<br>indicated (eg,<br>oxygen) | Life-threatening consequences OR Urgent intervention indicated (eg, vasoactive medications, ventricular assist device, heart transplant) |

h Modification of DAIDS toxicity table consistent with FDA guidance "Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials, September 2007

| Hemorrhage (with | NA | Symptoms AND No | Symptoms AND | Life-threatening |
|---|---|---|---|---|
| significant acute | | transfusion indicated | Transfusion of ≤2 | hypotension OR |
| blood loss) | | | units packed RBCs | Transfusion of >2 |
| | | | indicated | units packed RBCs |
| | | | | (for children, packed |
| | | | | RBCs >10 cc/kg) |
| | | | | indicated |

<sup>&</sup>lt;sup>1</sup> Blood pressure norms for children <18 years of age can be found in: Expert Panel on Integrated Guidelines for Cardiovascular Health and Risk Reduction in Children and Adolescents. *Pediatrics* 2011;128;S213; originally published online November 14, 2011; DOI: 10.1542/peds.2009 2107C

| PARAMETER | GRADE 1<br>MILD | GRADE 2<br>MODERATE | GRADE 3 SEVERE | GRADE 4 POTENTIALLY LIFE- THREATENING |
|---|---|---|---|---|
| Prolonged PR Interval or AV Block Report only one >16 years of age ≤16 years of age | PR interval 0.21 to<br><0.25 seconds<br>1st degree AV block<br>(PR interval > normal<br>for age and rate) | PR interval<br>≥0.25 seconds OR<br>Type I 2nd degree AV<br>block<br>Type I 2nd degree AV<br>block | Type II 2nd degree AV block OR Ventricular pause ≥3.0 seconds Type II 2nd degree AV block OR Ventricular pause ≥3.0 seconds | Complete AV block Complete AV block |
| Prolonged QTc<br>Interval <sup>2</sup> | 0.45 to 0.47 seconds | >0.47 to 0.50 seconds | >0.50 seconds OR<br>≥0.06 seconds above<br>baseline | Life-threatening<br>consequences (eg,<br>Torsade de pointes,<br>other associated<br>serious ventricular<br>dysrhythmia) |
| Thrombosis or<br>Embolism<br>Report only one | NA | Symptoms AND No intervention indicated | Symptoms AND<br>Intervention<br>indicated | Life-threatening<br>embolic event (eg,<br>pulmonary embolism,<br>thrombus) |

<sup>&</sup>lt;sup>2</sup> As per Bazett's formula.

| | | DERMATOLOGIC | | |
|---|---|---|---|---|
| PARAMETER | GRADE 1<br>MILD | GRADE 2<br>MODERATE | GRADE 3<br>SEVERE | GRADE 4 POTENTIALLY LIFE- THREATENING |
| Alopecia (scalp only) | Detectable by study participant, caregiver, or physician AND Causing no or minimal interference with usual social & functional activities | Obvious on visual inspection AND Causing greater than minimal interference with usual social & functional activities | NA | NA |
| Bruising | Localized to one area | Localized to more than one area | Generalized | NA |
| Cellulitis | NA | Non-parenteral<br>treatment indicated<br>(eg, oral antibiotics,<br>antifungals,<br>antivirals) | IV treatment indicated (eg, IV antibiotics, antifungals, antivirals) | Life-threatening<br>consequences (eg,<br>sepsis, tissue<br>necrosis) |
| Hyperpigmentation | Slight or localized<br>causing no or<br>minimal interference<br>with usual social &<br>functional activities | Marked or<br>generalized causing<br>greater than minimal<br>interference with<br>usual social &<br>functional activities | NA | NA |
| Hypopigmentation | Slight or localized<br>causing no or<br>minimal interference<br>with usual social &<br>functional activities | Marked or<br>generalized causing<br>greater than minimal<br>interference with<br>usual social &<br>functional activities | NA | NA |
| Petechiae | Localized to one area | Localized to more than one area | Generalized | NA |
| Pruritus³ (without skin lesions) | Itching causing no or<br>minimal interference<br>with usual social &<br>functional activities | Itching causing<br>greater than minimal<br>interference with<br>usual social &<br>functional activities | Itching causing inability to perform usual social & functional activities | NA |
| Rash<br>Specify type, if<br>applicable | Localized rash | Diffuse rash OR<br>Target lesions | Diffuse rash AND Vesicles or limited number of bullae OR superficial ulcerations of mucous membrane limited to one site | Extensive or generalized bullous lesions OR Ulceration of mucous membrane involving two or more distinct mucosal sites OR Stevens-Johnson syndrome OR Toxic epidermal necrolysis |

<sup>&</sup>lt;sup>3</sup> For pruritus associated with injections or infusions, see the Site Reactions to Injections and Infusions section.

| | END | OCRINE AND METABO | OLIC | |
|---|---|---|---|---|
| PARAMETER | GRADE 1<br>MILD | GRADE 2<br>MODERATE | GRADE 3<br>SEVERE | GRADE 4 POTENTIALLY LIFE- THREATENING |
| Diabetes Mellitus | Controlled without medication | Controlled with<br>medication OR<br>Modification of<br>current medication<br>regimen | Uncontrolled despite<br>treatment<br>modification OR<br>Hospitalization for<br>immediate glucose<br>control indicated | Life-threatening<br>consequences (eg,<br>ketoacidosis,<br>hyperosmolar non-<br>ketotic coma, end<br>organ failure) |
| Gynecomastia | Detectable by study participant, caregiver, or physician AND Causing no or minimal interference with usual social & functional activities | Obvious on visual inspection AND Causing pain with greater than minimal interference with usual social & functional activities | Disfiguring changes AND Symptoms requiring intervention or causing inability to perform usual social & functional activities | NA |
| Hyperthyroidism | No symptoms AND<br>Abnormal laboratory<br>value | Symptoms causing greater than minimal interference with usual social & functional activities OR Thyroid suppression therapy indicated | Symptoms causing inability to perform usual social & functional activities OR Uncontrolled despite treatment modification | Life-threatening<br>consequences (eg,<br>thyroid storm) |
| Hypothyroidism | No symptoms AND<br>Abnormal laboratory<br>value | Symptoms causing greater than minimal interference with usual social & functional activities OR Thyroid replacement therapy indicated | Symptoms causing inability to perform usual social & functional activities OR Uncontrolled despite treatment modification | Life-threatening<br>consequences (eg,<br>myxedema coma) |
| Lipoatrophy <sup>4</sup> | Detectable by study participant, caregiver, or physician AND Causing no or minimal interference with usual social & functional activities | Obvious on visual inspection AND Causing greater than minimal interference with usual social & functional activities | Disfiguring changes | NA |
| Lipohypertrophy <sup>5</sup> | Detectable by study participant, caregiver, or physician AND Causing no or minimal interference with usual social & functional activities | Obvious on visual inspection AND Causing greater than minimal interference with usual social & functional activities | Disfiguring changes | NA |

<sup>&</sup>lt;sup>4</sup> Definition: A disorder characterized by fat loss in the face, extremities, and buttocks.

<sup>&</sup>lt;sup>5</sup> Definition: A disorder characterized by abnormal fat accumulation on the back of the neck, breasts, and abdomen.

| | | GASTROINTESTINA | AL | |
|---|---|---|---|---|
| PARAMETER | GRADE 1<br>MILD | GRADE 2 MODERATE | GRADE 3 SEVERE | GRADE 4 POTENTIALLY LIFE- THREATENING |
| Anorexia | Loss of appetite without decreased oral intake | Loss of appetite<br>associated with<br>decreased oral intake<br>without significant<br>weight loss | Loss of appetite<br>associated with<br>significant weight<br>loss | Life-threatening<br>consequences OR<br>Aggressive intervention<br>indicated (eg, tube<br>feeding, total parenteral<br>nutrition) |
| Ascites | No symptoms | Symptoms AND Intervention indicated (eg, diuretics, therapeutic paracentesis) | Symptoms recur or persist despite intervention | Life-threatening consequences |
| Bloating or<br>Distension<br>Report only one | Symptoms causing no or<br>minimal interference<br>with usual social &<br>functional activities | Symptoms causing greater than minimal interference with usual social & functional activities | Symptoms causing inability to perform usual social & functional activities | NA |
| Cholecystitis | NA | Symptoms AND<br>Medical intervention<br>indicated | Radiologic,<br>endoscopic, or<br>operative<br>intervention<br>indicated | Life-threatening<br>consequences (eg,<br>sepsis, perforation) |
| Constipation | NA | Persistent constipation<br>requiring regular use of<br>dietary modifications,<br>laxatives, or enemas | Obstipation with manual evacuation indicated | Life-threatening<br>consequences (eg,<br>obstruction) |
| Diarrhea<br>≥1 year of<br>age | Transient or<br>intermittent episodes of<br>unformed stools OR<br>Increase of ≤3 stools<br>over baseline per 24-<br>hour period | Persistent episodes of<br>unformed to watery<br>stools OR Increase of 4<br>to 6 stools over<br>baseline per 24-hour<br>period | Increase of ≥7 stools<br>per 24-hour period<br>OR IV fluid<br>replacement<br>indicated | Life-threatening<br>consequences (eg,<br>hypotensive shock) |
| <1 year of<br>age | Liquid stools (more<br>unformed than usual)<br>but usual number of<br>stools | Liquid stools with<br>increased number of<br>stools OR Mild<br>dehydration | Liquid stools with moderate dehydration | Life-threatening<br>consequences (eg, liquid<br>stools resulting in severe<br>dehydration,<br>hypotensive shock) |
| Dysphagia or<br>Odynophagia<br>Report only one<br>and specify<br>location | Symptoms but able to eat usual diet | Symptoms causing altered dietary intake with no intervention indicated | Symptoms causing<br>severely altered<br>dietary intake with<br>intervention<br>indicated | Life-threatening reduction in oral intake |
| Gastrointestin<br>al Bleeding | Not requiring intervention other than iron supplement | Endoscopic intervention indicated | Transfusion indicated | Life-threatening<br>consequences (eg,<br>hypotensive shock) |
| Mucositis or<br>Stomatitis<br>Report only one<br>and specify<br>location | Mucosal erythema | Patchy<br>pseudomembranes or<br>ulcerations | Confluent pseudomembranes or ulcerations OR Mucosal bleeding with minor trauma | Life-threatening<br>consequences (eg,<br>aspiration, choking) OR<br>Tissue necrosis OR<br>Diffuse spontaneous<br>mucosal bleeding |
| Nausea | Transient (<24 hours) or intermittent AND No or minimal interference with oral intake | Persistent nausea<br>resulting in decreased<br>oral intake for 24 to<br>48 hours | Persistent nausea<br>resulting in minimal<br>oral intake for<br>>48 hours OR<br>Rehydration<br>indicated (eg, IV<br>fluids) | Life-threatening<br>consequences (eg,<br>hypotensive shock) |

# Clinical Protocol VAC89220HPX2004 Amendment 5

| PARAMETER | GRADE 1<br>MILD | GRADE 2<br>MODERATE | GRADE 3<br>SEVERE | GRADE 4 POTENTIALLY LIFE- THREATENING |
|---|---|---|---|---|
| Pancreatitis | NA | Symptoms with hospitalization not indicated | Symptoms with hospitalization indicated | Life-threatening<br>consequences (eg,<br>circulatory failure,<br>hemorrhage, sepsis) |
| Perforation<br>(colon or rectum) | NA | NA | Intervention indicated | Life-threatening consequences |
| Proctitis | Rectal discomfort<br>with no intervention<br>indicated | Symptoms causing greater than minimal interference with usual social & functional activities OR Medical intervention indicated | Symptoms causing inability to perform usual social & functional activities OR Operative intervention indicated | Life-threatening<br>consequences (eg,<br>perforation) |
| Rectal Discharge | Visible discharge | Discharge requiring the use of pads | NA | NA |
| Vomiting | Transient or intermittent AND No or minimal interference with oral intake | Frequent episodes<br>with no or mild<br>dehydration | Persistent vomiting resulting in orthostatic hypotension OR Aggressive rehydration indicated (eg, IV fluids) | Life-threatening<br>consequences (eg.<br>hypotensive shock) |

| | | MUSCULOSKELETAL | | |
|---|---|---|---|---|
| PARAMETER | GRADE 1<br>MILD | GRADE 2<br>MODERATE | GRADE 3<br>SEVERE | GRADE 4 POTENTIALLY LIFE- THREATENING |
| Arthralgia | Joint pain causing no<br>or minimal<br>interference with<br>usual social &<br>functional activities | Joint pain causing<br>greater than minimal<br>interference with<br>usual social &<br>functional activities | Joint pain causing inability to perform usual social & functional activities | Disabling joint pain<br>causing inability to<br>perform basic self-<br>care functions |
| Arthritis | Stiffness or joint<br>swelling causing no or<br>minimal interference<br>with usual social &<br>functional activities | Stiffness or joint<br>swelling causing<br>greater than minimal<br>interference with<br>usual social &<br>functional activities | Stiffness or joint<br>swelling causing<br>inability to perform<br>usual social &<br>functional activities | Disabling joint<br>stiffness or swelling<br>causing inability to<br>perform basic self-<br>care functions |
| Myalgia<br>(generalized) | Muscle pain causing<br>no or minimal<br>interference with<br>usual social &<br>functional activities | Muscle pain causing greater than minimal interference with usual social & functional activities | Muscle pain causing inability to perform usual social & functional activities | Disabling muscle<br>pain causing inability<br>to perform basic self-<br>care functions |
| Osteonecrosis | NA | No symptoms but<br>with radiographic<br>findings AND No<br>operative<br>intervention<br>indicated | Bone pain with<br>radiographic findings<br>OR Operative<br>intervention<br>indicated | Disabling bone pain<br>with radiographic<br>findings causing<br>inability to perform<br>basic self-care<br>functions |
| Osteopenia <sup>6</sup> ≥30 years of age | BMD t-score -2.5 to -1 BMD z-score -2 to -1 | NA<br>NA | NA<br>NA | NA<br>NA |
| <30 years of age Osteoporosis <sup>6</sup> ≥30 years of age <30 years of age | NA NA | BMD t-score <-2.5 | Pathologic fracture (eg, compression fracture causing loss of vertebral height) Pathologic fracture | Pathologic fracture<br>causing life-<br>threatening<br>consequences<br>Pathologic fracture |
| -30 yeurs of age | 1441 | Bird E-Score N-2 | (eg, compression<br>fracture causing loss<br>of vertebral height) | causing life-<br>threatening<br>consequences |

<sup>&</sup>lt;sup>6</sup> BMD t and z scores can be found in: Kanis JA on behalf of the World Health Organization Scientific Group (2007). Assessment of osteoporosis at the primary health care level. Technical Report. World Health Organization Collaborating Centre for Metabolic Bone Diseases, University of Sheffield, UK. 2007: Printed by the University of Sheffield.

| | NEUROLOGIC | | | |
|---|---|---|---|---|
| PARAMETER | GRADE 1 | GRADE 2 | GRADE 3 | GRADE 4 |
| | MILD | MODERATE | SEVERE | POTENTIALLY LIFE-<br>THREATENING |
| Acute CNS Ischemia | NA | NA | Transient ischemic attack | Cerebral vascular<br>accident (eg, stroke<br>with neurological<br>deficit) |
| Altered Mental Status (for Dementia, see Cognitive, Behavioral, or Attentional Disturbance below) | Changes causing no<br>or minimal<br>interference with<br>usual social &<br>functional activities | Mild lethargy or<br>somnolence causing<br>greater than minimal<br>interference with<br>usual social &<br>functional activities | Confusion, memory impairment, lethargy, or somnolence causing inability to perform usual social & functional activities | Delirium OR<br>Obtundation OR<br>Coma |
| Ataxia | Symptoms causing no or minimal interference with usual social & functional activities OR No symptoms with ataxia detected on examination | Symptoms causing greater than minimal interference with usual social & functional activities | Symptoms causing inability to perform usual social & functional activities | Disabling symptoms<br>causing inability to<br>perform basic self-<br>care functions |
| Cognitive, Behavioral, or Attentional Disturbance (includes dementia and attention deficit disorder) Specify type, if applicable | Disability causing no<br>or minimal<br>interference with<br>usual social &<br>functional activities<br>OR Specialized<br>resources not<br>indicated | Disability causing greater than minimal interference with usual social & functional activities OR Specialized resources on parttime basis indicated | Disability causing inability to perform usual social & functional activities OR Specialized resources on a full-time basis indicated | Disability causing inability to perform basic self-care functions OR Institutionalization indicated |
| Developmental Delay <18 years of age Specify type, if applicable | Mild developmental delay, either motor or cognitive, as determined by comparison with a developmental screening tool appropriate for the setting | Moderate developmental delay, either motor or cognitive, as determined by comparison with a developmental screening tool appropriate for the setting | Severe developmental delay, either motor or cognitive, as determined by comparison with a developmental screening tool appropriate for the setting | Developmental regression, either motor or cognitive, as determined by comparison with a developmental screening tool appropriate for the setting |
| Headache | Symptoms causing no<br>or minimal<br>interference with<br>usual social &<br>functional activities | Symptoms causing greater than minimal interference with usual social & functional activities | Symptoms causing inability to perform usual social & functional activities | Symptoms causing inability to perform basic self-care functions OR Hospitalization indicated OR Headache with significant impairment of alertness or other neurologic function |
| Neuromuscular Weakness (includes myopathy and neuropathy) Specify type, if applicable | Minimal muscle weakness causing no or minimal interference with usual social & functional activities OR No symptoms with decreased strength on examination | Muscle weakness<br>causing greater than<br>minimal interference<br>with usual social &<br>functional activities | Muscle weakness<br>causing inability to<br>perform usual social<br>& functional activities | Disabling muscle weakness causing inability to perform basic self-care functions OR Respiratory muscle weakness impairing ventilation |

| DADAMETER | CDADE 4 | CDADES | CDADES | CDAREA |
|---|---|---|---|---|
| PARAMETER | GRADE 1<br>MILD | GRADE 2<br>MODERATE | GRADE 3<br>SEVERE | GRADE 4 POTENTIALLY LIFE- THREATENING |
| Neurosensory Alteration (includes paresthesia and painful neuropathy) Specify type, if applicable | Minimal paresthesia causing no or minimal interference with usual social & functional activities OR No symptoms with sensory alteration on examination | Sensory alteration or<br>paresthesia causing<br>greater than minimal<br>interference with<br>usual social &<br>functional activities | Sensory alteration or<br>paresthesia causing<br>inability to perform<br>usual social &<br>functional activities | Disabling sensory<br>alteration or<br>paresthesia causing<br>inability to perform<br>basic self-care<br>functions |
| Seizures New Onset Seizure ≥18 years of age | NA | NA | 1 to 3 seizures | Prolonged and repetitive seizures (eg, status epilepticus) OR Difficult to control (eg, refractory epilepsy) |
| <18 years of age<br>(includes new or pre-<br>existing febrile<br>seizures) | Seizure lasting <5 minutes with <24 hours postictal state | Seizure lasting 5 to<br><20 minutes with<br><24 hours postictal<br>state | Seizure lasting<br>≥20 minutes OR<br>>24 hours postictal<br>state | Prolonged and repetitive seizures (eg, status epilepticus) OR Difficult to control (eg, refractory epilepsy) |
| Pre-existing<br>Seizure | NA | Increased frequency<br>from previous level of<br>control without<br>change in seizure<br>character | Change in seizure<br>character either in<br>duration or quality<br>(eg, severity or<br>focality) | Prolonged and repetitive seizures (eg, status epilepticus) OR Difficult to control (eg, refractory epilepsy) |
| Syncope | Near syncope without<br>loss of consciousness<br>(eg, pre-syncope) | Loss of consciousness with no intervention indicated | Loss of consciousness<br>AND Hospitalization<br>or intervention<br>required | NA NA |

| | PREGNANCY, PUERPERIUM, AND PERINATAL | | | |
|---|---|---|---|---|
| PARAMETER | GRADE 1<br>MILD | GRADE 2<br>MODERATE | GRADE 3<br>SEVERE | GRADE 4 POTENTIALLY LIFE- THREATENING |
| Fetal Death or<br>Stillbirth (report<br>using mother's<br>participant ID)<br>Report only one | NA | NA | Fetal loss occurring<br>at ≥20 weeks<br>gestation | NA |
| Preterm Delivery <sup>7</sup> (report using mother's participant ID) | Delivery at 34 to<br><37 weeks gestational<br>age | Delivery at 28 to<br><34 weeks<br>gestational age | Delivery at 24 to<br><28 weeks<br>gestational age | Delivery at <24<br>weeks gestational age |
| Spontaneous Abortion or Miscarriage <sup>8</sup> (report using mother's participant ID) Report only one | Chemical pregnancy | Uncomplicated<br>spontaneous abortion<br>or miscarriage | Complicated spontaneous abortion or miscarriage | NA |

<sup>&</sup>lt;sup>7</sup> Definition: A delivery of a live born neonate occurring at ≥20 to <37 weeks gestational age.

<sup>&</sup>lt;sup>8</sup> Definition: A clinically recognized pregnancy occurring at <20 weeks gestational age.

| | | PSYCHIATRIC | | |
|---|---|---|---|---|
| PARAMETER | GRADE 1<br>MILD | GRADE 2<br>MODERATE | GRADE 3<br>SEVERE | GRADE 4 POTENTIALLY LIFE- THREATENING |
| Insomnia | Mild difficulty falling<br>asleep, staying asleep,<br>or waking up early | Moderate difficulty<br>falling asleep, staying<br>asleep, or waking up<br>early | Severe difficulty<br>falling asleep, staying<br>asleep, or waking up<br>early | NA |
| Psychiatric Disorders (includes anxiety, depression, mania, and psychosis) Specify disorder | Symptoms with intervention not indicated OR Behavior causing no or minimal interference with usual social & functional activities | Symptoms with intervention indicated OR Behavior causing greater than minimal interference with usual social & functional activities | Symptoms with<br>hospitalization<br>indicated OR<br>Behavior causing<br>inability to perform<br>usual social &<br>functional activities | Threatens harm to<br>self or others OR<br>Acute psychosis OR<br>Behavior causing<br>inability to perform<br>basic self-care<br>functions |
| Suicidal Ideation or<br>Attempt<br>Report only one | Preoccupied with<br>thoughts of death<br>AND No wish to kill<br>oneself | Preoccupied with<br>thoughts of death<br>AND Wish to kill<br>oneself with no<br>specific plan or intent | Thoughts of killing oneself with partial or complete plans but no attempt to do so OR Hospitalization indicated | Suicide attempted |

| | | RESPIRATORY | | |
|---|---|---|---|---|
| PARAMETER | GRADE 1<br>MILD | GRADE 2<br>MODERATE | GRADE 3<br>SEVERE | GRADE 4 POTENTIALLY LIFE- THREATENING |
| Acute Bronchospasm | Forced expiratory<br>volume in 1 second or<br>peak flow reduced to<br>≥70 to <80% OR<br>Mild symptoms with<br>intervention not<br>indicated | Forced expiratory volume in 1 second or peak flow 50 to <70% OR Symptoms with intervention indicated OR Symptoms causing greater than minimal interference with usual social & functional activities | Forced expiratory<br>volume in 1 second or<br>peak flow 25 to <50%<br>OR Symptoms<br>causing inability to<br>perform usual social<br>& functional activities | Forced expiratory volume in 1 second or peak flow <25% OR Life threatening respiratory or hemodynamic compromise OR Intubation |
| Dyspnea or<br>Respiratory Distress<br>Report only one | Dyspnea on exertion with no or minimal interference with usual social & functional activities OR Wheezing OR Minimal increase in respiratory rate for age | Dyspnea on exertion causing greater than minimal interference with usual social & functional activities OR Nasal flaring OR Intercostal retractions OR Pulse oximetry 90 to <95% | Dyspnea at rest<br>causing inability to<br>perform usual social<br>& functional activities<br>OR Pulse oximetry<br><90% | Respiratory failure with<br>ventilator support<br>indicated (eg, CPAP,<br>BPAP, intubation) |

| | | SENSORY | | |
|---|---|---|---|---|
| PARAMETER | GRADE 1<br>MILD | GRADE 2<br>MODERATE | GRADE 3<br>SEVERE | GRADE 4 POTENTIALLY LIFE- THREATENING |
| Hearing Loss ≥12 years of age <12 years of age (based on a 1, 2, 3, 4, 6 and 8 kHz | NA >20 dB hearing loss at ≤4 kHz | Hearing aid or intervention not indicated >20 dB hearing loss at >4 kHz | Hearing aid or intervention indicated >20 dB hearing loss at ≥3 kHz in one ear with additional speech | Profound bilateral<br>hearing loss (>80 dB at<br>2 kHz and above) OR<br>Non serviceable<br>hearing (ie, >50 dB<br>audiogram and <50%<br>speech discrimination)<br>Audiologic indication<br>for cochlear implant<br>and additional speech |
| audiogram) | | | language related<br>services indicated<br>(where available) OR<br>Hearing loss sufficient<br>to indicate therapeutic<br>intervention, including<br>hearing aids | language related<br>services indicated<br>(where available) |
| Tinnitus | Symptoms causing no<br>or minimal<br>interference with usual<br>social & functional<br>activities with<br>intervention not<br>indicated | Symptoms causing greater than minimal interference with usual social & functional activities with intervention indicated | Symptoms causing inability to perform usual social & functional activities | NA |
| Uveitis | No symptoms AND<br>Detectable on<br>examination | Anterior uveitis with<br>symptoms OR<br>Medicamylasal<br>intervention indicated | Posterior or pan<br>uveitis OR Operative<br>intervention indicated | Disabling visual loss in affected eye(s) |
| Vertigo | Vertigo causing no or<br>minimal interference<br>with usual social &<br>functional activities | Vertigo causing greater<br>than minimal<br>interference with usual<br>social & functional<br>activities | Vertigo causing inability to perform usual social & functional activities | Disabling vertigo<br>causing inability to<br>perform basic self care<br>functions |
| Visual Changes<br>(assessed from<br>baseline) | Visual changes<br>causing no or minimal<br>interference with usual<br>social & functional<br>activities | Visual changes causing<br>greater than minimal<br>interference with usual<br>social & functional<br>activities | Visual changes<br>causing inability to<br>perform usual social &<br>functional activities | Disabling visual loss in affected eye(s) |

| | | SYSTEMIC | | |
|---|---|---|---|---|
| PARAMETER | GRADE 1<br>MILD | GRADE 2<br>MODERATE | GRADE 3<br>SEVERE | GRADE 4 POTENTIALLY LIFE- THREATENING |
| Acute Allergic<br>Reaction | Localized urticaria<br>(wheals) with no<br>medical intervention<br>indicated | Localized urticaria<br>with intervention<br>indicated OR Mild<br>angioedema with no<br>intervention indicated | Generalized urticaria OR Angioedema with intervention indicated OR Symptoms of mild bronchospasm | Acute anaphylaxis OR<br>Life threatening<br>bronchospasm OR<br>Laryngeal edema |
| Chills | Symptoms causing no<br>or minimal<br>interference with usual<br>social & functional<br>activities | Symptoms causing greater than minimal interference with usual social & functional activities | Symptoms causing inability to perform usual social & functional activities | NA |
| Cytokine Release<br>Syndrome <sup>9</sup> | Mild signs and<br>symptoms AND<br>Therapy (ie, antibody<br>infusion) interruption<br>not indicated | Therapy (ie, antibody infusion) interruption indicated AND Responds promptly to symptomatic treatment OR Prophylactic medications indicated for ≤24 hours | Prolonged severe signs<br>and symptoms OR<br>Recurrence of<br>symptoms following<br>initial improvement | Life threatening<br>consequences (eg,<br>requiring pressor or<br>ventilator support) |
| Fatigue or Malaise<br>Report only one | Symptoms causing no<br>or minimal<br>interference with usual<br>social & functional<br>activities | Symptoms causing greater than minimal interference with usual social & functional activities | Symptoms causing inability to perform usual social & functional activities | Incapacitating<br>symptoms of fatigue or<br>malaise causing<br>inability to perform<br>basic self care<br>functions |
| Fever (non axillary temperatures only) | 38.0 to <38.6°C or<br>100.4 to <101.5°F | ≥38.6 to <39.3°C or<br>≥101.5 to <102.7°F | ≥39.3 to <40.0°C or<br>≥102.7 to <104.0°F | ≥40.0°C or ≥104.0°F |
| Pain <sup>10</sup> (not associated<br>with study agent<br>injections and not<br>specified elsewhere)<br>Specify location | Pain causing no or<br>minimal interference<br>with usual social &<br>functional activities | Pain causing greater<br>than minimal<br>interference with usual<br>social & functional<br>activities | Pain causing inability<br>to perform usual social<br>& functional activities | Disabling pain causing inability to perform basic self care functions OR Hospitalization indicated |
| Serum Sickness <sup>11</sup> | Mild signs and symptoms | Moderate signs and<br>symptoms AND<br>Intervention indicated<br>(eg, antihistamines) | Severe signs and<br>symptoms AND<br>Higher level<br>intervention indicated<br>(eg, steroids or IV<br>fluids) | Life threatening<br>consequences (eg,<br>requiring pressor or<br>ventilator support) |
| Underweight <sup>12</sup> >5 to 19 years of age 2 to 5 years of age | NA<br>NA | WHO BMI z score $< 2$<br>to $\le 3$<br>WHO Weight for<br>height z score<br>$< 2$ to $\le 3$ | WHO BMI z score < 3 WHO Weight for height z score < 3 | WHO BMI z score < 3<br>with life threatening<br>consequences<br>WHO Weight for<br>height z score < 3 with<br>life threatening |
| <2 years of age | NA | WHO Weight for length z score < 2 to ≤ 3 | WHO Weight for length z score < 3 | consequences WHO Weight for length z score < 3 with life threatening consequences |

<sup>9</sup> Definition: A disorder characterized by nausea, headache, tachycardia, hypotension, rash, and/or shortness of breath.

http://www.who.int/childgrowth/standards/chart\_catalogue/en/ for those ≤5 years of age.

<sup>&</sup>lt;sup>10</sup> For pain associated with injections or infusions, see the *Site Reactions to Injections and Infusions* section.

<sup>&</sup>lt;sup>11</sup> Definition: A disorder characterized by fever, arthralgia, myalgia, skin eruptions, lymphadenopathy, marked discomfort, and/or dyspnea.

<sup>&</sup>lt;sup>12</sup> WHO reference tables may be accessed by clicking the desired age range or by accessing the following URLs: http://www.who.int/growthref/who2007\_bmi\_for\_age/en/ for participants >5 to 19 years of age and

# JNJ-55471468, JNJ-55471494, JNJ-55471520, JNJ-55471585, JNJ-64219324

# Clinical Protocol VAC89220HPX2004 Amendment 5

| PARAMETER | GRADE 1<br>MILD | GRADE 2<br>MODERATE | GRADE 3<br>SEVERE | GRADE 4 POTENTIALLY LIFE- THREATENING |
|---|---|---|---|---|
| Weight Loss<br>(excludes postpartum<br>weight loss) | NA | 5 to <9% loss in body<br>weight from baseline | ≥9 to <20% loss in<br>body weight from<br>baseline | ≥20% loss in body<br>weight from baseline<br>OR Aggressive<br>intervention indicated<br>(eg, tube feeding, total<br>parenteral nutrition) |

| URINARY | | | | |
|---|---|---|---|---|
| PARAMETER | GRADE 1<br>MILD | GRADE 2<br>MODERATE | GRADE 3<br>SEVERE | GRADE 4 POTENTIALLY LIFE- THREATENING |
| Urinary Tract<br>Obstruction | NA | Signs or symptoms of<br>urinary tract<br>obstruction without<br>hydronephrosis or renal<br>dysfunction | Signs or symptoms of<br>urinary tract<br>obstruction with<br>hydronephrosis or<br>renal dysfunction | Obstruction causing life threatening consequences |

| | SITE REACTION | ONS TO INJECTIONS A | ND INFUSIONS | |
|---|---|---|---|---|
| PARAMETER | GRADE 1<br>MILD | GRADE 2<br>MODERATE | GRADE 3<br>SEVERE | GRADE 4 POTENTIALLY LIFE- THREATENING |
| Injection Site Pain or<br>Tenderness<br>Report only one | Pain or tenderness<br>causing no or minimal<br>limitation of use of<br>limb | Pain or tenderness<br>causing greater than<br>minimal limitation of<br>use of limb | Pain or tenderness<br>causing inability to<br>perform usual social &<br>functional activities | Pain or tenderness<br>causing inability to<br>perform basic self care<br>function OR<br>Hospitalization<br>indicated |
| Injection Site Erythema or Redness <sup>13</sup> Report only one >15 years of age | 2.5 to <5 cm in<br>diameter OR 6.25 to<br><25 cm² surface area<br>AND Symptoms<br>causing no or minimal<br>interference with<br>usual social &<br>functional activities | ≥5 to <10 cm in<br>diameter OR ≥25 to<br><100 cm² surface area<br>OR Symptoms causing<br>greater than minimal<br>interference with usual<br>social & functional<br>activities | ≥10 cm in diameter OR ≥100 cm² surface area OR Ulceration OR Secondary infection OR Phlebitis OR Sterile abscess OR Drainage OR Symptoms causing inability to perform usual social & functional activities | Potentially life<br>threatening<br>consequences (eg,<br>abscess, exfoliative<br>dermatitis, necrosis<br>involving dermis or<br>deeper tissue) |
| ≤15 years of age | ≤2.5 cm in diameter | >2.5 cm in diameter<br>with <50% surface area<br>of the extremity<br>segment involved (eg,<br>upper arm or thigh) | ≥50% surface area of the extremity segment involved (eg, upper arm or thigh) OR Ulceration OR Secondary infection OR Phlebitis OR Sterile abscess OR Drainage | Potentially life<br>threatening<br>consequences (eg,<br>abscess, exfoliative<br>dermatitis, necrosis<br>involving dermis or<br>deeper tissue) |
| Injection Site Induration or Swelling Report only one >15 years of age ≤15 years of age | Same as for Injection<br>Site Erythema or<br>Redness, >15 years<br>of age<br>Same as for Injection | Same as for Injection Site Erythema or Redness, >15 years of age Same as for Injection | Same as for Injection Site Erythema or Redness, >15 years of age Same as for Injection | Same as for Injection Site Erythema or Redness, >15 years of age Same as for Injection |
| | Site Erythema or<br>Redness, ≤15 years of<br>age | Site Erythema or<br>Redness, ≤15 years of<br>age | Site Erythema or<br>Redness, ≤15 years of<br>age | Site Erythema or<br>Redness, ≤15 years of<br>age |
| Injection Site Pruritus | Itching localized to<br>the injection site that<br>is relieved<br>spontaneously or in<br><48 hours of<br>treatment | Itching beyond the injection site that is not generalized OR Itching localized to the injection site requiring ≥48 hours treatment | Generalized itching<br>causing inability to<br>perform usual social &<br>functional activities | NA |

treatment ≥48 hours treatment |

13 Injection Site Erythema or Redness should be evaluated and graded using the greatest single diameter or measured surface area.

| | LABORATORY VALUES | | | |
|---|---|---|---|---|
| | | CHEMISTRIES | 3 | |
| PARAMETER | GRADE 1<br>MILD | GRADE 2<br>MODERATE | GRADE 3<br>SEVERE | GRADE 4 POTENTIALLY LIFE- THREATENING |
| Acidosis | NA | pH ≥7.3 to <lln< td=""><td>pH &lt;7.3 without life<br/>threatening<br/>consequences</td><td>pH &lt;7.3 with life<br/>threatening<br/>consequences</td></lln<> | pH <7.3 without life<br>threatening<br>consequences | pH <7.3 with life<br>threatening<br>consequences |
| Albumin, Low (g/dL; g/L) | 3.0 to <lln<br>30 to <lln< td=""><td>≥2.0 to &lt;3.0<br/>≥20 to &lt;30</td><td>&lt;2.0<br/>&lt;20</td><td>NA</td></lln<></lln<br> | ≥2.0 to <3.0<br>≥20 to <30 | <2.0<br><20 | NA |
| Alkaline<br>Phosphatase, High | 1.25 to <2.5 x ULN | 2.5 to <5.0 x ULN | 5.0 to <10.0 x ULN | ≥10.0 x ULN |
| Alkalosis | NA | pH > ULN to ≤7.5 | pH >7.5 without life<br>threatening<br>consequences | pH >7.5 with life<br>threatening<br>consequences |
| ALT or SGPT, High<br>Report only one | 1.25 to <2.5 x ULN | 2.5 to <5.0 x ULN | 5.0 to <10.0 x ULN | ≥10.0 x ULN |
| Amylase (Pancreatic)<br>or Amylase (Total),<br>High<br>Report only one | 1.1 to <1.5 x ULN | 1.5 to < 3.0 x ULN | 3.0 to <5.0 x ULN | ≥5.0 x ULN |
| AST or SGOT, High<br>Report only one | 1.25 to <2.5 x ULN | 2.5 to <5.0 x ULN | 5.0 to <10.0 x ULN | ≥10.0 x ULN |
| Bicarbonate, Low (mEq/L; mmol/L) | 16.0 to <lln<br>16.0 to <lln< td=""><td>11.0 to &lt;16.0<br/>11.0 to &lt;16.0</td><td>8.0 to &lt;11.0<br/>8.0 to &lt;11.0</td><td>&lt;8.0<br/>&lt;8.0</td></lln<></lln<br> | 11.0 to <16.0<br>11.0 to <16.0 | 8.0 to <11.0<br>8.0 to <11.0 | <8.0<br><8.0 |
| Bilirubin Direct Bilirubin <sup>14</sup> , High >28 days of age | NA | NA | >ULN | >ULN with life<br>threatening<br>consequences (eg,<br>signs and symptoms of<br>liver failure) |
| ≤28 days of age<br>Total Bilirubin,<br>High | ULN to ≤1 mg/dL<br>1.1 to <1.6 x ULN | >1 to ≤1.5 mg/dL<br>1.6 to <2.6 x ULN | >1.5 to ≤2 mg/dL<br>2.6 to < 5.0 x ULN | >2 mg/dL<br>≥5.0 x ULN |
| >28 days of age<br>≤28 days of age | See Appendix A. Total<br>Bilirubin for Term and<br>Preterm Neonates | See Appendix A. Total<br>Bilirubin for Term and<br>Preterm Neonates | See Appendix A. Total<br>Bilirubin for Term and<br>Preterm Neonates | See Appendix A. Total<br>Bilirubin for Term and<br>Preterm Neonates |
| Calcium, High (mg/dL; mmol/L) ≥7 days of age <7 days of age | 10.6 to <11.5<br>2.65 to <2.88<br>11.5 to <12.4<br>2.88 to <3.10 | 11.5 to <12.5<br>2.88 to <3.13<br>12.4 to <12.9<br>3.10 to <3.23 | 12.5 to <13.5<br>3.13 to <3.38<br>12.9 to <13.5<br>3.23 to <3.38 | ≥13.5<br>≥3.38<br>≥13.5<br>≥3.38 |
| Calcium (Ionized),<br>High (mg/dL;<br>mmol/L) | >ULN to <6.0<br>>ULN to <1.5 | 6.0 to <6.4<br>1.5 to <1.6 | 6.4 to <7.2<br>1.6 to <1.8 | ≥7.2<br>≥1.8 |
| Calcium, Low<br>(mg/dL; mmol/L)<br>≥7 days of age | 7.8 to <8.4<br>1.95 to <2.10 | 7.0 to <7.8<br>1.75 to <1.95 | 6.1 to <7.0<br>1.53 to <1.75 | <6.1<br><1.53 |
| <7 days of age | 6.5 to <7.5<br>1.63 to <1.88 | 6.0 to <6.5<br>1.50 to <1.63 | 5.50 to <6.0<br>1.38 to <1.50 | <5.50<br><1.38 |
| Calcium (Ionized),<br>Low (mg/dL; mmol/L) | <lln 4.0<br="" to=""><lln 1.0<="" td="" to=""><td>3.6 to &lt;4.0<br/>0.9 to &lt;1.0</td><td>3.2 to &lt;3.6<br/>0.8 to &lt;0.9</td><td>&lt;3.2<br/>&lt;0.8</td></lln></lln> | 3.6 to <4.0<br>0.9 to <1.0 | 3.2 to <3.6<br>0.8 to <0.9 | <3.2<br><0.8 |
| Cardiac Troponin I,<br>High | NA NA | NA NA | NA NA | Levels consistent with<br>myocardial infarction<br>or unstable angina as<br>defined by the local<br>laboratory |

laboratory

14 Direct bilirubin >1.5 mg/dL in a participant <28 days of age should be graded as grade 2, if <10% of the total bilirubin.

| PARAMETER | GRADE 1<br>MILD | GRADE 2<br>MODERATE | GRADE 3<br>SEVERE | GRADE 4<br>POTENTIALLY |
|---|---|---|---|---|
| | | | ~= , ==== | LIFE- |
| | | | | THREATENING |
| Creatine Kinase,<br>High | 3 to <6 x ULN | 6 to <10 x ULN | 10 to <20 x ULN | ≥20 x ULN |
| Creatinine, High | 1.1 to 1.3 x ULN | >1.3 to 1.8 x ULN OR | >1.8 to <3.5 x ULN | ≥3.5 x ULN OR |
| | | Increase of >0.3 mg/dL | OR Increase of 1.5 to | Increase of $\geq 2.0 \text{ x}$ |
| | | above baseline | <2.0 x above baseline | above baseline |
| Creatinine | NA | <90 to 60 ml/min or | <60 to 30ml/min or | <30 ml/min or |
| Clearance <sup>15</sup> or | | ml/min/1.73 m <sup>2</sup> OR 10 | ml/min/1.73 m <sup>2</sup> OR | ml/min/1.73 m <sup>2</sup> OR |
| eGFR, Low | | to <30% decrease from | ≥30 to <50% decrease | ≥50% decrease from |
| Report only one | | baseline | from baseline | baseline or dialysis<br>needed |
| Glucose | 110 to 125 | >125 to 250 | >250 to 500 | >500 |
| (mg/dL; mmol/L) | 6.11 to <6.95 | 6.95 to <13.89 | 13.89 to <27.75 | ≥27.75 |
| Fasting, High | | | | |
| Nonfasting, High | 116 to 160 | >160 to 250 | >250 to 500 | >500 |
| | 6.44 to <8.89 | 8.89 to <13.89 | 13.89 to <27.75 | ≥27.75 |
| Glucose, Low | 55 to 64 | 40 to <55 | 30 to <40 | <30 |
| (mg/dL; mmol/L) | 3.05 to 3.55 | 2.22 to <3.05 | 1.67 to <2.22 | <1.67 |
| $\geq 1$ month of age | | | | |
| <1 month of age | 50 to 54 | 40 to < 50 | 30 to <40 | < 30 |
| | 2.78 to 3.00 | 2.22 to <2.78 | 1.67 to <2.22 | <1.67 |
| Lactate, High | ULN to <2.0 x ULN | ≥2.0 x ULN without | Increased lactate with | Increased lactate with |
| | without acidosis | acidosis | pH <7.3 without life | pH <7.3 with life |
| | | | threatening | threatening |
| | 44. 45 *** | 1.5. 0.0 27737 | consequences | consequences |
| Lipase, High | 1.1 to <1.5 x ULN | 1.5 to <3.0 x ULN | 3.0 to <5.0 x ULN | ≥5.0 x ULN |
| Lipid Disorders | | | | |
| (mg/dL; mmol/L) Cholesterol, | 200 to <240 | 240 to <300 | ≥300 | NA |
| Fasting, High | 5.18 to < 6.19 | 6.19 to <7.77 | ≥7.77 | NA |
| ≥18 years of age | 3.10 10 \0.19 | 0.1910 <7.77 | 27.77 | |
| <18 years of age | 170 to <200 | 200 to <300 | ≥300 | NA |
| 10 years of age | 4.40 to <5.15 | 5.15 to <7.77 | ≥7.77 | NA. |
| LDL, Fasting, High | 130 to <160 | 160 to <190 | ≥190 | NA |
| ≥18 years of age | 3.37 to <4.12 | 4.12 to <4.90 | ≥4.90 | 1411 |
| >2 to <18 years of | 110 to <130 | 130 to <190 | ≥190 | NA |
| age | 2.85 to <3.34 | 3.34 to <4.90 | ≥4.90 | |
| Triglycerides, | 150 to 300 | >300 to 500 | >500 to <1,000 | >1,000 |
| Fasting, High | 1.71 to 3.42 | >3.42 to 5.7 | >5.7 to 11.4 | >11.4 |
| Magnesium <sup>16</sup> , Low | 1.2 to <1.4 | 0.9 to <1.2 | 0.6 to <0.9 | <0.6 |
| (mEq/L; mmol/L) | 0.60 to <0.70 | 0.45 to < 0.60 | 0.30 to < 0.45 | < 0.30 |
| Phosphate, Low | 2.0 to < LLN | 1.4 to < 2.0 | 1.0 to <1.4 | <1.0 |
| (mg/dL; mmol/L) | 0.81 to < LLN | 0.65 to < 0.81 | 0.32 to < 0.65 | < 0.32 |
| >14 years of age | | | | |
| 1 to 14 years of age | 3.0 to <3.5 | 2.5 to <3.0 | 1.5 to <2.5 | <1.5 |
| | 0.97 to <1.13 | 0.81 to <0.97 | 0.48 to < 0.81 | <0.48 |
| <1 year of age | 3.5 to <4.5 | 2.5 to <3.5 | 1.5 to <2.5 | <1.5 |
| | 1.13 to <1.45 | 0.81 to <1.13 | 0.48 to <0.81 | <0.48 |
| Potassium, High | 5.6 to <6.0 | 6.0 to <6.5 | 6.5 to <7.0 | ≥7.0 |
| (mEq/L; mmol/L) | 5.6 to <6.0 | 6.0 to <6.5 | 6.5 to <7.0 | ≥7.0 |
| Potassium, Low | 3.0 to <3.4 | 2.5 to <3.0 | 2.0 to <2.5 | <2.0 |
| (mEq/L; mmol/L) | 3.0 to <3.4 | 2.5 to <3.0 | 2.0 to <2.5 | <2.0 |

<sup>15</sup> Use the applicable formula (ie, Cockroft Gault in mL/min or Schwatrz in mL/min/1.73m<sup>2</sup>).

16 To convert a magnesium value from mg/dL to mmol/L, laboratories should multiply by 0.4114.

# JNJ-55471468, JNJ-55471494, JNJ-55471520, JNJ-55471585, JNJ-64219324

# Clinical Protocol VAC89220HPX2004 Amendment 5

| PARAMETER | GRADE 1<br>MILD | GRADE 2<br>MODERATE | GRADE 3<br>SEVERE | GRADE 4 POTENTIALLY |
|---|---|---|---|---|
| | MED | MODERATE | SEVERE | LIFE-<br>THREATENING |
| Sodium, High | 146 to <150 | 150 to <154 | 154 to <160 | ≥160 |
| (mEq/L; mmol/L) | 146 to <150 | 150 to <154 | 154 to <160 | ≥160 |
| Sodium, Low | 130 to <135 | 125 to <130 | 121 to <125 | ≤120 |
| (mEq/L; mmol/L) | 130 to <135 | 125 to <135 | 121 to <125 | ≤120 |
| Uric Acid, High | 7.5 to <10.0 | 10.0 to <12.0 | 12.0 to <15.0 | ≥15.0 |
| (mg/dL; mmol/L) | 0.45 to <0.59 | 0.59 to <0.71 | 0.71 to < 0.89 | ≥0.89 |

| | HEMATOLOGY | | | |
|---|---|---|---|---|
| PARAMETER | GRADE 1<br>MILD | GRADE 2<br>MODERATE | GRADE 3<br>SEVERE | GRADE 4 POTENTIALLY LIFE- THREATENING |
| Absolute CD4+ | | | | THREATENING |
| Count, Low | | | | |
| (cell/mm <sup>3</sup> ; cells/L) | 300 to <400 | 200 to <300 | 100 to <200 | <100 |
| >5 years of age | 300 to <400 | 200 to <300 | 100 to <200 | <100 |
| (not HIV infected) | | | | |
| Absolute Lymphocyte | | | | |
| Count, Low | 6004-4650 | 500 4 - 4600 | 250 4 4500 | -250 |
| (cell/mm <sup>3</sup> ; cells/L)<br>>5 years of age | 600 to <650<br>0.600 x 10 <sup>9</sup> to <0.650 | 500 to <600<br>0.500 x 10 <sup>9</sup> to <0.600 | 350 to <500<br>0.350 x10 <sup>9</sup> to <0.500 x | <350<br><0.350 x 10 <sup>9</sup> |
| (not HIV infected) | $x 10^9$ | $\begin{array}{ c c c c c c c c c c c c c c c c c c c$ | $10^9$ | <0.550 x 10 |
| Absolute Neutrophil | x 10 | x 10 | 10 | |
| Count (ANC), Low | | | | |
| (cells/mm <sup>3</sup> ; cells/L) | 800 to 1,000 | 600 to 799 | 400 to 599 | <400 |
| >7 days of age | $0.800 \times 10^9 \text{ to } 1.000 \times$ | $0.600 \times 10^9 \text{ to } 0.799 \times$ | $0.400 \times 10^9 \text{ to } 0.599 \times$ | $< 0.400 \times 10^9$ |
| | $10^{9}$ | 109 | 109 | |
| 2 to 7 days of age | 1,250 to 1,500 | 1,000 to 1,249 | 750 to 999 | <750 |
| | $1.250 \times 10^9 \text{ to } 1.500 \times$ | $1.000 \times 10^9 \text{ to } 1.249 \times 10^9 \text{ to } 1.249 \times 10^9 \times$ | $0.750 \times 10^9 \text{ to } 0.999 \times$ | $< 0.750 \times 10^9$ |
| <1.1 | 109 | 10° | 10° | <1.500 |
| ≤1 day of age | 4,000 to 5,000<br>4.000 x 10 <sup>9</sup> to 5.000 x | 3,000 to 3,999<br>3.000 x 10 <sup>9</sup> to 3.999 x | 1,500 to 2,999<br>1.500 x 10 <sup>9</sup> to 2.999 x | <1,500<br><1.500 x 10 <sup>9</sup> |
| | $10^9$ | $10^9$ | $1.300 \times 10^{\circ} 10 \ 2.999 \times 10^{9}$ | <1.500 x 10° |
| Fibrinogen, | 100 to <200 | 75 to <100 | 50 to <75 | <50 |
| Decreased (mg/dL; | 1.00 to <2.00 | 0.75 to <1.00 | 0.50 to < 0.75 | <0.50 |
| g/L) | OR | OR | OR | OR |
| | 0.75 to <1.00 x LLN | ≥0.50 to <0.75 x LLN | 0.25 to <0.50 x LLN | <0.25 x LLN |
| | | | | OR Associated with |
| ** *** 17 * | | | | gross bleeding |
| Hemoglobin <sup>17</sup> , Low | | | | |
| $(g/dL; mmol/L)^{18}$<br>$\geq 13 \text{ years of age}$ | 10.0 to 10.9 | 9.0 to <10.0 | 7.0 to <9.0 | <7.0 |
| (male only) | 6.19 to 6.76 | 5.57 to < 6.19 | 4.34 to <5.57 | <4.34 |
| ≥13 years of age | 9.5 to 10.4 | 8.5 to <9.5 | 6.5 to <8.5 | <6.5 |
| (female only) | 5.88 to 6.48 | 5.25 to <5.88 | 4.03 to <5.25 | <4.03 |
| 57 days of age to | 9.5 to 10.4 | 8.5 to <9.5 | 6.5 to <8.5 | <6.5 |
| <13 years of age | 5.88 to 6.48 | 5.25 to <5.88 | 4.03 to <5.25 | <4.03 |
| (male and female) | | l | | |
| 36 to 56 days of | 8.5 to 9.6 | 7.0 to <8.5 | 6.0 to <7.0 | <6.0 |
| age (male and | 5.26 to 5.99 | 4.32 to <5.26 | 3.72 to <4.32 | <3.72 |
| female) 22 to 35 days of | 9.5 to 11.0 | 8.0 to <9.5 | 6.7 to <8.0 | <6.7 |
| age (male and | 5.88 to 6.86 | 4.94 to <5.88 | 4.15 to <4.94 | <4.15 |
| female) | 2.50 10 0.00 | | 10 -1127 | .,,,,, |
| 8 to ≤21 days of | 11.0 to 13.0 | 9.0 to <11.0 | 8.0 to <9.0 | <8.0 |
| age (male and | 6.81 to 8.10 | 5.57 to <6.81 | 4.96 to <5.57 | <4.96 |
| female) | | | | |
| ≤7 days of age | 13.0 to 14.0 | 10.0 to <13.0 | 9.0 to <10.0 | <9.0 |
| (male and female) | 8.05 to 8.72 | 6.19 to <8.05 | 5.59 to <6.19 | <5.59 |
| INR, High | 1.1 to <1.5 x ULN | 1.5 to <2.0 x ULN | 2.0 to <3.0 x ULN | ≥3.0 x ULN |
| (not on anticoagulation therapy) | | | | |
| Methemoglobin (% | 5.0 to <10.0% | 10.0 to <15.0% | 15.0 to <20.0% | ≥20.0% |
| hemoglobin) | 2.0 10 -10.0/0 | 10.0 10 \15.0/0 | 15.0 10 \20.0/0 | _20.070 |
| | I | I | l | I |

<sup>&</sup>lt;sup>17</sup> Male and female sex are defined as sex at birth.

 $<sup>^{18}</sup>$  The conversion factor used to convert g/dL to mmol/L is 0.6206 and is the most commonly used conversion factor. For grading hemoglobin results obtained by an analytic method with a conversion factor other than 0.6206, the result must be converted to g/dL using the appropriate conversion factor for the particular laboratory.

# Clinical Protocol VAC89220HPX2004 Amendment 5

| PARAMETER | GRADE 1<br>MILD | GRADE 2<br>MODERATE | GRADE 3<br>SEVERE | GRADE 4 POTENTIALLY LIFE- THREATENING |
|---|---|---|---|---|
| PTT, High<br>(not on anticoagulation<br>therapy) | 1.1 to <1.66 x ULN | 1.66 to <2.33 x ULN | 2.33 to <3.00 x ULN | ≥3.00 x ULN |
| Platelets, Decreased (cells/mm³; cells/L) | 100,000 to <124,999<br>100.000 x 10 <sup>9</sup> to<br><124.999 x 10 <sup>9</sup> | 50,000 to <100,000<br>50.000 x 10 <sup>9</sup> to<br><100.000 x 10 <sup>9</sup> | 25,000 to <50,000<br>25.000 x 10 <sup>9</sup> to<br><50.000 x 10 <sup>9</sup> | <25,000<br><25.000 x 10 <sup>9</sup> |
| PT, High<br>(not on anticoagulation<br>therapy | 1.1 to <1.25 x ULN | 1.25 to <1.50 x ULN | 1.50 to <3.00 x ULN | ≥3.00 x ULN |
| WBC, Decreased<br>(cells/mm³; cells/L)<br>>7 days of age | 2,000 to 2,499<br>2.000 x 10 <sup>9</sup> to 2.499 x | 1,500 to 1,999<br>1.500 x 10 <sup>9</sup> to 1.999 x | 1,000 to 1,499<br>1.000 x 10 <sup>9</sup> to 1.499 x | <1,000<br><1.000 x 10 <sup>9</sup> |
| ≤7 days of age | 10°<br>5,500 to 6,999<br>5.500 x 10° to 6.999 x<br>10° | 10°<br>4,000 to 5,499<br>4.000 x 10° to 5.499 x<br>10° | 10 <sup>9</sup> 2,500 to 3,999 2,500 x 10 <sup>9</sup> to 3,999 x 10 <sup>9</sup> | <2,500<br><2.500 x 10 <sup>9</sup> |

| URINALYSIS | | | | |
|---|---|---|---|---|
| PARAMETER | GRADE 1<br>MILD | GRADE 2<br>MODERATE | GRADE 3<br>SEVERE | GRADE 4 POTENTIALLY LIFE- THREATENING |
| Glycosuria (random<br>collection tested by<br>dipstick) | Trace to 1+ or ≤250 mg | 2+ or >250 to ≤500 mg | >2+ or >500 mg | NA |
| Hematuria (not to be<br>reported based on<br>dipstick findings or on<br>blood believed to be of<br>menstrual origin) | 6 to <10 RBCs per<br>high power field | ≥10 RBCs per high<br>power field | Gross, with or without<br>clots OR With RBC<br>casts OR Intervention<br>indicated | Life threatening consequences |
| Proteinuria (random<br>collection tested by<br>dipstick) | 1+ | 2+ | 3+ or higher | NA |

### APPENDIX A: TOTAL BILIRUBIN TABLE FOR TERM AND PRETERM NEONATES

| PARAMETER | GRADE 1 | GRADE 2 | GRADE 3 | GRADE 4 |
|---|---|---|---|---|
| TAKAMETEK | MILD | MODERATE | SEVERE | POTENTIALLY |
| | WILL | MODERATE | SEVERE | LIFE- |
| | | | | THREATENING |
| Total Bilirubin <sup>19</sup> , | | | | |
| High (mg/dL; μmol/L) | | | | |
| 20 | | | | |
| Term Neonate <sup>21</sup> | | | | |
| <24 hours of age | 4 to <7 | 7 to <10 | 10 to <17 | ≥17 |
| | 68.4 to <119.7 | 119.7 to <171 | 171 to <290.7 | >290.7 |
| 24 to <48 hours of | 5 to <8 | 8 to <12 | 12 to <19 | ≥19 |
| age | 85.5 to <136.8 | 136.8 to <205.2 | 205.2 to <324.9 | <i>≥324.9</i> |
| 48 to <72 hours of | 8.5 to <13 | 13 to <15 | 15 to <22 | >22 |
| age | 145.35 to < 222.3 | 222.3 to <256.5 | 256.5 to <376.2 | _<br>≥376.2 |
| 72 hours to | 11 to <16 | 16 to <18 | 18 to <24 | >24 |
| <7 days of age | 188.1 to <273.6 | 273.6 to <307.8 | 307.8 to <410.4 | <i>-</i><br>≥410.4 |
| 7 to 28 days of age | 5 to <10 | 10 to <20 | 20 to <25 | ≥25 |
| (breast feeding) | 85.5 to <171 | 171 to <342 | 342 to <427.5 | ≥427.5 |
| 7 to 28 days of age | 1.1 to < 1.6 x ULN | 1.6 to <2.6 x ULN | 2.6 to <5.0 x ULN | ≥5.0 x ULN |
| (not breast | | | | |
| feeding) | | | | |
| Preterm Neonate <sup>21</sup> | | | | |
| 35 to <37 weeks | Same as for Total | Same as for Total | Same as for Total | Same as for Total |
| gestational age | Bilirubin, High, Term | Bilirubin, High, Term | Bilirubin, High, Term | Bilirubin, High, Term |
| | Neonate (based on | Neonate (based on | Neonate (based on | Neonate (based on |
| | days of age). | days of age). | days of age). | days of age). |
| 32 to <35 weeks | NA | NA | 10 to <14 | ≥14 |
| gestational age | | | 171 to <239.4 | ≥239.4 |
| and <7 days of age | | | | |
| 28 to <32 weeks | NA | NA | 6 to <10 | ≥10 |
| gestational age | | | 102.6 to <171 | ≥171 |
| and <7 days of age | | | | |
| <28 weeks | NA | NA | 5 to <8 | ≥8 |
| gestational age | | | 85.5 to <136.8 | ≥136.8 |
| and <7 days of age | | | | |
| 7 to 28 days of age | 5 to <10 | 10 to <20 | 20 to <25 | ≥25 |
| (breast feeding) | 85.5 to <171 | 171 to <342 | 342 to <427.5 | ≥427.5 |
| 7 to 28 days of age | 1.1 to < 1.6 x ULN | 1.6 to <2.6 x ULN | 2.6 to <5.0 x ULN | ≥5.0 x ULN |
| (not breast | | | | |
| feeding) | | | | |

<sup>19</sup> Severity grading for total bilirubin in neonates is complex because of rapidly changing total bilirubin normal ranges in the first week of life followed by the benign phenomenon of breast milk jaundice after the first week of life. Severity grading in this appendix corresponds approximately to cut offs for indications for phototherapy at grade 3 and for exchange transfusion at grade 4.  $^{20}$  A laboratory value of 1 mg/dL is equivalent to 17.1  $\mu$ mol/L.

<sup>&</sup>lt;sup>21</sup> Definitions: Term is defined as ≥37 weeks gestational age; near term, as ≥35 weeks gestational age; preterm, as <35 weeks gestational age; and neonate, as 0 to 28 days of age.

#### Attachment 2: HIV-risk Assessment

The following are intended as guidelines for the investigator to help identify potential vaccine trial participants at "low risk" for HIV infection in the US and Switzerland. Outside these countries, in addition to minimum requirements specified by the first two criteria defined below ("Have oral, vaginal or anal intercourse with an HIV-infected partner, or a partner who uses injection drugs" and "Give or receive money, drugs, gifts or services in exchange for oral, vaginal or anal sex"), low risk criteria as defined by local standards would be applicable.



# HVTN Low Risk Guidelines August 1, 2013

The following are intended as guidelines for the investigator to help identify potential vaccine trial participants at "low risk" for HIV infection in the US and Switzerland. These guidelines are based on behaviors within the last 6-12 months prior to enrollment; however, it may be appropriate to consider a person's behavior over a longer period of time than specified to assess the person's likelihood of maintaining low risk behavior. *Some volunteers may not be appropriate for enrollment even if they meet these guidelines*. These guidelines should be supplemented and interpreted with local epidemiologic information about HIV prevalence in your area and community networks. The investigator may review the risk level of any volunteer with the site PI and/or the Protocol Safety Review Team.

A volunteer may be appropriate for inclusion if he/she meets these guidelines:

#### SEXUAL BEHAVIORS

#### In the last 12 months did not:

- Have oral, vaginal, or anal intercourse with an HIV-infected partner, or a partner who uses injection drugs
- Give or receive money, drugs, gifts, or services in exchange for oral, vaginal, or anal sex

#### **AND**

In the last 6 months has abstained from penile/anal or penile/vaginal intercourse, OR

#### In the last 6 months:

• Had 4 or fewer partners of the opposite birth sex for vaginal and/or anal intercourse, OR

Is an MSM (person born male with partner(s) born male) who, in the **last 12 months**:

- Had 2 or fewer MSM partners for anal intercourse and had no unprotected anal sex with MSM, OR
- Had unprotected anal intercourse with only 1 MSM partner, within a monogamous relationship lasting at least 12 months (during which neither partner had any other partners). If the monogamous relationship ended, the volunteer may then have had protected anal intercourse with 1 other MSM partner (total 2 or fewer partners in the last 12 months).

Is a transgender person, regardless of the point on the transition spectrum, having sex with men (born male) and/or other transgender persons, who **in the last 12 months**:

- Had 2 or fewer partners for anal or vaginal intercourse, and had no unprotected anal or vaginal sex, OR
- Had unprotected anal or vaginal intercourse sex with 1 partner only within a monogamous relationship lasting at least 12 months (during which neither partner had any other partners). If the monogamous relationship ended, may then have had protected anal or vaginal sex with 1 other partner (total 2 or fewer partners in the last 12 months).

#### **AND**

Uses or intends to use condoms in situations which may include penile/anal or penile/vaginal intercourse with new partners of unknown HIV status, occasional partners, partners outside a primary relationship, and/or partners known to have other partners.

#### 2. NON-SEXUAL BEHAVIORS

#### In the **last 12 months** did not:

- Inject drugs or other substances without a prescription
- Use cocaine, methamphetamine, or excessive alcohol, which in the investigator's judgment, rendered the participant at greater than low risk for acquiring HIV infection

The investigator's judgment should consider local epidemiologic information about HIV prevalence in the area and community networks.

A volunteer is NOT appropriate for inclusion if he/she:

Acquired an STI (ie, new infection) in the last 12 months:

- Syphilis
- Gonorrhea
- Non-gonococcal urethritis
- HSV-2
- Chlamydia
- Pelvic inflammatory disease (PID)
- Trichomonas
- Mucopurulent cervicitis
- Epididymitis
- Proctitis
- Lymphogranuloma venereum
- Chancroid
- Hepatitis B

# Attachment 3: Test of Understandingi

Please read each question and answer whether the statement is True or False.

| True | False | 1. | The vaccines you will receive in this study protect against HIV. |
|---|---|---|---|
| True | False | 2. | You will need to come to the clinic for 4 scheduled visits over the next 1.5 years. |
| True | False | 3. | The vaccines in this study can give you HIV. |
| True | False | 4. | One purpose of this study is to determine if these vaccines are safe to administer to humans. |
| True | False | 5. | Participants in this study will need to avoid engaging in activities that may expose them to HIV infection. |
| True | False | 6. | You may take other experimental (test) products while you are taking part in this study. |
| True | False | 7. | You may withdraw from the study at any time if you choose or your participation may be stopped if the study team decides it is in your best interest. |
| True | False | 8. | Women participating in this study are permitted to become pregnant starting 3 months after the last vaccination. |
| True | False | 9. | A participant in this study may experience side effects after vaccination. |
| True | False | 10. | Some participants in this study may develop a positive HIV-test result, despite the fact that they are not HIV infected. |

CONFIDENTIAL - FOIA Exemptions Apply in U.S.

<sup>&</sup>lt;sup>i</sup> Adaptations to the TOU are allowed for local purposes, after IRB and sponsor approval.

# **Attachment 4: Social Impact Questionnaire**

# Vaccine Research Center (VRC) Social Impact Case Report Form<sup>j</sup>

| | Social Impact Question | Yes or No | If Yes, did you consider this to be harmful to you? |
|---|---|---|---|
| 1. Personal | Did you have problems with family, friends, significant others or sex partners because of participation in this clinical trial? | □ Yes □ No | □ Yes □ No |
| Relationships | Comment: resolved; | □ continuing | □ mild; □ moderate; □ major |
| 2. Travel or Immigration | Did you have problems getting legal permission to travel to or from another country, such as being denied a visa, or having problems with immigration/naturalization because of participation in this clinical trial? | □ Yes □ No | □ Yes □ No |
| | Comment: resolved; | □ continuing | □ mild; □ moderate; □ major |
| 3. Employment | Have you been turned down for a new job, lost a job, or had other problems at work because of participation in this clinical trial? | □ Yes □ No | □ Yes □ No |
| | Comment: resolved; | □ continuing | ☐ mild; ☐ moderate; ☐ major |
| 4. Education | Have you been turned down by an educational program, told to leave an educational program, or had other problems at school because of participation in this clinical trial? | □ Yes □ No | □ Yes □ No |
| | Comment: resolved; | □ continuing | □ mild; □ moderate; □ major |
| 5. Medical or<br>Dental | Have you been refused medical or dental care or treated negatively by a health care provider because of participation in this clinical trial? | □ Yes □ No | □ Yes □ No |
| | Comment: resolved; | continuing | □ mild; □ moderate; □ major |
| 6. Health<br>Insurance | Have you lost health insurance, had a problem getting new health insurance, or had other problems related to health insurance because of participation in this clinical trial? | □ Yes □ No | □ Yes □ No |
| | Comment: resolved; | □ continuing | ☐ mild; ☐ moderate; ☐ major |
| 7. Life Insurance | Have you lost life insurance, had a problem getting new life insurance, or had other problems related to life insurance because of participation in this clinical trial? | ☐ Yes ☐ No | □ Yes □ No |
| | Comment: resolved; | □ continuing | □ mild; □ moderate; □ major |
| 8. Housing | Have you had trouble getting or keeping housing, or had other problems related to housing because of participation in this clinical trial? | □ Yes □ No | □ Yes □ No |
| | Comment: resolved; | □ continuing | □ mild; □ moderate; □ major |
| 9. Military/Other<br>Government<br>Agency | Have you had a problem with the military or any other government agency because of participation in this clinical trial? | ☐ Yes ☐ No | □ Yes □ No |
| Agency | Comment: resolved; | □ continuing | □ mild; □ moderate; □ major |
| 10. Other | Have you had any other problem not covered by the other questions because of anything related to participation in this clinical trial? | □ Yes □ No | □ Yes □ No |
| | Comment: resolved; | continuing | ☐ mild; ☐ moderate; ☐ major |

-

<sup>&</sup>lt;sup>j</sup> Adaptations to the social impact questionnaire are allowed for local purposes, after IRB and sponsor approval.

### **INVESTIGATOR AGREEMENT**

I have read this protocol and agree that it contains all necessary details for carrying out this study. I will conduct the study as outlined herein and will complete the study within the time designated.

I will provide copies of the protocol and all pertinent information to all individuals responsible to me who assist in the conduct of this study. I will discuss this material with them to ensure that they are fully informed regarding the study intervention, the conduct of the study, and the obligations of confidentiality.

| <b>Coordinating Investigato</b> | or (where required): | | |
|---|---|---|---|
| Name (typed or printed): | | | |
| Institution and Address: | | | |
| Signature: | | Date: | |
| | | | (Day Month Year) |
| Principal (Site) Investiga | tor: | | |
| Name (typed or printed): | | | |
| Institution and Address: | | | |
| Telephone Number: | | | |
| Signature: | | Date: | |
| | | | (Day Month Year) |
| Sponsor's Responsible M | | | |
| Name (typed or printed): | PPD | | |
| Institution: | Janssen Research & Development | | |
| Signature: electronic sig | nature appended at the end of the protocol | Date: | |
| | | | (Day Month Year) |

**Note:** If the address or telephone number of the investigator changes during the study, written notification will be provided by the investigator to the sponsor, and a protocol amendment will not be required.

#### **LAST PAGE**

# **Signature**

| User | Date | Reason |
|------|----------------------------------|-------------------|
| PPD | 29-Oct-2021<br>13:47:24<br>(GMT) | Document Approval |